A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Effects of Multiple Subcutaneous Injections of Elamipretide on Left Ventricular Function in Subjects with Stable Heart Failure with Reduced Ejection Fraction

NCT02788747

**04 DECEMBER 2017** 



## STATISTICAL ANALYSIS PLAN

**Trial Sponsor:** Stealth BioTherapeutics, Inc.

**Protocol Number:** SPIHF-201 **IND Number:** N/A **EUDRACT** 

Number: 2014-005724-10 Investigational Drug: Elamipretide (MTP-131)

**Indication:** Heart Failure with reduced Ejection

Fraction (HFrEF)

Dosage Form/Strength: Elamipretide (MTP-131) 40 mg/1 mL of

sterile solution for subcutaneous injection

with doses of 4 mg or 40 mg administered once daily

**Protocol Title:** A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Effects of Multiple Subcutaneous Injections of Elamipretide on Left Ventricular Function in Subjects with Stable Heart Failure with Reduced Ejection Fraction

\_\_\_\_\_

The information in this document is confidential and is proprietary to Stealth Biotherapeutics. It is understood that information in this document shall not be disclosed to any third party, in any form, without prior written consent of an authorized officer of Stealth Biotherapeutics.

Version 1.0 Page 1 of 37 CONFIDENTIAL



# Statistical Analysis Plan Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

## FINAL SIGN-OFF APPROVAL

| Author<br>Biostatistician: | Meleana Dunn<br>Principal Biostatistician<br>Everest Clinical Research | |
|---|---|---|
| | Meleana Dunn<br>Signature | 05 Oec20f |
| Peer Review<br>Biostatistician: | Dean Rutty Executive Director, Biometrics Everest Clinical Research | |
| | Signature | 05 DEC 2017<br>Date |
| Approved by: | Douglas Weaver Chief Medical Officer Stealth BioTherapeutics Signature | 5 Dec 2017 |
| Approved by: | James Carr Chief Clinical Development Officer Stealth BioTherapeutics | 5 Dec 2017 |
| | Signature | Date |
| Approved by: | Jeffrey Finman Statistical Consultant Stealth BioTherapeutics | |
| | 6: 25 | 05-Duc-201 |
| | Signature | Date |

Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

#### CHANGE LOG FOR CHANGES MADE AFTER THE INITIAL APPROVAL

| Revision<br>Date* | Section(s)<br>Modified | Brief Description of Revision(s) or<br>Reason(s) for Revision | Modifications Reviewed and Approved by** |
|---|---|---|---|
| | | | Sponsor, Everest |

<sup>\*</sup> Update the Last Revision Dates on the cover page and the document header.

#### **TABLE OF CONTENTS**

| 1. INTRODUCTION | 8 |
|--------------------------------------------------|----|
| 2. STUDY OBJECTIVES | 9 |
| 2.1 Primary Objective | 9 |
| 2.2 Secondary Objectives | |
| 2.3 Exploratory Objectives | |
| 3. STUDY DESIGN | 10 |
| 3.1 Study Design | 10 |
| 3.2 Randomization | 11 |
| 3.3 Hypothesis Testing | 12 |
| 3.4 Interim Analysis | |
| 3.5 Sample Size | |
| 3.6 Schedule of Assessments and Study Procedures | 12 |
| 4. DATA AND ANALYTICAL QUALITY ASSURANCE | 16 |
| 5. ANALYSIS POPULATIONS | 16 |
| 5.1 Safety Population | 16 |
| 5.2 Intent-to-Treat (ITT) Population | 16 |
| 5.3 Per-Protocol (PP) Population | |
| 6. SPECIFICATION OF ENDPOINTS AND VARIABLES | 16 |
| 6.1 Demographic and Baseline Characteristics | 16 |

<sup>\*\*</sup> Provide person's initial and last name.

Statistical Analysis Plan Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

| 6.2 Efficacy | 17 |
|-------------------------------------------------|----|
| 6.2.1 Study Day and Visit Window Definitions | 17 |
| 6.2.2 Primary Efficacy Variables | 18 |
| 6.2.3 Secondary Efficacy Variables | 18 |
| 6.2.4 Exploratory Efficacy Variables | 19 |
| 6.2.5 Plasma Concentration | 19 |
| 6.3 Safety | 20 |
| 6.3.1 Study Day and Visit Window Definitions | 20 |
| 6.3.2 Extent of Exposure to Study Medication | 21 |
| 6.3.3 Adverse Events | 21 |
| 6.3.4 Laboratory Data | 23 |
| 6.3.5 Vital Signs | |
| 6.3.6 Electrocardiogram (ECG) | 25 |
| 6.3.7 Physical Examination | 25 |
| 6.3.8 Pregnancy Test | |
| 6.3.9 Concomitant Medications/Treatments | 25 |
| 7. STATISTICAL ANALYSIS | |
| 7.1 General Data Handling Rules and Definitions | 27 |
| 7.2 Subject Disposition | 28 |
| 7.3 Demographic and Baseline Characteristics | |
| 7.4 Efficacy Analyses | |
| 7.4.1 Primary Efficacy | |
| 7.4.2 Secondary Efficacy | |
| 7.4.3 Exploratory Efficacy | 30 |
| 7.4.4 Efficacy Subgroup Analyses | |
| 7.5 Plasma Concentration Analyses | |
| 7.6 Safety Analyses | |
| 7.6.1 Extent of Exposure to Study Medication | |
| 7.6.2 Adverse Events | |
| 7.6.3 Deaths | |
| 7.6.4 Clinical Laboratory Evaluations | |
| 7.6.5 Vital Signs | |
| 7.6.6 Electrocardiogram (ECG) | |
| 7.6.7 Physical Examination | |
| 7.6.8 Concomitant Medications/Treatments | |
| 8. ANALYSES PERFORMED BEFORE DATABASE CLOSURE | |
| 9. CHANGES FROM METHODS PLANNED IN THE PROTOCOL | |
| 10. STATISTICAL SOFTWARE | |
| 11. REFERENCES | |
| APPENDIX 1 DATA HANDLING RULES | |
| APPENDIX 2 SAS CODE FOR STATISTICAL ANALYSES | 36 |




| APPENDIX | 3 | REFERENCE | RANGES | AND | CLINICALLY | RELEVANT | CHANGES | FROM |
|---|---|---|---|---|---|---|---|---|
| BASELINE I | FOR | MARKED LA | BORATOR | Y ABN | ORMALITIES | | | 37 |
| APPENDIX 4 | 4 M | OCKUP TABLI | ES. LISTIN | GS. AN | ID GRAPHS (TI | LGS) | | 38 |

#### 6-minute walk test

AE Adverse event

ATP Adenosine triphosphate

ATP<sub>max</sub> Maximal ATP synthetic mitochondrial energy coupling AUC Area under the plasma concentration versus time curve

BMI Body mass index

BP Blood pressure

BSA Body surface area

BUN Blood urea nitrogen

CK Creatine kinase

ECG Electrocardiogram

eCRF electronic Case Report Form

EF Ejection fraction

DBP Diastolic blood pressure

HFrEF Heart failure with reduced ejection fraction

Hgb Hemoglobin

IMP Investigational medicinal product

ITT Intent-to-treat
IV Intravenous

IWRS Interactive web-based response system

KCCQ Kansas City Cardiomyopathy Questionnaire

LA Left atria

LV Left ventricle

LV EDV Left ventricular end diastolic volume

LVEF Left ventricular ejection fraction



## Statistical Analysis Plan Protocol No. SPIHF-201


| 6MWT | |
|--------------|--------------------------------------|
| Abbreviation | Term |
| Mb | Myoglobin |
| LV ESV | Left ventricular end systolic volume |

**GLOSSARY OF ABBREVIATIONS** 




MedDRA Medical Dictionary for Regulatory Activities

MRI Magnetic resonance imaging

MRS Magnetic resonance spectroscopy

MTP-131 Elamipretide

NAD Nicotine adenine dinucleotide

NT-pro-BNP N-terminal pro-brain natriuretic peptide

PCr Phosphocreatine

31P Phosphorus-31

P/O Mitochondrial coupling

PT Preferred term

RBC Erythrocyte count

RV Right ventricle

RVSP Right ventricular systolic pressure

SAE Serious adverse event

SAP Statistical analysis plan

SBP Systolic blood pressure

SC Subcutaneous

SOC System organ class

TEAE Treatment-emergent adverse event

US United States

WBC Leukocytes

WHO-DD World Health Organization Drug Dictionary

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) outlines the planned statistical methods for the display, summary and analysis of data collected within the scope of Stealth BioTherapeutics, Inc. protocol SPIHF-201 version 8.0 dated 21 March 2017. The analysis of the data should allow




changes in the plan to the extent that deviations from the original plan would provide a more reliable and valid analysis of the data. As such, deviations from this SAP must be substantiated by a sound statistical rationale and described in the clinical study report (CSR).

The SAP should be read in conjunction with the study protocol and the electronic Case Report Forms (eCRFs). This version of the SAP has been developed using the final version of the protocol mentioned above and the final version of the annotated eCRFs dated 16 June 2016.

The SAP details the analysis of the data collected in the study and the presentation of the results of the analyses. The table, listing, and figure (TLF) shells are displayed in a companion document which provides information on the layout of the data displays. Analysis dataset specifications will be developed to detail the programming specifications and mapping rules needed to create the analysis datasets and the TLFs.

All statistical analyses will be performed using SAS® version 9.3, or higher. Adverse events will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA 19.1 or newer).

This study is a Phase 2, randomized, double-blind, placebo-controlled, multiple dose study, conducted in up to 20 centers in Europe, enrolling 66 subjects with previous evidence of stable heart failure with reduced ejection fraction (HFrEF) to evaluate the effects of multiple subcutaneous (SC) doses of elamipretide on left ventricular end systolic volume (LV ESV).

#### 2. STUDY OBJECTIVES

#### 2.1 Primary Objective

To evaluate the effects of multiple SC doses of elamipretide on LV ESV assessed by cardiac Magnetic Resonance Imaging (MRI).

#### 2.2 Secondary Objectives

- To evaluate the safety and tolerability of multiple SC doses of elamipretide.
- To evaluate the effects of multiple SC doses of elamipretide on left ventricular (LV) systolic and diastolic function to include: LV volumes, LV global longitudinal strain, left atrial (LA) volume, LV mass, extent of mitral and tricuspid regurgitation severity, and right ventricular (RV) function (original and indexed to BSA).


#### 2.3 Exploratory Objectives

To evaluate the effects of multiple SC doses of elamipretide on:

- 6-minute walking distance
- Quality of life using the KCCQ
- N-terminal pro-brain natriuretic peptide (NT-pro-BNP) levels

#### 3. STUDY DESIGN

#### 3.1 Study Design

This is a randomized, double-blinded, placebo-controlled, multiple dose Phase 2 study in subjects with HFrEF. The objectives are to evaluate the effects of multiple SC doses of elamipretide on LV ESV, LV systolic and diastolic function, LV volumes, LV global longitudinal strain, LA volume, LV mass, mitral and tricuspid regurgitation severity, and RV function in subjects with stable heart failure with reduced ejection fraction. After completing the screening period, approximately 66 subjects will be randomized, in a 1:1:1 ratio, to receive either placebo, 4 mg elamipretide, or 40 mg elamipretide once daily for 28 consecutive days.

Efficacy will be assessed with the following measurements:

- LV ESV assessed by MRI
- Left ventricular ejection fraction (LVEF) and left ventricular end diastolic volume (LV EDV) assessed by MRI
- The following parameters by echocardiography:
  - o E/A (ratio between early and late mitral inflow velocity),
  - E/e' (Ratio between early mitral inflow velocity and mitral annular early diastolic velocity)
  - o LV EDV, LV ESV and biplane ejection fraction (EF)
  - LV global longitudinal strain
  - o LA volume o LV mass
  - Mitral regurgitation severity o Tricuspid regurgitation severity o RV fractional area change o RV systolic pressure (RVSP)
- Distance walked (meters) on the 6-minute walk test (6MWT)




- Kansas City Cardiomyopathy Questionnaire (KCCQ) score
- Levels of NT-pro-BNP

Subjects will be screened for reduced EF, defined as LVEF  $\leq$  40%, by 2-D echocardiography.

There are 3 study treatment groups randomized in equal ratio:

- Elamipretide (MTP-131) 40 mg of 40 mg/1 mL of sterile solution, administered as a once daily SC injection for 28 consecutive days.
- Elamipretide (MTP-131) 4 mg of 40 mg/1 mL of sterile solution, administered as a once daily SC injection for 28 consecutive days.
- Placebo (excipients used to manufacture the investigational drug but without the active drug substance) administered as a once daily SC injection for 28 consecutive days.

#### 3.2 Randomization

Randomization will be used in this study to avoid bias in the assignment of study treatments to subjects, to increase the likelihood that known and unknown subject attributes (e.g., demographics and baseline characteristics) are balanced across treatment groups, and to enhance the possible validity of statistical comparisons across treatment groups. Blinded treatment will be used to reduce potential bias during data collection and evaluation of endpoints. Only those subjects who meet protocol-specified criteria for stable heart failure with reduced ejection fraction will be randomized to study treatment.

At Day 1, after the eligibility criteria have been confirmed, a treatment kit number will be assigned to each subject on the basis of a centralized computer-generated randomization schedule administered by IWRS. Subjects will be randomized into 1 of 3 treatment groups in a 1:1:1 fashion to receive either elamipretide 4 mg, elamipretide 40 mg, or placebo, so that a target of 22 subjects will be randomized to the elamipretide 4 mg dose group, 22 subjects will be randomized to the elamipretide 40 mg dose group, and 22 subjects will be randomized to the placebo treatment group. Treatment kits for placebo will specify injection volumes of either 0.1 or 1 mL in order to maintain the blind. This will be accomplished by administering a randomization schedule in randomized blocks of 6 with a ratio of 2:2:1:1 (elamipretide 4 mg [0.1 mL], elamipretide 40 mg [1 mL], placebo [0.1 mL] or placebo [1 mL]). This design maintains the 1:1:1 ratio of elamipretide 4 mg, elamipretide 40 mg, and placebo in addition to ensuring the complete blind to study treatment.


#### 3.3 Hypothesis Testing

Primary hypothesis:

<u>Null hypothesis  $H_0$ </u>: There is no difference between the elamipretide 40 mg and placebo treatment groups in change in LV ESV at Week 4 from baseline.

Alternative hypothesis  $H_a$ : There is a difference between the elamipretide 40 mg and placebo treatment groups in change in LV ESV at Week 4 from baseline.

The elamipretide 4 mg treatment will also be compared to placebo as a secondary hypothesis.

#### 3.4 Interim Analysis

No formal interim analyses are planned for this study.

### 3.5 Sample Size

The target sample size of 22 subjects per treatment group provides 80% power to detect an 8 mL difference between treatment groups in LV ESV, as measured by MRI, assuming a standard deviation of 9.4 mL.

#### 3.6 Schedule of Assessments and Study Procedures



Protocol No.: SPIHF-201

Last Revision Date: 04 DECEMBER 2017

| | Screening Period | | Treatn | nent Period | Follow-Up Period | |
|---|---|---|---|---|---|---|
| | Days -28 to -1<br>(Screening Visit) | Day 1 <sup>a</sup><br>(Baseline) | Week 1 (Day 8 + 3) | Week 2<br>(Day 15 ± 3) | Week 4/ED <sup>b</sup> (Day 29 + 3) | Week 6<br>(Day 43 ± 3) |
| Informed Consent | X | | | | | |
| Demographics | X | | | | | |
| Randomization | | X | | | | |
| Review of Inclusion/Exclusion Criteria | X | X | | | | |
| Relevant Medical History <sup>c</sup> | X | X | | | | |
| Concomitant Medication Review | X | X | X | X | X | X |
| Review AEs | | X | X | X | X | X |
| Cardiovascular Physical Examination <sup>d</sup> | X | X | X | X | X | X |
| Vital Signs <sup>e</sup> | X | X | X | X | X | X |
| 12-Lead ECG | X | X | X | X | X | X |
| Blood Chemistry & Hematology | X | X | X | X | X | X |
| PK Samples <sup>f</sup> | | X | X | X | X | X |
| Urinalysis | X | X | | | X | |
| Pregnancy Test <sup>g</sup> | X | X | | | X | |
| Echocardiography <sup>h</sup> | X | X | | | X | X |
| Cardiac MRI <sup>i</sup> | X | | X | | X | |
| KCCQ | | X | | | X | |
| NT-pro-BNP | | X | X | X | X | X |
| 6-Minute Walk Test | | X | | | X | |
| Study Medication Dispensing | | X | X | X | | |
| Study Medication Injection <sup>j</sup> | | X | | | X | |
| ISR Self-Assessment Questionnaire | | X | | | X | |
| Visiting Nurse/Investigator ISR Assessment <sup>k</sup> | | X | | | X | |

Protocol No.: SPIHF-201 Last Revision Date: 04 DECEMBER 2017

- <sup>a</sup> All Day 1 assessments should be performed prior to administering the first dose of study medication except the ISR assessments (as described in Section 6.3.9) and blood drawn for plasma analysis of elamipretide and metabolites (45 minutes post-injection ±15 minutes) (as described in Section 6.3.8.5) which should be completed after study medication administration. <sup>b</sup> If a subject discontinues study medication early, the subject will have an Early Discontinuation Visit and will be asked to complete the Week 4 assessments. <sup>c</sup> At the Screening Visit, a relevant medical history will be taken. Relevant medical history will be updated at the Day 1 visit. <sup>d</sup> Cardiovascular physical examination including lung auscultation and weight. Height will only be measured at the Screening Visit. <sup>e</sup> Vital signs measurements will include temperature, heart rate, respiration rate and blood pressure, recorded in the sitting position after at least 10 minutes rest.
- Blood samples for PK determinations of elamipretide and metabolites concentrations will be collected before administration of study medication and at 45 minutes (±15 minutes) post-dose at the Day 1, Week 1, and Week 2 visits, and at any time point at the Week 4 and 6 visit.
- Serum pregnancy test will be done for women of childbearing potential at the Screening visit. Urine pregnancy test will be done for women of childbearing potential on Day 1 and Week 4. The results of the Day 1 pre-dose pregnancy test must be evaluated before randomization to ensure eligibility.
- At the Screening Visit, only a 2-D echocardiography will be performed and it will be performed prior to Step 2 (blood draw, urinalysis) and Step 3 (cardiac MRI) screening procedures. Both 2-D and 3-D echocardiography will be performed at the Day 1, Week 4 and Week 6 visits.
- At the Screening visit, subjects will undergo delayed gadolinium-enhanced cardiac MRI prior to study medication injection. At the Week 1 visit, subjects will undergo cardiac MRI approximately 1 to 6 hours following injection of study medication.
- At Day 1, study medication injection will occur after the completion of baseline procedures (as noted in footnote a). Study medication will be administered daily by a Visiting Nurse, except on Study Visits, at Days 1 through 3 and during the Week 1 and Week 2 visits. The last dose of study medication will be administered on the day prior to the Week 4 visit.
- At each home visit, the Visiting Nurse will assess the current day's injection site. At Days 1 through 3, Week 1 and Week 2 visits, the Investigator (or designee) will assess the current day's injection site. The assessment will evaluate erythema, pain, swelling, and pruritus at the injection site at approximately 15 minutes post-injection. If any reaction is apparent, the injection site will also be evaluated at 30 minutes post-injection.






#### 4. DATA AND ANALYTICAL QUALITY ASSURANCE

The overall quality assurance procedures for the study data, statistical programming and analyses are described in the Everest's Standard Operating Procedures. Detailed data management procedures are documented in the Data Management Plan, Data Validation Check Specifications, and Data Review Plan. Detailed statistical and programming quality control and quality assurance procedures are documented in the Statistical Analysis and Programming QC/QA Plan.

#### 5. ANALYSIS POPULATIONS

#### 5.1 Safety Population

Safety population includes all subjects receiving at least one dose of the investigational medicinal product (IMP). Safety analyses will be conducted on the safety population according to the treatment received.

## 5.2 Intent-to-Treat (ITT) Population

The Intent-To-Treat Population (ITT) will consist of all subjects who were randomized and receive at least 1 dose of IMP. The ITT population will be the primary analysis for efficacy assessments. Efficacy analyses will be conducted on the ITT Population according to the treatment group to which the subjects were randomized.

#### 5.3 Per-Protocol (PP) Population

The Per-Protocol Population (PP) will consist of all randomized subjects receiving at least one dose of the IMP without major protocol violations/deviations. The list of major protocol violations/deviations will be identified by the Sponsor prior to final database lock for the study that would lead to exclusion from the PP analysis. The PP population will be a sensitivity analysis to the ITT analysis for efficacy assessments. If there are no major deviations which exclude data from the PP population, the PP analysis will not be reported.

#### 6. SPECIFICATION OF ENDPOINTS AND VARIABLES

#### 6.1 Demographic and Baseline Characteristics

Demographic variables consist of the following:

- Age in years (continuous) derived as the integer of (informed consent date date of birth + 1)/365.25
- Gender


- Race
- Ethnicity

Baseline characteristics consist of the following:

- Weight (kg)
- Height (cm)
- BMI (kg/m²) derived as
- weight in kg divided by (height in m)<sup>2</sup>
- Vital signs (heart rate, systolic blood pressure, diastolic blood pressure, and temperature [oral or tympanic])
- Physical cardiovascular examination (any clinically significant abnormalities (yes, no))
- Medical and surgical history
- Prior medications

#### 6.2 Efficacy

The effect of multiple SC doses of elamipretide on left ventricular end systolic volume is assessed using the change in LVESV between Baseline and Week 4.

#### 6.2.1 Study Day and Visit Window Definitions

The date the subject is randomized and is expected to receive the first dose of study medication will be used as the Study Day 1.

Study day will be calculated as follows:

```
Before study day 1: Study Day = date of assessment – date of study day 1.
On or after study day 1: Study Day = date of assessment – date of study day 1 + 1.
```

The last study date is the last visit date of any scheduled, unscheduled or early discontinuation visits. The last Study Day is calculated as:

Last Study Day = last study date - date of study day 1 + 1.

The target study days are summarized in Table 1 below:

#### **Table 1. Visit Windows for Efficacy Assessments**


| Scheduled<br>Visit Number | Visit (label) | Time<br>Interval<br>(day) | Target Time<br>Point (day) |
|---|---|---|---|
| 0 | Screening | -28 to -1 | -28 to -1 |
| 1 | Baseline/Day 1 | 1 | 1 |
| 2 | Week 1 | 1 (postdose)<br>to 11 | 8 |
| 3 | Week 2 | 12 to 22 | 15 |
| 4 | Week 4 | 23 to 36 | 29 |
| 5 | Week 6 | ≥37 | 43 |

The baseline assessment is defined as the last assessment prior to the first dose of study medication. In some cases, these baseline measurements are obtained at the screening visit.

If multiple assessments fall in the same visit window, the non-missing assessment closest to target time point will be selected for analysis. Data obtained during unscheduled visits will be allocated to the scheduled visit corresponding to the visit window they fall in. If an unscheduled visit is closer to the target time point than the scheduled visit, a blinded review will be done at the end of the study to determine which visit to use. The choice will depend on how far off the scheduled visit occurred and what data was collected at each of the visits.

## **6.2.2** Primary Efficacy Variables

The primary efficacy endpoint is change in LV ESV assessed by MRI at Week 4 from baseline.

#### **6.2.3** Secondary Efficacy Variables

Secondary efficacy endpoints are changes from baseline for the following measures:

- LVEF and LV EDV assessed by MRI
- The following parameters by echocardiography:
  - o E/A (ratio between early and late mitral inflow velocity),
  - o E/e' (Ratio between early mitral inflow velocity and mitral annular early diastolic velocity) o LV EDV, LV ESV and biplane ejection fraction (EF)




- LV global longitudinal strain
- LA volume
- o LV mass
- Mitral regurgitation severity o Tricuspid regurgitation severity o RV fractional area change o RV systolic pressure (RVSP)

Change from baseline for the above MRI measures will be assessed at Week 1 (approximately 1 to 6 hours following injection of study medication) and at Week 4, and for the echocardiography measures at Weeks 4 and 6.

The measures of volume, LV ESV, LV EDV, LA volume, LV mass, RV ESV, RV EDV, and RV myocardial mass, will be indexed to body surface area (BSA) by dividing the measures by BSA. All analyses will be done on the indexed values. Listings will include both indexed and nonindexed values.

#### **6.2.4** Exploratory Efficacy Variables

Exploratory efficacy endpoints are changes from screening for the following measures:

- Distance walked (meters) during 6MWT
- Levels of NT-pro-BNP
- KCCO score

Change from baseline for the Distance walked measure will be assessed at Week 4, the levels of NT-pro-BNP measure at Weeks 1, 2, 4, and 6, and as an AUC for visits Baseline, Weeks 1, 2, 4, and 6, and for the KCCQ measure at Week 4.

#### 6.2.5 Plasma Concentration

Blood samples for PK determinations of elamipretide and metabolites (M1, M2) concentrations will be collected before administration of study medication and at 45 minutes  $\pm 15$  minutes postdose at the Day 1, Week 1 and Week 2 visits, and at any time point at the Week 4 and Week 6 visits.

Plasma samples will be analyzed for MTP-131 concentrations using a validated liquid chromatography/ tandem mass spectrometry assay.


#### 6.3 Safety

The safety profile of elamipretide will be assessed through the recording, reporting, and analyzing of AEs, clinical evaluations, and laboratory tests. Safety variables include the following:

- Adverse events and serious adverse events
- Local laboratory measurements clinical chemistry and hematology with specific attention to Na+ and K+
- Urinalysis
- Vital signs
- Electrocardiogram (ECG)
- Physical examination
- Pregnancy
- Concomitant medications/treatments
- Injection site reaction (ISR)

#### 6.3.1 Study Day and Visit Window Definitions

The term "Safety analysis period" is from the first dose of study medication to 30 days after the last dose of study drug.

Study day is defined as in Section 6.2.1.

The date at the first dose of study medication is used as Study Day 1. The target study days are summarized in Table 2 below:

| Table 2. Visit Windows for Safety Assessments | | | |
|---|---|---|---|
| Scheduled Visit<br>Number | Visit (label) | Time Interval (day) | Target Time Point (day) |
| 0 | Screening | -28 to -1 | -28 to -1 |
| 1 | Baseline/Day 1 | 1 | 1 |
| 2 | Week 1 | 1 (postdose) to 11 | 8 |
| 3 | Week 2 | 12 to 18 | 15 |
| 4 | Week 4 | 23 to 36 | 29 |
| 5 | Week 6 | >37 | 43 |




Data obtained during unscheduled visits will be allocated to the scheduled visit corresponding to the visit window they fall in. If multiple assessments fall in the same visit window, the nonmissing assessment closest to target time point will be selected for analysis.

Baseline values for clinical laboratory tests, vital signs and ECGs will be defined as the last evaluation performed prior to the first dose of study medication.

#### **6.3.2** Extent of Exposure to Study Medication

Elamipretide 4 mg or 40 mg, or Placebo (excipients used to manufacture the investigational drug but without the active drug substance) will be administered as a once daily SC injection for 28 consecutive days.

The study medication exposure variables include:

- Study treatment exposure (days) = Treatment end date treatment start date number of days of missed doses + 1
- Study treatment compliance (%) = Average over total time of exposure (Treatment start date to treatment end date):

For each day:

100 × Day X Total Volume Expected Day X Total Volume Injected

The average calculation should include all days from the treatment start date to the treament end date, including days with missed doses.

#### **6.3.3** Adverse Events

The AE reporting period begins when the subject signs the ICF and continues through the clinical study's post treatment follow-up period, defined as 14 days after last administration of study medication. Within the study, all subjects who took at least 1 dose of IMP, whether they completed the treatment period or not, should enter the 14-day period as defined above. If a subject is documented as lost-to follow-up, ongoing/unknown outcome AEs will not be followedup.

Adverse events will be collected and coded using the latest version of the Medical Dictionary for




Regulatory Activities (MedDRA 19.1 or newer). An adverse event is considered treatmentemergent if the date of onset is on or after the date of first dose of study medication, or worsening during the treatment period (intensity/severity changed to worsen grades). All reported AEs will be listed, but only treatment-emergent adverse events (TEAEs) will be summarized. All adverse events are assessed by investigators on intensity, relationship to study drug, and seriousness according to the definitions in protocol Sections 9.7.1.1 and 9.7.1.2.

Intensity: AEs will be rated as Mild, Moderate or Severe.

Relationship to study AEs will be qualified as either related (unlikely, probably or drug: possibly related) or non-related (unrelated) to study drug. Seriousness: AEs will be categorized as serious or non-serious

#### **Adverse Events Counting Rules:**

- 1. A subject with more than one different adverse event in a particular system organ class (SOC) will be counted only once in the total of subjects experiencing adverse events in that particular SOC.
- 2. A subject having experienced the same event (AE preferred term) more than once during the study will be counted only once in the number of subjects with that event.
- 3. A subject having experienced the same event (AE preferred term) more than once during the study with a different intensity or seriousness, it will be counted only once with the worst grade and seriousness respectively.
- 4. A subject having experienced the same event (AE preferred term) more than once during the study with a different causal relationship to the study drug, it will be counted only once by considering the most-related documented degree of relationship.

#### **Events with Irregular Start or End Dates:**

Partial dates may be imputed when appropriate. Imputed dates will be used to determine Study Day.

If a partial date is reported for the start of an adverse event, a complete date will be estimated by the following algorithm:

- 1. Only the year is reported: If the subject started receiving study medication in the previous year, then January 1 will be used as the starting date of the event. If the subject started receiving study medication in the year reported, then the date of the first dose of study medication will be used as the start of the event.
- 2. The month and year is reported: If the subject started receiving study medication prior to the month and year reported, then the first day of the month will be used as the starting date




of the event. If the subject started receiving study medication during the month and year reported, then the date of the first dose of study medication will be used as the start of the event.

If a partial date is reported for the end of an adverse event and the adverse event is not continuing, a complete date will be estimated by the following algorithm:

- 1. Only the year is reported: If the subject started receiving study drug in the previous year, then the date of final study contact with the subject will be used as the end of the adverse event. If the subject started receiving study medication in the year reported, then the earlier of December 31 or the date of final study contact with the subject will be used as the end of the adverse event.
- 2. The month and year reported: The earlier of the last date of the month or the date of final contact with the subject will be used as the end of the adverse event.

The above rules are subject to logical sense (for example, imputed start date should be on or prior to imputed end date and vice-versa).

#### 6.3.4 Laboratory Data

Clinical laboratory tests on hematology, chemistry, urinalysis, and HF biomarkers will be performed according to the schedule in Section 3.6. Investigators will assess whether there are any clinically significant abnormalities and record the abnormality on medical and surgical history or adverse event forms. The lists of laboratory parameters collected are as follows:

#### Hematology:

- Hemoglobin
- Hematocrit
- Erythrocyte count (RBC)
- Leukocytes (WBC)
- Neutrophils, segmented
- Lymphocytes
- Monocytes
- Eosinophils
- Basophils
- Platelets

#### Clinical Chemistry (Serum Concentrations of):

- Sodium
- Potassium




- Total bilirubin
- Alkaline phosphatase (ALP)
- Alanine aminotransferase (ALT)
- Aspartate aminotransferase (AST)
- Blood urea nitrogen (BUN)
- Creatinine
- Calcium
- Glucose, nonfasting
- Albumin
- Chloride
- Bicarbonate
- Total Protein
- Triglycerides
- eGFR calculated with the MDRD study equation
- hsTroponin I Urinalysis:
- Specific gravity
- pH
- Protein
- Glucose
- Ketones
- Blood
- Sodium
- Chloride
- Creatinine
- Microalbuminuria HF Biomarker:
- NT-pro-BNP

#### **Conversion to the International System of Units**

All laboratory data will be stored in the database with the units in which they are originally reported. Laboratory data in summary tables and subject data listings will be presented in the International System of Units (SI units; Système International d'Unités). Laboratory data not reported in SI units will be converted to SI units before further processing or data analysis.

#### **Abnormal Values**

Based upon laboratory normal ranges, laboratory test results will be categorized according to the normal range as low, normal and high. Subjects with laboratory data outside the normal range will be listed with abnormal values flagged.


#### 6.3.5 Vital Signs

Vital signs include heart rate (beats per minute [BPM]), respiration rate, systolic and diastolic blood pressure (mmHg) and oral or tympanic temperature (°C). Vital signs will be collected at each scheduled visit.

Baseline values are those measured at last evaluation prior to the first dose of study medication.

Change from baseline to time point t, denoted Changet, will be calculated as:

Changet = Value - ValueBaseline.

#### 6.3.6 Electrocardiogram (ECG)

Baseline ECGs will be defined as the last evaluation performed prior to the first dose of study medication. Electrocardiogram results (normal versus abnormal), intervals of HR, PR, QRS, QT, and RR in msec are reported on eCRF at screening, Day 1 (Baseline), Week 1, Week 2, Week 4, and Week 6. The Fridericia corrected QT interval (QTcF) will be calculated as: QTcF = QT/(RR)<sup>1</sup>/<sub>3</sub>.

#### 6.3.7 Physical Examination

A cardiovascular physical examination, including lung auscultation and weight, will be measured at screening, Day 1 (Baseline), Week 1, Week 2, Week 4, and Week 6. Height will only be measured at the Screening Visit.

The results of the physical examination with any clinical significant abnormalities (yes/no) are reported on the eCRF.

#### 6.3.8 Pregnancy Test

All pregnancies with an estimated conception date that occurred during the AE reporting period, as defined in Section 6.3.3, must be recorded in the AE section of the eCRF. For this study, this applies to pregnancies in female subjects and in female partners of male subjects.

#### **6.3.9** Concomitant Medications/Treatments

Prior and concomitant medications will be recorded at Screening and during the study. Prior medication is defined as any medication taken before the first dose of the IMP. Concomitant




medication is defined as any medication taken during the study between the date of the first dose of IMP and the last study date of the subject. Any medications started after the last study date of the subject will not be considered concomitant medications.

All relevant information, including reason for use, dose, frequency and route, will be recorded for any medication administered or received prior and during the study.

Summaries of all concomitant therapies taken during the course of the study will be presented in tabular form using Anatomical Therapeutic Chemical 3 classification codes and preferred drug name via the World Health Organization Drug Dictionary (WHO-DD) with latest version to be specified in the Clinical Study Report.

All medications will be summarized by treatment group and sorted alphabetically by medication class and medication subclass. For the summary tables, if a subject has taken a concomitant medication more than once, the subject will be counted only once in the total.

The concomitant medication listing will be reviewed as part of the identification of protocol deviations to identify subjects who took medications which may affect the efficacy of the study drug. Medications of interest include beta blockers, ACE or ARBS, Spironolactone, diuretics (specifically furosemide), and oral long acting nitrates.

#### **Medications with Incomplete Dates:**

For medications with incomplete dates, imputation will be used to convert to a complete date. Imputed dates will be used to determine Study Day.

Partial medication start dates will be imputed as follows:

- 1. Only the year is reported: If the subject started to receive study drug in the year reported, then the date of the first dose of study drug will be used as the starting date of the medication. Otherwise, January 1 will be used as the start of the medication.
- 2. The month and year is reported: If the subject started to receive study drug during the month and year reported, then the date of first dose of study drug will be used as the starting date of the medication. Otherwise, the first day of the month will be used as the start of the medication.

Partial medication end dates will be imputed for non-ongoing medications as follows:




- 1. Only the year is reported: If the subject stopped to receive study drug in the year reported, then the date of the last dose of study drug will be used as the end date of the medication. Otherwise, December 31 will be used as the end of the medication.
- 2. The month and year is reported: If the subject stopped to receive study drug during the month and year reported, then the date of last dose of study drug will be used as the end date of the medication. Otherwise, the last day of the month will be used as the end of the medication.

The above rules are subject to logical sense (for example, imputed start date should be on or prior to imputed end date and vice-versa).

#### 7. STATISTICAL ANALYSIS

#### 7.1 General Data Handling Rules and Definitions

All data collected on case report forms will be provided in listings, except data collected only for confirmation of study entry criteria and for study administrative purposes. If any randomized subject is found to not have valid documented informed consent, the subject's data will be excluded from the report, except as necessary to document the error.

Except where specified all continuous variables will be summarized with descriptive statistics (the number of non-missing values, mean, standard deviation, median, minimum and maximum) and all categorical variables will be summarized with frequency counts and percentages, by treatment group. Unless otherwise specified, the mean and median will be displayed to one more decimal place than the original data, and standard deviation and standard error of the mean should be displayed to two more decimal place than the original data. All percentages for frequencies will be rounded to 1 decimal place.

When statistical hypothesis testing is performed, the treatment comparison will be two-sided and tested at an alpha=0.05 level of significance. Although, this provides for experiment-wise alpha at the strict 0.05 level, for the primary endpoint (LV ESV), significant results on LV EF would also be considered positive. In addition, if both endpoints are statistically significant at the 0.10 level of statistical significance, the study will similarly be considered positive. This effectively implements a Hochberg's adjustment for a primary endpoint family (of LV ESV and LV EF) at the 0.10 family-wise alpha-level.




Missing data will be maintained as missing unless specified otherwise. For variables where missing data is imputed, the analysis dataset will contain one variable with the imputed value and the original variable with missing maintained as missing.

#### 7.2 Subject Disposition

Subject disposition summaries will include the number of subjects randomized and the numbers included in the Safety, ITT, and Per-Protocol populations by treatment group for all subjects. The number and percentage of subjects who complete or discontinue from the study will be summarized by reason for discontinuation for each treatment group.

The frequency distribution of the extent of subject participation in the study (last study date – randomization date – number of days of missed doses + 1) will be provided by treatment group for all randomized subjects.

## 7.3 Demographic and Baseline Characteristics

Subject's age, gender, race, ethnicity, weight, height, BMI, and baseline characteristics, vital signs, cardiovascular physical examination results (any clinically significant abnormalities (yes, no)), and ischemic/non-ischemic status will be summarized by treatment group and for all subjects in the Safety, ITT, and Per-Protocol populations. The medical and surgical history will be listed.

#### 7.4 Efficacy Analyses

Efficacy analyses will be conducted on the ITT population, along with the Per-Protocol population for sensitivity; according to the treatment the subjects were assigned.

Since imaging may be performed after a clinic visit there will be an allowable 5 day window from the clinic visit. Any imaging that is collected more than 5 days after the clinic visit will not be included in the analysis.

#### 7.4.1 Primary Efficacy

The primary efficacy endpoint is change in LV ESV assessed by MRI at Week 4 from baseline.

Actual values and change from baseline values will be summarized by treatment group in the ITT and Per-Protocol populations. Mean change in LV ESV measurements of all three treatment groups together will be analyzed using a mixed-effect model for repeated measures (MMRM), in order to study trends in the treatment effects over 4 weeks, with the primary time point of interest




being at Week 4. The model will include treatment (4 mg elamipretide, 40 mg elamipretide, placebo), visit (week numbers), treatment-by-visit interaction, and ischemic/non-ischemic as fixed effects, baseline LV ESV and baseline LV ESV by visit interaction as covariates, and subject as a random effect. An unstructured covariance matrix will be used to model the covariance of withinpatient results. The Kenward Roger method will be used to compute the denominator degrees of freedom. All LV ESV data at Week 1 and Week 4 will be included in the MMRM model. All pairwise comparisons among treatment groups for change from baseline in LV ESV and the corresponding 2-sided 95% confidence interval (CI) will be calculated based on the MMRM model for each visit. In addition a linear contrasts (at each visit) will be constructed to test for trend over dose levels, such that differences in contrast coefficients are proportional to differences in dose level (0 mg, 4 mg and 40 mg).

The primary comparison for the primary analysis involves the comparison of 40 mg elamipretide vs. placebo at Week 4. This provides for experiment-wise alpha at the strict 0.05 alpha-level for this comparison, only.

Nevertheless, a failure of the primary comparison for the primary endpoint will not automatically be considered a "failed study" for internal decision making, where the decision will necessarily be made based on the totality of the data. Accordingly, nominal significance on key secondary endpoints (such as LV EF) or even strong trends in a preponderance of endpoints with key secondary endpoints significant at a slightly inflated alpha-level of, say, 0.10, may be considered sufficient for progression of the compound in this indication, despite an outcome not generally considered to represent "substantial evidence of effectiveness".

The normality and homogeneity of variances assumptions will be checked graphically by residual plot. If these model assumptions fail despite data transformation (e.g. log) a non-parametric approach (e.g. Kruskal-Wallis test) may be used.

#### 7.4.2 Secondary Efficacy

Secondary analyses to address the secondary objective will include comparisons in change from baseline between treatment groups for the following endpoints. The MRI endpoints will be analyzed in the same manner as the primary efficacy measures. The model will include the same terms as for the primary analysis, but will include the baseline (pre-treatment) assessment of the same endpoint. The echocardiography endpoints (except those endpoints noted below) will be analyzed with the same MMRM model as the primary endpoint, with the exception that Week 4


and Week 6 (two week post-treatment follow-up visit) will be included in the model (instead of Week 1 and Week 4). The model will include the same terms as for the primary analysis, but will include the baseline (pre-treatment) assessment of the same endpoint. Due to the high degree of measurement error associated with echocardiography measurements, only descriptive statistics will be produced for select echocardiography parameters as described below.

Secondary Endpoints Assessed by MRI:

- LVEF LV EDV LVSV
- o LVCO
- LV myocardial mass RV ESV RV EDV
- o RVEF

Secondary Endpoints Assessed by Echocardiography:

- o E/A (ratio between early and late mitral inflow velocity),
- E/e' (Ratio between early mitral inflow velocity and mitral annular early diastolic velocity)
- LA volume LV GLS

The following secondary endpoints assessed by echocardiography with descriptive statistics only:

- LV EDV LV ESV LVEF (biplane)
- o LV mass
- Mitral regurgitation severity
- Tricuspid regurgitation severity o RV fractional area change o RV systolic pressure (RVSP)

#### 7.4.3 Exploratory Efficacy

Exploratory analyses to address the exploratory objective will include comparisons in change from baseline between treatment groups for the following endpoints. hsTroponin and the log of NT-proBNP levels will be analyzed in the same manner as the primary efficacy measures, with a MMRM model. The distance walked (meters) during 6MWT and the KCCQ score only have one postbaseline assessment so they will not be analyzed as repeated measures. Instead, the change




from baseline of these two endpoints will be analyzed with an ANCOVA model. The model terms will include terms for treatment, baseline (pre-treatment) value, and ischemic/non-ischemic. Treatment difference estimates using least square means along with the 95% confidence intervals for the estimates will be presented for scheduled visits. The difference in mean change from baseline between the elamipretide treatment groups and placebo will be tested at a 2-sided significance level of 0.05.

- Distance walked (meters) during 6MWT
- Levels of NT-pro-BNP (log transformed)
- KCCO score

Additionally, the LV myocardial mass, LV stroke volume, LV cardiac output, RV end systolic volume, RV end diastolic volume, RV myocardial mass, and the RV ejection fraction, assessed by MRI, will be analyzed in the same manner as the primary efficacy measures, including comparisons in change from baseline between treatment groups.

#### 7.4.4 Efficacy Subgroup Analyses

The primary efficacy endpoint, change in LV ESV assessed by MRI at Week 4 from baseline, will be summarized by treatment group for subgroups of subjects with baseline ischemic/non-ischemic status, high versus low baseline hsTroponin, subgroups of baseline NT-pro-BNP levels. The values of the endpoint for the subgroups will also be plotted by treatment group over time for Screening, Week 1, and Week 4. The analyses and plots will be done using the ITT population.

#### 7.5 Plasma Concentration Analyses

Plasma concentration analyses will be conducted on the Safety population. Plasma samples will be analyzed for elamipretide, M1, and M2 concentrations. No formal statistical analyses will be performed.

Individual concentration time data for elamipretide will be listed, sorted by subject, and summarized for each nominal time point (as determined by nominal hour).

The plasma concentration data for elamipretide, M1, and M2 at each time point will be listed and summarized for the safety population. Descriptive statistics will include the number of observations (n), mean, standard deviation, coefficient of variation, median, minimum, maximum, geometric mean, and geometric coefficient of variation.




The plasma concentration-time profiles for individual and mean (+/-SD) plasma concentrations of elamipretide, M1, and M2 will be presented on both linear/linear and semi-logarithmic (log/linear) scales. For individual profiles, three figures will be presented with all individual profiles, one each for elamipretide, M1, and M2, superimposed on a same profile panel. For the mean linear-linear and semi-logarithmic profiles, three figures will be created with the mean concentrations of elamipretide, M1, and M2 at each nominal time-point for all subjects displayed.

#### 7.6 Safety Analyses

Except where otherwise specified, safety analyses will be performed using the safety population. Safety measurements will include AEs, clinical laboratory tests (i.e. serum chemistry, hematology, urinalysis, and hsTroponin), ECGs, physical exams and vital signs. All safety data will be summarized by treatment group. Baseline values for clinical laboratory tests, vital signs and ECGs will be defined as the last evaluation performed prior to administration of study drug.

#### 7.6.1 Extent of Exposure to Study Medication

The following study medication exposure variables as listed in Section 6.3.2 will be summarized by treatment groups.

- Study treatment exposure (days)
- Study treatment compliance (%)

Study medication dosing information will be listed by subject.

#### 7.6.2 Adverse Events

All AEs will be coded to system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA version 19.1 or newer) coding dictionary (version to be specified in the clinical study report). All reported AEs will be listed, but only treatmentemergent adverse events (TEAEs) will be summarized.

Frequency and percentage of subjects experiencing a specific adverse event will be tabulated by system organ class, preferred term, and treatment group. Summary tables will be provided for adverse events by maximum intensity, relationship to study drug, serious adverse events, and adverse events causing discontinuation of study medication.

The incidence of all TEAEs, drug relationship with TEAEs, and severity of TEAE will be summarized by treatment group and all subjects in the safety population with frequencies and




percentages. In the summary tables, subjects may be counted under multiple SOCs and PTs, but for each SOC and PT, subjects are only counted once. If a subject has the same AE on multiple occasions, the highest intensity (severe > moderate > mild) or drug relationship (probable > possibly related > unlikely related > unrelated) recorded for the event will be presented. If severity is missing, subjects will be included as Grade 3 (for severity). If drug relationship is missing, subjects will be included in related tables (i.e., considered related). Summary tables will be sorted by SOC, and then PT.

The following summaries will be presented for TEAEs:

- 1. Summary of Adverse Events by Treatment Group;
- 2. Incidence of Adverse Events by System Organ Class and Preferred Term;
- 3. Incidence of Serious Adverse Events by System Organ Class and Preferred Term;
- 4. Incidence of Adverse Events by System Organ Class, Preferred Term and Intensity;
- 5. Incidence of Study Drug Related Adverse Events by System Organ Class, Preferred Term and Intensity;
- 6. Incidence of Adverse Events by System Organ Class, Preferred Term and Relationship to Study Drug;
- 7. Incidence of Adverse Events Leading to Discontinuation of Study Drug by System Organ Class and Preferred Term

#### **7.6.3** Deaths

Summary of deaths will be provided as a listing, displaying treatment group, date of death, study day of death and reason for death.

## 7.6.4 Clinical Laboratory Evaluations

Summary tables for laboratory parameters (including hematology, chemistry, urinalysis, and hsTroponin) will include descriptive statistics for values and change from baseline for all continuous variables for each treatment group. Subjects with laboratory data outside the normal range will be listed with abnormal values flagged.

Shift tables (i.e., tables that show the number of subjects who are low, normal, or high at baseline versus each post-baseline scheduled assessment, Section 3.6) will be produced.

The number and percentage of subjects with urinalysis results outside the normal range will be presented by parameter and time point for each treatment group. Shift tables for urinalysis will




show the number of subjects who are normal/abnormal at baseline and normal/abnormal at the end of study.

Laboratory test reference ranges, flags for values outside of the normal ranges, as well as investigators assessment of these values as non-clinically or clinically significant are all displayed in subject data listings by treatment group and measurement time point for all subjects from the safety population.

#### 7.6.5 Vital Signs

Vital sign changes from baseline tables will be summarized by treatment group and visit time point. Listing of vital signs will be provided for all subjects in the safety population.

## 7.6.6 Electrocardiogram (ECG)

ECG changes from baseline tables will be summarized by treatment group and visit time point, and a subgroup table for low and high QRS interval duration. ECG results (normal versus abnormal) and an assessment of the clinical significance of any abnormalities (in the opinion of the Investigator) will be listed for individual subjects. Intervals of HR, PR, QRS, QT, and QTc will also be listed. Patients who have either an increase of >60 msec between baseline and end of treatment in their QT or an absolute QT value >500 msec at any point in time during the study will be listed separately.

#### 7.6.7 Physical Examination

The number and percentage of subjects experiencing clinically significant abnormalities (yes, no, not done) in the cardiovascular physical examination will be tabulated at every visit by treatment group and for all subjects combined. The number and percentage of subjects experiencing clinically significant abnormalities (yes, no, not done), and the weight, height, and BMI, in the physical measurements will be summarized at every visit by treatment group and for all subjects combined. Physical examinations results will be presented in individual subject data listings.

#### 7.6.8 Concomitant Medications/Treatments

The number and percentage of subjects have reported concomitant therapies during the course of the study will be tabulated by using Anatomical Therapeutic Chemical 3 classification codes and preferred drug name via the World Health Organization Drug Dictionary (WHO-DD) in latest version (version 3Q2016 WHODRUG DDE in addition to WHODRUG HD, or later), with version to be specified in the Clinical Study Report.


All medications will be summarized by treatment group and sorted alphabetically by medication class and medication subclass. For the summary tables, if a subject has taken a concomitant medication more than once, the subject will be counted only once in the total.

All prior and concomitant medication data will be presented in individual subject data listings.

#### 8. ANALYSES PERFORMED BEFORE DATABASE CLOSURE

No interim analyses are planned for this study.

#### 9. CHANGES FROM METHODS PLANNED IN THE PROTOCOL

Any changes to methods planned in this statistical analysis plan will be documented in a revision to this statistical plan prior to database lock, or identified in the clinical study report.

#### 10. STATISTICAL SOFTWARE

The statistical software to be used for generation of the tables, listings, and figures is SAS® version 9.3 or higher.

#### 11. REFERENCES

#### APPENDIX 1 DATA HANDLING RULES

| Category | Description | Data Handling Rules |
|---|---|---|
| Demographics | Age at informed consent | Age = integer ((date of informed consent signed – date of birth+1)/365.25) |
| | | For some sites (Italy and U.K.) only month and year of birth are collected, and day of birth is imputed as the 1 <sup>st</sup> of the month. |
| | | For some sites (Netherlands) only year of birth is collected, and day and month of birth are imputed as the 1 <sup>st</sup> of January. This same imputation rule will apply for all missing day of birth to the 1 <sup>st</sup> of the month, and month of birth to January. |
| Baseline | Baseline assessment | Baseline assessment is defined as last assessment prior to first dose of study medication. |
| Timing | Study Day 1 | Date subject is randomized and expected to receive the first dose of study medication. |


| Timing | Study Day | Before study day 1: study day = date of assessment – date of study day 1. |
|---|---|---|
| | | On or after study day 1: study day = date of assessment – date of study day $1 + 1$ . |
| Timing | Day 1 and Hour 0 | The date and time at first dose of study medication. |
| Timing | Time from first dose of study medication | The time from first dose of study medication = time of assessment – time of first dose of study medication. |
| Outcome<br>measures/Vita<br>1 Signs/Lab | Change from baseline | $Change_t = Value_t - Value_{Baseline}.$ |
| Exposure | Extent of study drug exposure | Extent of exposure to study medication (days) = Treatment end date – treatment start date – number of days of missed doses + 1. |

#### APPENDIX 2 SAS CODE FOR STATISTICAL ANALYSES

The following table presents the SAS code for the statistical analyses. This section will be finalized after examining the existing data and prior to the final signoff of this SAP.

| Test | Table/Figure | SAS Codes |
|---|---|---|
| MMRM with<br>baseline value as<br>covariate | Primary and secondary MRI and exploratory endpoints- requiring MMRM | proc mixed; class treatment timepoint patient; model cfb = treatment baseline timepoint baseline*timepoint treatment*timepoint ischemic / residual ddfm=kenwardroger; ** cfb is change from baseline **; repeated timepoint / type=un subject=patient; lsmeans treatment*timepoint / pdiff cl; run; |
| ANCOVA with baseline value as covariate | Secondary and Exploratory endpoints requiring ANCOVA | <pre>proc glm; class treatment; model cfb = treatment baseline baseline_MRI ischemic; **cfb is change from baseline; lsmeans treatment / cl pdiff; run;</pre> |

| Linear trend test<br>for MMRM<br>models | Primary, and secondary MRI, and exploratory endpoints-requiring MMRM | proc mixed; class treatment timepoint patient; model cfb = treatment baseline timepoint baseline*timepoint treatment*timepoint ischemic; **A contrast 'linear trend test' will involve the following coefficients to test treatment effects at each visit -0.470757 -0.342368 0.8131249; ** coefficients calculated from SAS PROC IML; ** in order of placebo, 4, 40; If treatment=3 is placebo, code treatment as 0 so placebo will go first. Coefficients are applied to estimates of treatment effect for each treatment group at each visit, which will consist of main effect and interaction terms, specific for the visit under consideration. run; |
|---|---|---|
| Linear trend test<br>for ANCOVA<br>models | Secondary and Exploratory endpoints requiring ANCOVA | proc glm; class treatment; model cfb = treatment baseline baseline_MRI ischemic; contrast 'linear trend test' treatment -0.470757 -0.342368 0.8131249; ** coefficients calculated from SAS PROC IML; ** in order of placebo, 4, 40; If treatment=3 is placebo, code treatment as 0 so placebo will go first. run; |

APPENDIX 3 REFERENCE RANGES AND CLINICALLY RELEVANT CHANGES FROM BASELINE FOR MARKED LABORATORY ABNORMALITIES

Not applicable.




## APPENDIX 4 MOCKUP TABLES, LISTINGS, AND GRAPHS (TLGS)

Mockup tables, listings, and graphs are presented in a separate document.




# SPECIFICATION OF END OF TEXT STANDARD OUTPUT TABLES, LISTINGS, AND FIGURES (TLFs)

**Trial Sponsor:** Stealth BioTherapeutics, Inc.

**Protocol Number:** SPIHF-201 **IND Number:** N/A **EUDRACT Number:** 2014-005724-10

**Investigational Drug:** Elamipretide<sup>TM</sup> (MTP-131)

**Indication:** Heart Failure with reduced Ejection Fraction

(HFrEF)

**Dosage Form/Strength:** Elamipretide<sup>TM</sup> (MTP-131) 40 mg/1 mL of

sterile solution for subcutaneous injection with doses of 4 mg or 40 mg administered

as a once daily SC injection

**Protocol Title:** A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Effects of Multiple Subcutaneous Injections of Elamipretide on Left Ventricular Function in Subjects with Stable Heart Failure with Reduced Ejection Fraction

\_\_\_\_\_\_

The information in this document is confidential and is proprietary to Stealth Biotherapeutics. It is understood that information in this document shall not be disclosed to any third party, in any form, without prior written consent of an authorized officer of Stealth Biotherapeutics.

#### CHANGE LOG FOR CHANGES MADE AFTER THE INITIAL APPROVAL


| Revision | Section(s) | Brief Description of Revision(s) or<br>Reason(s) for Revision | Modifications Reviewed and Approved by* |
|---|---|---|---|
| Date** | Modified | | Sponsor, Everest |

<sup>\*</sup> Provide person's initial and last name. \*\* Update the Last Revision Dates

on the cover page and the document header.


#### General Instructions for End-of-Text TFLs

Following are the specifications for end-of-text standard tables, figures and listings (TFLs).

#### **Header**

The following header should appear at the very top of each page of a table, a figure, or a listing (TFL):

Stealth Protocol SPIBioTherapeuticsHF-201 Inc. ElamipretidePage n of N  $^{\text{TM}}$  (MTP-131 for SC Injection)

#### Footer

The following footer should appear at the bottom of each page of a TFL generated in SAS:

Program: /sasdir/pgname.sas Version 2014-01-25 13:37

where: PGNAME = SAS program name. Version will be replaced by "Draft" or "Final".

#### Title

At least three (3) lines should be reserved for the whole title. The first line is for the TFL number (i.e., title index #); the second line is for the actual title (title); and the third line is reserved for the analysis population descriptor (population). All titles should be centered, as shown in the following example:

Table 1.1
Demographics
Safety Population

#### Footnotes

In general, a footnote serves as a brief explanation/clarification/definition/concept of a flag symbol or a character, an abbreviation, a terminology, etc., that appears in, or related directly to the displayed content of a TFL. Detailed/technical elaboration of, for example, a mathematical/statistical formula, a statistical term/test, or an algorithm for deriving a parameter value, should be addressed in the text of the statistical analysis plan (SAP).

All footnotes should follow immediately after a horizontal solid line. There should be one and only one space between the last footnote and the footer.

When an abbreviation (e.g., TEAE, SAE, etc.) appears for the first time in the entire set of TFLs for a study, a footnote should be provided at least once; it is up to the Study Biostatistician, Scientist, and Study Programmer to decide whether there is a need to repeat the same footnote for the rest of TFLs (if applicable).

Each line of a complete footnote should end with a period. When a footnote needs more than 1 line, one (1) period is needed.




#### Footnotes should be in the format shown in the following example:

<abbreviations> <notes>
[a]
[b]
[c]
Source: Listings 2.1.1, 2.1.2, 2.3

#### Page Layout

All output should be in landscape orientation.

All efforts should be made to present all treatment groups in one page.

The Scientist and Study Biostatistician will pre-determine the order for the display of the treatment groups.

#### Page Format

There should be a solid line at the top of the tables and listings just below the title.

There should be a solid line just below the column headings that runs completely across the width of the tables and listings.

There should be a solid line at the bottom of the tables and listings just above the footnote(s) on every page.

#### Font

The default font to be used in the actual study tables/listings should be Courier New 8 point which is approximately equivalent to the acceptable font size of Times New Roman 9-10 in accordance with the FDA's guidance on Electronic Common Technical Document Specification.

#### Descriptive Statistics

By default, descriptive statistics in this template covers: n, mean, median, standard deviation (SD), minimum (min), and maximum (max). Unless otherwise specified in the actual table shells, the mean and median should be displayed to one more decimal place than the original data, and standard deviation and standard error of the mean should be displayed to two more decimal place than the original data.

#### Rounding for Percentage

All percentages will be rounded to 1 decimal place in all TFLs. P-values will be presented with 4 decimal places.

#### Alignment of Decimals

It is recommended that all the decimal places be aligned in summary tables, as shown in the following example:




#### Decimal Align

n xxx

Mean xx.xx

SD xx.xxx

Median xx.xx

Min, Max xx.x, xx.x

When numbers with decimal points are included in brackets (e.g., percentages), the brackets should be aligned to the right and then padded to allow for all possible percentages and then the left brackets will also be aligned. For example:

Brackets Align (99.9%) (xx.x%) (9.9%) (x.x%)

It is recommended that all column entries in a summary tables and listings are aligned to the center. Columns for text fields are all left justified. Columns with whole numbers are all right justified. For graphs, the lines are distinguishable and that the symbols for each line are appropriate. Legend is consistent across output for treatment names and abbreviations.

#### Use of N Versus n

N = total number of subjects in the defined analysis set. n

= total number of subjects in the specific category.

If N is specified in the column heading then any reference to the number of subjects in the body should be small n, as shown in the following example:

| Demographic Parameter | <pre>Treatment Group A (N = xxx)</pre> | Treatment Group B (N = xxx) | Total (N = xxx) |
|---|---|---|---|
| | XX | XX | XX |
| Age (years) n | XX.X | XX.X | XX.X |
| Mean SD | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |

#### A Note for Subject Data Listings

Observed Dates/AE Severity/Relationship to investigational product are used in subject data listings.

Observed values or raw assessment scores are used in data listings along with their derived values used in analyses, e.g., raw assessment scores and derived total scores.

#### TABLE OF CONTENTS FOR TABLES, FIGURES AND LISTINGS

CONFIDENTIAL

Statistical Analysis Plan Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

| 1. | SUBJECT DISPOSITION | 19 |
|-----|-------------------------------------------------------------|----|
| | Table 1.1 | 19 |
| | Subject Disposition | |
| | All Randomized Subjects | |
| | Table 1.2 | 20 |
| | Extent of Participation in the Study | |
| | All Randomized Subjects | |
| 2. | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 21 |
| | Table 2.1a | 21 |
| | Demographic and Non-Imaging Baseline Characteristics | |
| | Safety Population | |
| | Table 2.1b | 25 |
| | Baseline Characteristics from MRI | |
| | Safety Population | |
| | Table 2.1c | 27 |
| | Baseline Characteristics from Echocardiography Safety | |
| | Population | |
| | Table 2.2a | 29 |
| | Demographic and Non-Imaging Baseline Characteristics ITT | |
| | Population | |
| | Table 2.2b | 29 |
| | Baseline Characteristics from MRI ITT | |
| | Population | |
| | Table 2.2c | 29 |
| | Baseline Characteristics from Echocardiography ITT | |
| | Population | |
| | Table 2.3a | 29 |
| | Demographic and Non-Imaging Baseline Characteristics | 29 |
| | Per-Protocol Population | |
| | Table 2.3b | 29 |
| | Baseline Characteristics from MRI | 2) |
| | Per-Protocol Population | |
| | Table 2.3c | 29 |
| | Baseline Characteristics from Echocardiography Per-Protocol | 2) |
| | Population | |
| 3. | EFFICACY ANALYSIS | 30 |
| 3.1 | EFFICACY ANALYSIS | |
| 5.1 | | |
| | Table 3.1 | 31 |
| | Assessed by MRI | |
| | • | |
| | ITT Population Table 3.2 | 32 |
| | I auic J.Z | |



| Summary of Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), |
|---|
| Assessed by MRI |
| Per-Protocol Population |
| Table 3.3 |
| Summary of Change From Baseline in Left Ventricular Ejection Fraction (LVEF), Assessed by |
| MRI |
| ITT Population |
| Table 3.4 |
| Summary of Change From Baseline in Left Ventricular Ejection Fraction (LVEF), Assessed by |
| MRI |
| Per-Protocol Population |
| Table 3.5 |
| Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV), |
| Assessed by MRI ITT |
| Population |
| Table 3.6 |
| Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV), |
| Assessed by MRI |
| Per-Protocol Population |
| Table 3.7 |
| Summary of Change From Baseline in Left Ventricular Stroke Volume (LVSV), Assessed by |
| MRI |
| ITT Population |
| Table 3.8 |
| Summary of Change From Baseline in Left Ventricular Stroke Volume (LVSV), Assessed by |
| MRI |
| Per-Protocol Population |
| Table 3.9 |
| Summary of Change From Baseline in Left Ventricular Cardiac Output (LVCO), Assessed by |
| MRI |
| ITT Population |
| Table 3.10 |
| Summary of Change From Baseline in Left Ventricular Cardiac Output (LVCO), Assessed by |
| MRI |
| Per-Protocol Population |
| Table 3.11 |
| Summary of Change From Baseline in Left Ventricular Myocardial Mass (LV Mass), |
| Assessed by MRI ITT |
| Population |
| Table 3.12 |
| Summary of Change From Baseline in Left Ventricular Myocardial Mass (LV Mass), |
| Assessed by MRI |



| Per-Protocol Population | |
|---|---|
| Table 3.13 | 35 |
| Summary of Change From Baseline in Right Ventricular End Systolic Volume (RV ESV), | |
| Assessed by MRI ITT | |
| Population | |
| Table 3.14 | 35 |
| Summary of Change From Baseline in Right Ventricular End Systolic Volume (RV ESV), | |
| Assessed by MRI | |
| Per-Protocol Population | |
| Table 3.15 | 35 |
| Summary of Change From Baseline in Right Ventricular End Diastolic Volume (RV EDV), | |
| Assessed by MRI ITT | |
| Population | |
| Table 3.16 | 35 |
| Summary of Change From Baseline in Right Ventricular End Diastolic Volume (RV EDV), | |
| Assessed by MRI | |
| Per-Protocol Population | |
| Table 3.17 | 36 |
| Summary of Change From Baseline in Right Ventricular Ejection Fraction (RVEF), | |
| Assessed by MRI ITT | |
| Population | |
| Table 3.18 | 36 |
| Summary of Change From Baseline in Right Ventricular Ejection Fraction (RVEF), | |
| Assessed by MRI | |
| Per-Protocol Population | |
| Table 3.19 | 36 |
| Summary of Change From Baseline in E/A (Ratio Between Early And Late Mitral Inflow | |
| Velocity), Assessed by Echocardiography ITT | |
| Population | |
| Table 3.20 | 36 |
| Summary of Change From Baseline in E/A (Ratio Between Early And Late Mitral Inflow | |
| Velocity), Assessed by Echocardiography | |
| Per-Protocol Population | |
| Table 3.21 | 37 |
| Summary of Change From Baseline in E/e' (Ratio Between Early Mitral Inflow Velocity and | |
| Mitral Annular Early Diastolic Velocity), Assessed by Echocardiography ITT Population | |
| Table 3.22 | 37 |
| Summary of Change From Baseline in E/e' (Ratio Between Early Mitral Inflow Velocity and | |
| Mitral Annular Early Diastolic Velocity), Assessed by Echocardiography | |
| Per-Protocol Population | |
| Table 3.23 | 37 |



| Summary of Change From Baseline in Left Atrial Volume, Assessed by Echocardiography ITT | Γ |
|---|---|
| Population | |
| Table 3.24 | |
| Summary of Change From Baseline in Left Atrial Volume, Assessed by Echocardiography Protocol Population | Per- |
| Table 3.25 | . 38 |
| Summary of Change From Baseline in Left Ventricular Global Longitudinal Strain,<br>Assessed by Echocardiography ITT<br>Population | |
| Table 3.26 | 20 |
| Summary of Change From Baseline in Left Ventricular Global Longitudinal Strain, | . 38 |
| Assessed by Echocardiography | |
| Per-Protocol Population | |
| Table 3.27 | . 39 |
| Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV),<br>Assessed by Echocardiography ITT | |
| Population | |
| Table 3.28 | . 40 |
| Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV), | |
| Assessed by Echocardiography | |
| Per-Protocol Population | |
| Table 3.29 | . 40 |
| Summary of Change From Baseline in Left Ventricular End Systolic Volume (LV ESV),<br>Assessed by Echocardiography ITT | |
| Population | |
| Table 3.30 | . 40 |
| Summary of Change From Baseline in Left Ventricular End Systolic Volume (LV ESV),<br>Assessed by Echocardiography | |
| Per-Protocol Population | |
| Table 3.31 | . 40 |
| Summary of Change From Baseline in Biplane Ejection Fraction (EF), Assessed by Echocardiography ITT | |
| Population | |
| Table 3.32 | 41 |
| Summary of Change From Baseline in Biplane Ejection Fraction (EF), Assessed by | |
| Echocardiography | |
| Per-Protocol Population | |
| Table 3.33 | 41 |
| Summary of Change From Baseline in Left Ventricular Mass, Assessed by | |
| Echocardiography ITT | |
| Population Population | |
| Table 3 34 | 41 |



| Summary of Change From Baseline in Left Ventricular Mass, Assessed by | |
|---|---|
| Echocardiography | |
| Per-Protocol Population | |
| Table 3.35 | 41 |
| Summary of Change From Baseline in Mitral Regurgitation Severity, Assessed by | |
| Echocardiography | |
| ITT Population | |
| Table 3.36 | 41 |
| Summary of Change From Baseline in Mitral Regurgitation Severity, Assessed by | |
| Echocardiography | |
| Per-Protocol Population | |
| Table 3.37 | 41 |
| Summary of Change From Baseline in Tricuspid Regurgitation Severity, Assessed by | |
| Echocardiography ITT | |
| Population | |
| Table 3.38 | 42 |
| Summary of Change From Baseline in Tricuspid Regurgitation Severity, Assesse | |
| Echocardiography | |
| Per-Protocol Population | |
| Table 3.39 | 42 |
| Summary of Change From Baseline in Right Ventricular Fractional Area Change, Assessed | |
| by Echocardiography ITT Population | |
| Table 3.40 | 42 |
| Summary of Change From Baseline in Right Ventricular Fractional Area Change, Assessed | |
| by Echocardiography Per-Protocol Population | |
| Table 3.41 | 42 |
| Summary of Change From Baseline in Right Ventricular Systolic Pressure (RVSP), | |
| Assessed by Echocardiography ITT | |
| Population | |
| Table 3.42 | 42 |
| Summary of Change From Baseline in Right Ventricular Systolic Pressure (RVSP), | |
| Assessed by Echocardiography | |
| Per-Protocol Population | |
| Table 3.43 | 42 |
| Summary of Change From Baseline in Distance Walked (meters) During 6-minute Walking | |
| Test (6MWT) | |
| ITT Population | |
| Table 3.44 | |
| Summary of Change From Baseline in Distance Walked (meters) During 6-minute Walking T | est |
| (6MWT) | |
| Per-Protocol Population | |
| Table 3 45 | 43 |

Statistical Analysis Plan Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

| | Summary of Change From Baseline in Levels of NT-pro-BNP ITT | |
|---|---|---|
| | Population | |
| | Table 3.46 | 44 |
| | Summary of Change From Baseline in Levels of NT-pro-BNP | |
| | Per-Protocol Population | |
| | Table 3.47 | 44 |
| | Summary of Change From Baseline in Levels of hsTroponin | |
| | ITT Population | |
| | Table 3.48 | 44 |
| | Summary of Change From Baseline in Levels of hsTroponin | |
| | Per-Protocol Population | |
| | Table 3.49 | 45 |
| | Summary of Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score ITT Population | |
| | Table 3.50 | 45 |
| | Summary of Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) | |
| | Overall Summary Score | |
| | Per-Protocol Population | |
| 4. | PLASMA CONCENTRATION ANALYSIS | 46 |
| | Table 4.1 | 46 |
| | Summary of Plasma Concentrations of Elamipretide and Metabolites (M1, M2) by Time | |
| | Point | |
| | Safety Population | |
| 5. | EXTENT OF EXPOSURE TO STUDY MEDICATION | 48 |
| | Table 5.1 | 48 |
| | Extent of Exposure to Study Medication by Treatment Group Safety | |
| | Population | |
| 6. | ADVERSE EVENTS | 49 |
| | Table 6.1 | 49 |
| | Overall Summary of Treatment-Emergent Adverse Events by Treatment Group Safety | |
| | Population | |
| | Table 6.2 | 50 |
| | Incidence of Treatment-Emergent Adverse Events by System Organ Class and Preferred | |
| | Term | |
| | Safety Population | |
| | Table 6.3 | 51 |
| | Incidence of Treatment-Emergent Serious Adverse Events by System Organ Class and | |
| | Preferred Term | |
| | Safety Population | |
| | Table 6.4 | 52 |
| | Incidence of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Intensity Safety Population | |

| | Table 6.5 | |
|---|---|---|
| | Incidence of Study Treatment Related Adverse Events by System Organ Class, Preferred T | Term, |
| | and Intensity | |
| | Safety Population | |
| | Table 6.6 | |
| | Incidence of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term Relationship to Study Drug | , and |
| | Safety Population | |
| | Table 6.7 | 55 |
| | Incidence of Treatment-Emergent Adverse Events Leading to Discontinuation of Study<br>Drug by System Organ Class and Preferred Term | |
| | Safety Population | |
| | Table 6.8 | 56 |
| | Deaths | |
| | Safety Population | |
| 7. | CLINICAL LABORATORY EVALUATIONS | 57 |
| | Table 7.1a | 57 |
| | Change From Baseline in Hematology Parameters by Visit | |
| | Safety Population | |
| | Table 7.1b | 59 |
| | Shift Table of Hematology Parameters From Baseline to Post Baseline Visits Safety | |
| | Population | |
| | Table 7.2a | 60 |
| | Change From Baseline in Blood Chemistry Parameters by Visit | |
| | Safety Population | |
| | Table 7.2b | 60 |
| | Shift Table of Blood Chemistry Parameters From Baseline to Post Baseline Visits Safety | |
| | Population | |
| | Table 7.3a | 60 |
| | Change From Baseline in Urinalysis Parameters by Visit Safety | |
| | Population | |
| | Table 7.3b | 60 |
| | Shift Table of Urinalysis Parameters From Baseline to Post Baseline Visits Safety | |
| | Population | |
| | Table 7. 4a | 61 |
| | Change From Baseline in Levels of hsTroponin by Visit Safety | |
| | Population | |
| 8. | ELECTROCARDIOGRAM EVALUATIONS | 62 |
| 0. | Table 8.1 | |
| | Change From Baseline in Electrocardiogram (ECG) Parameters by Visit Safety Population | 02 |

| 9. | VITAL SIGNS | 64 |
|---|---|---|
| | Table 9.1 | 64 |
| | Change From Baseline in Vital Signs | |
| | Safety Population | |
| 10. | PHYSICAL EXAMINATION | 66 |
| | Table 10.1 | 66 |
| | Cardiovascular Physical Examination Results by Visit | |
| | Safety Population | |
| | Table 10.2 | 67 |
| | Physical Measurement Results by Visit | |
| | Safety Population | |
| 11. | CONCOMITANT MEDICATIONS/TREATMENTS | 70 |
| | Table 11.1 | 70 |
| | Concomitant Medications by ATC and Preferred Drug Name Safety | |
| | Population | |
| LIST | TINGS | 71 |
| LIST | TINGS – SUBJECT DISPOSITION, DEMOGRAPHICS, AND BASELINE | |
| | CHARACTERISTICS | 71 |
| | Listing 1.1 | 72 |
| | Study Completion or Early Discontinuation Status | |
| | All Randomized Subjects | |
| | Listing 1.2 | 73 |
| | Violations of Inclusion/Exclusion Criteria | |
| | All Subjects | |
| | Listing 1.3 | 74 |
| | Randomization Status | |
| | All Subjects | |
| | Listing 1.4 | 75 |
| | Demographic Information | |
| | All Randomized Subjects | |
| | Listing 1.5 | 76 |
| | Medical and Surgical History | |
| | All Randomized Subjects | |
| LIST | TINGS – EFFICACY | 77 |
| | Listing 2.1 | 77 |
| | Cardiac MRI Assessments – Actual and Change from Baseline Values ITT | |
| | Population | |
| | Listing 2.2 | 79 |
| | Echocardiography Assessments- Actual and Change from Baseline Values ITT | |
| | Population | |
| | Listing 2.3 | 81 |

Statistical Analysis Plan Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

| Exploratory Assessments – Actual and Change from Baseline Values ITT | |
|-----------------------------------------------------------------------|-----|
| Population | 02 |
| Listing 2.4.1 | 82 |
| Six-Minute Walk Test – Part I ITT | |
| Population | 0.2 |
| Listing 2.4.2 | 83 |
| Six-Minute Walk Test – Part II ITT | |
| Population | |
| Listing 2.5.1 | 84 |
| Kansas City Cardiomyopathy Questionnaire – Page 1 ITT | |
| Population | |
| Listing 2.5.2 | 85 |
| ITT Population | |
| Listing 2.5.3 | 86 |
| Kansas City Cardiomyopathy Questionnaire – Page 3 ITT | |
| Population | |
| Listing 2.5.4 | 87 |
| Kansas City Cardiomyopathy Questionnaire – Page 4 ITT | |
| Population | |
| Listing 2.5.5 | 88 |
| Kansas City Cardiomyopathy Questionnaire – Summary Scores ITT | |
| Population | |
| LISTINGS – STUDY DRUG AND PRIOR/CONCOMITANT MEDICATIONS | |
| Listing 3.1 | 89 |
| Study Drug Injection Records | |
| Safety Population | |
| Listing 3.2 | 90 |
| Prior and Concomitant Medications by Subject Safety | |
| Population | |
| LISTINGS – PLASMA CONCENTRATION | 91 |
| Listing 4.1 | 91 |
| Plasma Concentrations of Elamipretide and Metabolites (M1, M2) Safety | |
| Population | |
| LISTINGS – ADVERSE EVENTS | 92 |
| Listing 5.1 | 92 |
| Adverse Events | |
| Safety Population | |
| Listing 5.2 | 93 |
| Serious Adverse Events Safety | |
| Population | |
| Listing 5.3 | 94 |
| <del>-</del> | |

Statistical Analysis Plan Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

| Adverse Events Leading to Discontinuation of Study Drug Safety | |
|---|---|
| Population | |
| LISTINGS – LABORATORY DATA | 95 |
| Listing 6.1 | 95 |
| Hematology Results by Subject and Visit | |
| Safety Population | |
| Listing 6.2 | 96 |
| Blood Chemistry Results by Subject and Visit | |
| Safety Population | |
| Listing 6.3 | 96 |
| Urinalysis Results by Subject and Visit | |
| Safety Population | |
| Listing 6.4 | 96 |
| Levels of hsTroponin by Subject and Visit Safety | |
| Population | |
| LISTINGS – OTHER SAFETY DATA | 97 |
| Listing 7.1 | 97 |
| Vital Signs by Subject and Visit | |
| Safety Population | |
| Listing 7.2a | 98 |
| Electrocardiogram (ECG) by Subject and Visit | |
| Safety Population | |
| Listing 7.2b | 98 |
| Electrocardiogram (ECG) by Subject and Visit with QRS Duration of <= 110 msec Saf | ety |
| Population | |
| Listing 7.2c | 98 |
| Electrocardiogram (ECG) by Subject and Visit with QRS Duration of >110 msec Safet | y |
| Population | |
| Listing 7.3 | 99 |
| Electrocardiogram (ECG) by Subject and Visit | |
| Subjects with Either an Increase of >60 msec Between Baseline and End of Treatment is | n |
| Their QT or QTcF or an Absolute QT or QTcF value >500 msec at Any Point in Time | During |
| the Study | |
| Safety Population | |
| Listing 7.4 | |
| Cardiovascular Physical Examination and Physical Measurements by Subject and Visit | Safety |
| Population | |
| Listing 7.5 | 101 |
| Injection Site Reaction (Nurse/Investigator Assessment) | |
| Safety Population | |
| Listing 7.6 | 102 |



| | Injection Site Reaction Self-Assessment Questionnaire Safety | |
|---|---|---|
| | Population | |
| | Listing 7.7 | 103 |
| | Comments | |
| | All Subjects | |
| FIGUR | RES | 104 |
| | Figure 1a | 104 |
| | Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Elamipretide 4 mg Group (By Subject) ITT Population | |
| | Figure 1b | 105 |
| | Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Elamipretide 4 mg Group (By Subject) | |
| | Per-Protocol Population | |
| | Figure 1c | 105 |
| | Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by | |
| | MRI, for Elamipretide 40 mg Group (By Subject) | |
| | ITT Population | |
| | Figure 1d | 105 |
| | Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by | |
| | MRI, for Elamipretide 40 mg Group (By Subject) | |
| | Per-Protocol Population | |
| | Figure 1e | 105 |
| | Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Placebo Group (By Subject) ITT | |
| | Population | |
| | Figure 1f | 105 |
| | Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI | , |
| | for Placebo Group (By Subject) | |
| | Per-Protocol Population | |
| | Figure 1g | 105 |
| | LS Mean Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), | |
| | Assessed by MRI, (By Treatment Group) ITT | |
| | Population | |
| | Figure 1h | 105 |
| | LS Mean Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assesse<br>by MRI, (By Treatment Group) | d |
| | Per-Protocol Population | |

Statistical Analysis Plan Protocol No. SPIHF-201 Last Revision Date: 04 DECEMBER 2017

| Figure 2a to Figure 2h (LVEF assessed by MRI) | 106 |
|---|---|
| Figure 3a to Figure 2h (LV EDV assessed by MRI) | |
| Figure 4a to Figure 4h (LVSV assessed by MRI) | |
| Figure 5a to Figure 5h (LVCO assessed by MRI) | |
| Figure 6a to Figure 6h (LV Myocardial Mass assessed by MRI) | |
| Figure 7a to Figure 7h (RV ESV assessed by MRI) | |
| Figure 8a to Figure 8h (RV EDV assessed by MRI) | |
| Figure 9a to Figure 9h (RVEF assessed by MRI) | |
| Figure 10a to Figure 10h (E/A assessed by Echocardiography) | |
| Figure 11a to Figure 11h (E/e' assessed by Echocardiography) | |
| Figure 12a to Figure 12h (LA Volume assessed by Echocardiography) | |
| Figure 13a to Figure 13h (LV GLS assessed by Echocardiography) | |
| Figure 14a to Figure 14f (LV EDV assessed by Echocardiography) | |
| Figure 15a to Figure 15f (LV ESV assessed by Echocardiography) | |
| Figure 16a to Figure 16f (LVEF Biplane assessed by Echocardiography) | |
| Figure 17a to Figure 17f (LV Mass assessed by Echocardiography) | |
| Figure 18a to Figure 18f (Mitral Regurgitation Severity assessed by Echocardiography) | |
| Figure 19a to Figure 19f (Tricuspid Regurgitation Severity assessed by Echocardiography) | 106 |
| Figure 20a to Figure 20f (RV fractional area change assessed by Echocardiography) | 106 |
| Figure 21a to Figure 21f (RV systolic pressure assessed by Echocardiography) | 106 |
| Figure 22a to Figure 22h (6MWT) | 106 |
| Figure 23a to Figure 23f (NT-pro-BNP) | 106 |
| Figure 24a to Figure 24h (Log10 NT-pro-BNP) | 107 |
| Figure 25a to Figure 25h (hs Troponin) | 107 |
| Figure 26a to Figure 26h (KCCQ) | 107 |
| Figure 27a | 108 |
| Mean Plasma Concentration-Time Profile of Elamipretide (Linear Scale) | |
| Safety Population | |
| Figure 27b | 109 |
| Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M1 (Linear Scale) S | afety |
| Population | |
| Figure 27c | 109 |
| Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M2 (Linear Scale) S | afety |
| Population | |
| Figure 27d | 110 |
| Log Mean Plasma Concentration-Time Profile of Elamipretide (Semi-logarithmic Scale) S | afety |
| Population | |
| Figure 27e | 110 |
| Log Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M1 | |
| (Semilogarithmic Scale) Safety Population | |
| Figure 27f | 110 |



| Log Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M2 |
|---|
| (Semilogarithmic Scale) Safety Population |
| Figure 27g |
| Individual Plasma Concentration-Time Profile of Elamipretide (Linear Scale) Safety |
| Population |
| Figure 27h |
| Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M1 (Linear |
| Scale) |
| Safety Population |
| Figure 27i |
| Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M2 (Linear |
| Scale) |
| Safety Population |
| Figure 27j |
| Individual Plasma Concentration-Time Profile of Elamipretide (Semi-logarithmic Scale) Safety |
| Population |
| Figure 27k |
| Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M1 |
| (Semilogarithmic Scale) Safety Population |
| Figure 271 |
| Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M2 |
| (Semilogarithmic Scale) Safety Population |
| Figure 28a |
| QTc for Subjects with a QTc value >500 msec at Any Point in Time During the Study (By |
| Subject) |
| Safety Population |

#### 1. SUBJECT DISPOSITION

Table 1.1 Subject Disposition All Randomized Subjects

| | Elamipretide 4 mg<br>(N=xx) | Elamipretide 40 mg (N=xx) | Placebo<br>(N=xx) | All Subjects (N=xx) |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n_(%) |
| Subjects Randomized Safety Population [a] | ( xx.x%)<br>( xx.x%) | ( xx.x%)<br>( xx.x%) | ( xx.x%)<br>( xx.x%) | ( xx.x%)<br>( xx.x%) |
| ITT Population [b] | XX | XX | XX | XX |
| Per-Protocol Population [c] | XX ( XX.X%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Treated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | XX | xx | xx | XX |
| Completed Study | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Early Discontinuation from the Study Primary Reason for Discontinuation Adverse | XX ( XX.X%) | xx (xx.x%) | XX ( XX.X%) | XX ( XX.X%) |
| Event Subject Withdrawal of Consent Sponsor Decision Investigator Decision Pregnancy Subject Lost to Follow-up | xx<br>xx ( xx.x%) | xx<br>xx ( xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>( xx.x%) |

<sup>% = 100\*</sup>n/N, where n = number of subjects in the specific row category and N = number of subjects in the column category.

Table 1.2
Extent of Participation in the Study
All Randomized Subjects

Report generated by program: /sasdir/xxxx.sas

<sup>[</sup>a] Safety Population = all subjects who received at least 1 dose of the investigational medicinal product (IMP), summarized according to the treatment received.

<sup>[</sup>b] ITT Population = all subjects who were randomized and receive at least 1 dose of IMP, summarized according to the treatment group to which the subjects were randomized

<sup>[</sup>c] Per-Protocol Population = all randomized subjects receiving at least one dose of the IMP without major protocol violations/deviations, summarized according to the treatment group to which the subjects were randomized. Source: Listing 1.1

| | Elamipretide 4 mg | Elamipretide 40 mg | Placebo | All Subjects |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | | xx xx<br>(xx.x%) | | xx xx<br>(xx.x%) |
| | | XX | | XX XX |
| whent of Darticipation in the study [a] | | (xx.x%) | | (xx.x%) |
| xtent of Participation in the study [a] | | XX | | XX |
| Treatment Period | | (xx.x%) | | (xx.x%) |
| n<br>. – . | xx xx | XX | XX XX | XX |
| 1-5 days | (xx.x%) xx | (xx.x%) | (xx.x%) xx | (xx.x%) |
| 6-10 days | (XX.X%) XX | XX | (xx.x%) xx | XX |
| 11-15 days | (xx.x%) xx | (xx.x%) | (xx.x%) xx | (xx.x%) |
| 16-20 days | (xx.x%) xx | XX | (xx.x%) xx | XX |
| 21-25 days | (xx.x%) xx | (xx.x%) | (xx.x%) xx | (xx.x%) |
| 26-28 days | (xx.x%) xx | XX | (xx.x%) xx | XX |
| >28 days | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| <del>-</del> | , , | , | , | , |
| Mean | XX.X | XX.X | XX.X | XX.X |
| D | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x xx, | XX.X XX, | xx.x xx, | xx.x xx, |
| Min, Max | XX | XX | XX | XX |
| , | AA | AA | AA | ** |
| | xx xx | xx xx | xx xx | xx xx |
| | (xx.x%) xx | (xx.x%) | (xx.x%) xx | (xx.x%) |
| Follow-up Period | (xx.x%) xx | xx | (xx.x%) xx | XX |
| n | (xx.x%) xx | (xx.x%) | (xx.x%) xx | (xx.x%) |
| 1-5 days after last dose | (xx.x%) | xx | (xx.x%) | xx |
| 6-10 days after last dose | | (xx.x%) | | (xx.x%) |
| 11-14 days after last dose | | XX | | XX |
| >14 days after last dose | | (xx.x%) | | (xx.x%) |

<sup>[</sup>a] Extent of Participation in the Study = Treatment Period: last treatment date - randomization date + 1. Follow-up Period: last study date - last treatment date + 1.

Source: Listing 1.1

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY

Draft Version 

#### 2. DEMOGRAPHIC AND BASELINE CHARACTERISTICS

Table 2.1a

Demographic and Non-Imaging Baseline Characteristics Safety

Population

| Elamipretide 4 m | g Elamipretide 40 mg | Placebo | All Subjects |
|------------------|----------------------|-----------|--------------|
| - <u>-</u> | · · · | | _ |
| (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| (14 2323) | (11 2121) | (14 2323) | (17 2121) |

| | Elamipretide<br>(N=xx) | 4 mg Eramipretide 40 (N=xx) | (N=xx) | (N=xx) |
|---|---|---|---|---|
| | XX<br>Elaminretide | xx 4 mg Elamipretide 40 | mq Placebo | xx<br>All Subjects |
| | хх, | XX, | xx, | XX, |
| | XX.X | XX . X | XX.X | XX . X |
| | XX.XX | XX . XX | XX.XX | XX.XX |
| | XX.X | XX.X | XX.X | XX.X |
| | | | XX | XX |
| | (xx.x%)<br>xx | (xx.x%)<br>xx | (xx.x%) | (xx.x%) |
| Min, Max | XX (VV V%) | (VV V%) | XX | XX |
| Median | | | (xx.x%) | |
| Mean SD | xx<br>(xx.x%) | xx<br>(xx.x%) | XX | xx<br>(xx.x%) |
| aseline Weight (kg) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| | XX | XX (**** ****) | XX ( | XX ( |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Unknown | XX XX | XX XX | XX XX | XX XX |
| Not reported | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Not Hispanic or Latino | XX | XX | XX | XX |
| Hispanic or Latino | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| | XX | XX | XX | XX |
| thnicity | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Unknown | XX | XX | XX | XX |
| Other | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Native Hawaiian or other Pacific Islander | XX | xx | XX | XX |
| American Indian or Alaska Native | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Asian | XX | xx | XX | XX |
| Black or African American | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| White | XX | XX | XX | XX |
| pri. I u . | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Race | XX XX | XX XX | XX XX | XX XX |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Female | XX | XX | XX | XX |
| n<br>Male | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Gender | XX XX | XX XX | XX XX | XX XX |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| ≥ 65 | XX | xx | XX | XX |
| < 65 | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| l | xx xx | xx xx | xx xx | xx xx |
| age (years) | xx | xx | XX | xx |
| Min, Max | xx, | xx, | xx, | xx, |
| Median | xx.x | XX.X | XX.X | XX.X |
| D | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| age (years) | XX | XX | XX | XX |

Draft YYYY

Report generated by program: /sasdir/xxxx.sas

-MM-DD HH:MM

| | XX | XX | XX | XX |
|---|---|---|---|---|
| | XX.X | XX.X | XX.X | xx.x |
| Baseline Height (cm) | xx.xx | xx.xx | xx.xx | xx.xx |
| n Mean SD | XX.X | XX.X | XX.X | xx.x |
| Median | xx, | XX, | xx, | XX, |
| Min, Max | XX | XX | XX | XX |
| | XX | XX | XX | XX |
| Body Mass Index (kg/m²) | XX.X | XX.X | XX.X | XX.X |
| Baseline | XX.XX | xx.xx | XX.XX | xx.xx |
| n Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX, | xx, | XX, | xx, |
| Median | XX | XX | XX | XX |
| Min, Max | XX | XX | XX | XX |
| | XX.X | XX.X | XX.X | XX.X |
| 2) | XX.XX | XX.XX | XX.XX | XX.XX |
| Body Surface Area (m | XX.X | XX.X | XX.X | XX.X |
| n Mean SD | XX, | XX, | XX, | XX, |
| Median | XX | XX | XX | XX |
| Min, Max | | | | |
| riii, rida | | | | |
| Non-Imaging Efficacy Assessments | xx xx.x | xx xx.x | xx xx.x | XX |
| Baseline Distance Walked (meters) During 6-minute | XX XX.X | XX XX.X | XX XX.X | XX<br>XX.X |
| Walking Test | XX.X | XX.X | XX.X | XX.XX |
| n Mean SD | XX, XX | XX, XX | XX, XX | XX.X |
| Median | XX | XX | XX | XX, XX |
| Min, Max | XX.X | XX.X | XX.X | XX |
| · | XX.XX | XX.XX | XX.XX | XX.X |
| | XX.X | XX.X | XX.X | XX.XX |
| Baseline Levels of Log10 [NT-pro-BNP (ng/mL)] | XX, | XX, | xx, | XX.X |
| n Mean SD | XX | xx | XX | xx, |
| Median | xx xx.x | xx xx.x | xx xx.x | xx |
| Min, Max | (xx.xx) | (xx.xx) | (xx.xx) | xx xx.x |
| | xx.x xx.xx | xx.x xx.xx | xx.x xx.xx | (xx.xx) |
| Baseline Levels of NT-pro-BNP (ng/mL) | xx.x xx, xx | xx.x xx, xx | xx.x xx, xx | XX.X XX.XX |
| n | | | | xx.x xx, xx |
| Geometric Mean (CV%) | | | | |
| Mean | | | | |
| SD | | | | |
| Median | | | | |
| Min, Max | | | | |
| • | | | | |

| Baseline eGFR (ml/min) | XX XX | XX XX | XX XX | XX XX |
|---|---|---|---|---|
| n | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| < 60 | XX | XX | (AA.A.o.) | XX |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| ≥ 60 | XX.X | XX.X | XX.X | XX.X |
| Mean SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X XX, | XX.X XX, | XX.X XX, | XX.X XX, |
| Min, Max | XX | XX | XX | XX XX |
| | 2121 | 717 | 222 | 7171 |
| Baseline Kansas City Cardiomyopathy Questionnai | .re | | | |
| (KCCQ) Overall Summary Score | XX XX.X | xx xx.x | XX XX.X | XX |
| n | XX.XX | XX.XX | XX.XX | XX.X |
| | XX.X | XX.X | XX.X | XX.XX |
| | XX, XX | XX, XX | XX, XX | XX.X |
| | , | , | , | XX, XX |
| M' - Mari | | | | , |
| Min, Max | | | | |
| | XX | xx | xx | |
| Vital Signs | XX.X | XX.X | XX.X | XX |
| | XX.XX | XX.XX | XX.XX | XX.X |
| Deceline Heart Date (hom) | XX.X | XX.X | XX.X | XX.XX |
| Baseline Heart Rate (bpm) | XX, | XX, | xx, | XX.X |
| n Mean SD<br>Median | XX | XX | XX | XX, |
| | XX | XX | XX | XX |
| Min, Max | XX.X | XX.X | XX.X | XX |
| | XX.XX | XX.XX | XX.XX | XX.X |
| Baseline Respiration Rate (breaths/min) | XX.X | XX.X | XX.X | XX.XX |
| n Mean SD | xx, | XX, | XX, | XX.X |
| Median | XX | XX | XX | XX, |
| Min, Max | XX | XX | XX | XX |
| , | XX.X | XX.X | XX.X | XX |
| | XX.XX | XX.XX | XX.XX | XX.X |
| Baseline Systolic Blood Pressure (mmHg) | XX.X | XX.X | XX.X | XX.XX |
| n Mean SD | xx, | XX, | XX, | XX.X |
| Median | XX | XX | XX | XX, |
| Min, Max | XX | XX | XX | XX |
| | XX.X | XX.X | XX.X | XX |
| Decelled Dischalls Disch December (matter) | XX.XX | XX.XX | XX.XX | XX.X |
| Baseline Diastolic Blood Pressure (mmHg) | XX.X | XX.X | XX.X | XX.XX |
| n Mean SD | XX, | XX, | xx, | XX.X |
| Median | XX | XX | XX | XX, |
| Min, Max | | | | XX |

| Elamipretide 4 mg | Elamipretide 40 mg | Placebo | All Subjects |
|-------------------|--------------------|---------|--------------|
| (N=xx) | (N=xx) | (N=xx) | (N=xx) |

| | Elamipretide 4 mg | Elamipretide 40 mg | Placebo (N=xx) | 2 |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | | (N=xx) |
| oC) Stealth BioTherapeutics (Oral or Tympanic) ( PTPtqGan SPIJF-201 Median Min, Max | xx<br>xx.x<br>xx.xx<br>xx.x | xx<br>xx.x<br>xx.xx<br>xx.x<br>xx, xx | Elämipretide™ (MTP-<br>xx.x<br>xx.xx<br>xx.x<br>xx.<br>xx, | -131 <sup>xf</sup> or SC Injection) xx.x Page n of N xx.xx xx.x xx, xx, |
| Baseline Cardiovascular Physical Examination with<br>Clinically Significant Abnormalities<br>n Yes<br>No | xx xx<br>(xx.x%) xx<br>(xx.x%) | xx xx (%x.xx) | xx xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx xx<br>(%x.x%)<br>xx<br>(%x.x%) |

Baseline value is the last available measure prior to treatment.

SD = Standard deviation. Age is age at informed consent. n represents the number of subjects contributing to summary statistics. Percentages are based on n for each characteristic.

Source: Listings 1.4, 2.3, 7.1, 7.4.

Table 2.1b

Baseline Characteristics from MRI Safety
Population

| <br>Elamipretide 4 n | mg Elamipretide 40 mg | Placebo | All Subjects |
|----------------------|-----------------------|---------|--------------|
| (N=xx) | (N=xx) | (N=xx) | (N=xx) |

| Baseline Left Ventricular End Systolic Volume (LV ESV) (mL) [a] | | |
|---|---|---|
| n Mean SD | xx xx.x | XX |
| Median | XX.XX | XX.X |
| Min, Max | XX.X | XX.XX |
| HIII, HGA | xx, xx | XX.X |
| | | xx, xx |
| Baseline Left Ventricular Ejection Fraction (LVEF) (%) n Mean | | |
| SD | xx xx.x | XX |
| Median | xx.xx | XX.X |
| Min, Max | XX.X | XX.XX |
| | xx, xx | XX.X |
| | | xx, xx |
| Baseline Left Ventricular End Diastolic Volume (LV EDV) (mL) [a] n Mean SD | | |
| Median | XX XX.X | XX |
| Min, Max | XX.XX | XX.X |
| | XX.X | XX.XX |
| | XX, XX | XX.X |
| | | xx, xx |
| Percent Scarring of LV Mass (%) | | |
| n Mean SD | XX | |
| Median | XX.X<br>XX.XX | XX<br>XX.X |
| Min, Max | XX.XX<br>XX.X | xx.xx<br>xx.xx |
| | | XX.X |
| | XX, XX | |
| Ischemic/Non-ischemic Status [b] | | XX,<br>XX |
| n | | |
| Ischemic | | xx xx<br>(xx.x%) |
| Non-ischemic | | (XX.X%)<br>XX |
| | | (xx.x%) |
| | XX XX | (AA.AO) |
| | (xx.x%) xx | |
| | (xx.x%) | |

| Elamipretide 4 mg | g Elamipretide 40 mg | Placebo | All Subjects |
|-------------------|----------------------|---------|--------------|
| (N=xx) | (N=xx) | (N=xx) | (N=xx) |

Baseline value is the last available measure prior to treatment.

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

 ${\tt SD}={\tt Standard}$  deviation. n represents the number of subjects contributing to summary statistics. Percentages are based on n for each characteristic.

- [a] Value indexed by body surface area [BSA].
- [b] Ischemic status as determined by scar pattern. Source: Listings 2.1.

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM


#### Table 2.1c Baseline Characteristics from Echocardiography Safety Population

| Elamipretide 4 m | mg Elamipretide 40 mg | Placebo | All Subjects |
|------------------|-----------------------|---------|--------------|
| (N=xx) | (N=xx) | (N=xx) | (N=xx) |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

| Baseline E/A (Ratio Between Early And Late Mitral Inflow Velocity) | | |
|---|---|---|
| n Mean SD | XX XX.X | XX |
| Median | XX.XX | XX.X |
| Min, Max | XX.X | XX.XX |
| 11211/ 11011 | xx, xx | XX.X |
| | | XX, XX |
| Baseline E/e' (Ratio Between Early Mitral Inflow<br>Velocity And Mitral Annular Early Diastolic<br>Velocity) | | |
| n Mean | XX XX.X | XX |
| SD | XX.XX | XX.X |
| Median | XX.X | XX.XX |
| Min, Max | xx, xx | XX.X |
| | | XX, XX |
| Baseline Left Ventricular Ejection Fraction (LVEF) Biplane (%) n Mean SD Median Min, Max | xx xx.x<br>xx.xx<br>xx.x<br>xx. x | xx<br>xx.x<br>xx.xx<br>xx.xx |
| Baseline Left Ventricular Global Longitudinal<br>Strain (%)<br>n Mean<br>SD | | xx, xx |
| Median | xx xx.x | XX |
| Min, Max | xx.xx | XX.X |
| | xx.x | XX.XX |
| | xx, xx | XX.X |
| Baseline Left Atrial Volume (mL) [a] | xx | XX, XX |
| n Mean SD | xx.x | XX |
| Median | xx.xx | XX.X |
| Min, Max | XX.X | XX.XX |
| | xx, xx | XX.X |
| Baseline Left Ventricular Mass (g) [a] | | XX, |
| basetine bett ventifeutat Mass (g) [a] | | XX |

Draft YYYY


| | Elamipretide 4 mg Elamipretide 40 mg (N=xx) (N=xx) | | Placebo (N=xx | All Subjects (N=xx) |
|---|---|---|---|---|
| Maria | | | | , , , |
| n Mean | XX XX.X | XX XX.X | XX XX.X | XX XX.X |
| SD<br>Stealth BioTherapeutics, Inc.<br>Median<br>Protocol SPIHF-201 | XX.XX | XX.XX | <sup>XX</sup> Elamipretide™ (MTP | -131 for SC Injection) |
| Protocol, SPIHF-201 | XX.X | XX.X | XX.X | XX.X Page n of N |
| Min, Max Dol | XX, XX | xx, xx | XX, XX | xx, xx |
| | XX | XX | XX | XX |
| Baseline Mitral Regurgitation Severity (cm <sup>2</sup> ) | XX.X | XX.X | XX.X | XX.X |
| n Mean SD | XX.XX | xx.xx | xx.xx | XX.XX |
| Median | xx.x | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, | XX, |
| Tilly Han | | | XX | XX |
| | XX | XX | XX | xx |
| Baseline Tricuspid Regurgitation Severity (cm2) | XX.X | XX.X | XX.X | XX.X |
| n Mean SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, | XX, |
| | | | XX | xx |
| Baseline Right Ventricular Fractional Area Change | | | | |
| (%) n | XX XX.X | XX XX.X | XX XX.X | XX XX.X |
| Mean | xx.xx | XX.XX | XX.XX | XX.XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX, XX | xx, xx | XX, XX | xx, xx |
| Min, Max | | | | |
| Baseline Right Ventricular Systolic Pressure | | | | |
| (RVSP) (mmHg) | | | | |
| n Mean SD | vv vv v | VV VV V | vv vv v | vv vv v |
| Median | XX XX.X<br>XX.XX | XX XX.X<br>XX.XX | XX XX.X<br>XX.XX | XX XX.X<br>XX.XX |
| Min, Max | XX.X | XX.X | XX.X | XX.X |
| | XX, XX | XX, XX | XX, XX | XX, XX |
| | , **** | , | , | , **** |

Baseline value is the last available measure prior to treatment.

age at informed consent.

Source: Listings 2.2.

Table 2.2a

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

SD = Standard deviation. Age is

n represents the number of subjects contributing to summary statistics. Percentages are based on n for each characteristic.

<sup>[</sup>a] Value indexed by body surface area [BSA].

Demographic and Non-Imaging Baseline Characteristics ITT Population

Table 2.2b
Baseline Characteristics from MRI
ITT Population

Table 2.2c Baseline Characteristics from Echocardiography ITT Population

Table 2.3a

Demographic and Non-Imaging Baseline Characteristics Per-Protocol
Population

Table 2.3b
Baseline Characteristics from MRI
Per-Protocol Population

Table 2.3c Baseline Characteristics from Echocardiography Per-Protocol Population

#### 3. EFFICACY ANALYSIS

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

### 3.1 EFFICACY ANALYSIS

| | | | | | | | | | Linear<br>ence Between Trend |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | etween Elamipretide 40 | ) mg Test LV ESV |
| | _ | _ | | _ | _ | _ | _ | mipretide 4 P- | 3 m' |
| 5 - 1 - E - E - E | (mL) | 4 mg 40 | - | | acebo (95% | | Placebo (95% | mg (95% CI), P- | value Time |
| Point [a | | , , , | | alue [D] | CI), P-valu | | value [b] | [c] | |
| Baseline | | XX | XX | | Madian | Mean | XX.X | XX.X | |
| SD x | XX.XX | XX.XX | | | Median xx.x | | XX.X | | |
| | Min, | XX, XX | | xx, xx | | | | | |
| | Max | | | | | | | | |
| | | | | | Week 1 | | XX | XX | |
| | XX.X | XX.X | | | SD xx.x | X | XX.XX | | Median xx.x |
| X | XX.X | | | | | | | | |
| | Min, | xx, xx | | xx, xx | | | | | |
| | Max | | | | | | | | |
| | | | | | Change | | | from Baseline to | Week 1 |
| [d] | n | XX | | XX | | | | | |
| | Mean | XX.X | | XX.X | xx.x (xx.x, | xx.x)x.x | XXX | xx.x (xx.x, xx | .x)x.xxxx xx. |
| (xx.x, x | x.x)x.xxxx | x.xxxx | | | , , | • | | , , | , |
| • | | | | | | | | | |
| SD xx.xx | x xx.xx | Median xx.x | XX.X | | | | | | |
| | Min, | xx, xx | | xx, xx | | | | | |
| | Max | | | | | | | | |
| | | | | | 1 4 | | | | |
| _ | | | | | Week 4 | n | XX | XX | |
| | XX.X | XX.X | | | SD xx.x | ΪX | XX.XX | | Median xx.x |
| X | XX.X | | | | | | | | |
| | Min, | XX, XX | | xx, xx | | | | | |
| | Max | | | | | | | | |
| | | | | | Chang | е | n xx | XX | |
| | | | | | Table 3.1 | | | | |

Summary of Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI ITT Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

| Time Point | LV ESV | Elamipretide 4 mg (N=xx) | Elamipretide 40 mg Pl (N=xx) | acebo (N=xx) | Difference Between<br>Elamipretide 4 mg and<br>Placebo (95% CI), P-<br>value [b] | | Difference Between<br>Elamipretide 40 mg<br>and Elamipretide 4<br>mg (95% CI), Pvalue<br>[b] | Linear<br>Trend<br>Test<br>Pvalue |
|---|---|---|---|---|---|---|---|---|
| from<br>Baseline<br>to Week 4 | | | | | | | | |
| [d] | | | | | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | |
| | | | | | | , , , | | X.XXXX |
| | Mean | xx.x | | | X.XXX | X.XXXX | X.XXXX | |
| | | | | XX.X | | | | |
| | SD | XX.XX | | | | | | |
| | Median | XX.X XX, | XX.XX | XX.X | | | | |
| | Min, Max | XX | | XX, XX | | | | |

ITT Population = all subjects who were randomized and receive at least 1 dose of IMP, according to the treatment group to which the subjects were randomized.

Baseline value is the last available measure prior to treatment.

- [a] Value indexed by body surface area [BSA].
- [b] 95% confidence interval is based on the t-distribution and Lsmean of between treatment group difference from a mixed model repeated measures for the change from baseline which includes treatment group, treatment-by-visit interaction, and ischemic/non-ischemic as factors and the baseline value and baseline value-by-visit interaction as continuous covariates. P-value corresponds to a 2-sided significance level of the between treatment group difference from the mixed model repeated measures. [c] Linear trend test.
- [d] Change from Baseline at time point t: Changet = Value t ValueBaseline. Source:

Listings 2.1

# Table 3.2 Summary of Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.3
Summary of Change From Baseline in Left Ventricular Ejection Fraction (LVEF), Assessed by MRI ITT Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM
[Change 2nd column header to: LVEF]

[Remove footnote for indexing to BSA]

## Table 3.4 Summary of Change From Baseline in Left Ventricular Ejection Fraction (LVEF), Assessed by MRI Per-Protocol Population

[Change 2nd column header to: LVEF]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

[Remove footnote for indexing to BSA]

Table 3.5 Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV), Assessed by MRI ITT Population

[Change 2nd column header to: LV EDV]

Table 3.6
Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV), Assessed by MRI
Per-Protocol Population

[Change 2nd column header to: LV EDV]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.7
Summary of Change From Baseline in Left Ventricular Stroke Volume (LVSV), Assessed by MRI ITT Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


[Change 2nd column header to: LVSV] [Remove footnote for indexing to BSA]

# Table 3.8 Summary of Change From Baseline in Left Ventricular Stroke Volume (LVSV), Assessed by MRI Per-Protocol Population

[Change 2nd column header to: LVSV] [Remove footnote for indexing to BSA]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.9
Summary of Change From Baseline in Left Ventricular Cardiac Output (LVCO), Assessed by MRI ITT Population

[Change 2nd column header to: LVCO]
[Remove footnote for indexing to BSA]

Table 3.10
Summary of Change From Baseline in Left Ventricular Cardiac Output (LVCO), Assessed by MRI
Per-Protocol Population

[Change 2nd column header to: LVCO] [Remove footnote for indexing to BSA]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

#### Table 3.11 Summary of Change From Baseline in Left Ventricular Myocardial Mass (LV Mass), Assessed by MRI ITT Population

[Change 2nd column header to: LV Mass]

Table 3.12 Summary of Change From Baseline in Left Ventricular Myocardial Mass (LV Mass), Assessed by MRI Per-Protocol Population

[Change 2nd column header to: LV Mass]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.13
Summary of Change From Baseline in Right Ventricular End Systolic Volume (RV ESV), Assessed by MRI ITT Population

[Change 2nd column header to: RV ESV]

Table 3.14
Summary of Change From Baseline in Right Ventricular End Systolic Volume (RV ESV), Assessed by MRI
Per-Protocol Population

[Change 2nd column header to: RV ESV]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Report generated by program: /sasdir/xxxx.sas

Draft YYYY


# Table 3.15 Summary of Change From Baseline in Right Ventricular End Diastolic Volume (RV EDV), Assessed by MRI ITT Population

[Change 2nd column header to: RV EDV]

# Table 3.16 Summary of Change From Baseline in Right Ventricular End Diastolic Volume (RV EDV), Assessed by MRI Per-Protocol Population

[Change 2nd column header to: RV EDV]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.17
Summary of Change From Baseline in Right Ventricular Ejection Fraction (RVEF), Assessed by MRI ITT Population

[Change 2nd column header to: RVEF]
[Remove footnote for indexing to BSA]

Table 3.18
Summary of Change From Baseline in Right Ventricular Ejection Fraction (RVEF), Assessed by MRI
Per-Protocol Population

[Change 2nd column header to: RVEF]

[Remove footnote for indexing to BSA]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

### Table 3.19 Summary of Change From Baseline in E/A (Ratio Between Early And Late Mitral Inflow Velocity), Assessed by Echocardiography ITT Population

[Change 2nd column header to: E/A, Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

[Remove footnote for indexing to BSA]

#### Table 3.20

Summary of Change From Baseline in E/A (Ratio Between Early And Late Mitral Inflow Velocity), Assessed by Echocardiography Per-Protocol Population

[Change 2nd column header to: E/A, Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.] [Remove

footnote for indexing to BSA]

#### Table 3.21

Summary of Change From Baseline in E/e' (Ratio Between Early Mitral Inflow Velocity and Mitral Annular Early Diastolic Velocity), Assessed by Echocardiography ITT Population

[Change 2nd column header to: E/e', Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

[Remove footnote for indexing to BSA]

#### Table 3.22

Summary of Change From Baseline in E/e' (Ratio Between Early Mitral Inflow Velocity and Mitral Annular Early Diastolic Velocity), Assessed by Echocardiography Per-Protocol Population

[Change 2nd column header to: E/e', Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

[Remove footnote for indexing to BSA]

## Table 3.23 Summary of Change From Baseline in Left Atrial Volume, Assessed by Echocardiography ITT Population

[Change 2nd column header to: LAV, Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

### Table 3.24 Summary of Change From Baseline in Left Atrial Volume, Assessed by Echocardiography Per-Protocol Population

[Change 2nd column header to: LAV, Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.25
Summary of Change From Baseline in Left Ventricular Global Longitudinal Strain, Assessed by Echocardiography ITT Population

[Change 2nd column header to: LV GLS, Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

[Remove footnote for indexing to BSA]

Table 3.26
Summary of Change From Baseline in Left Ventricular Global Longitudinal Strain, Assessed by Echocardiography
Per-Protocol Population

Report generated by program: /sasdir/xxxx.sas -MM-DD +H+:MM

[Change 2nd column header to: LV GLS, Change Timepoints to Weeks 4 and 6, Change footnote to Listing 2.2]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

[Remove footnote for indexing to BSA]

Table 3.27
Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV), Assessed by Echocardiography ITT
Population

LV EDV Elamipretide Elamipretide (mL) 4 mg 40 mg Placebo Time Point [a] (N=xx) (N=xx)

Draft YYYY

| | SD | XX.XX | XX.X |
|-----------|-------------|---------|--------|
| | Median | XX.X | XX.XX |
| | Min, | XX, XX | xx.x |
| | Max | | XX, XX |
| | n | xx | |
| | Mean | xx.x | XX |
| | SD | XX.XX | XX.X |
| | Median | XX.X | XX.XX |
| Week 4 | Min,<br>Max | xx, | XX.X |
| week 4 | Max | XX | XX, |
| | | | XX |
| | n Mean | | |
| | SD | XX XX.X | |
| | Median | XX.XX | XX |
| Change | Min, | XX.X | XX.X |
| from | Max | xx, xx | XX.XX |
| Baseline | n | | XX.X |
| to Week 4 | Mean | | XX, XX |
| [a] | SD | XX | |
| [d] | Median | | |
| | Min, | XX.X | XX |
| | Max | XX.XX | XX.X |
| | | XX.X | XX.XX |
| | | XX, | XX.X |
| | | xx | xx, |
| | n Mean | | XX |
| | SD | | |
| | Median | | |
| Week 6 | | XX XX.X | |
| | | XX.XX | |
| | | XX.X | XX |
| | | | XX.X |
| | | | XX.XX |
| | | | XX.X |
| Change | | | |
| from | | | |

Baseline n Mean xx xx.x


Baseline to Week 6 XX

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

| | LV EDV | Elamipretide | Elamipretide | |
|------------|--------|--------------|--------------|---------|
| | (mL) | 4 mg | 40 mg | Placebo |
| Time Point | [a] | (N=xx) | (N=xx) | (N=xx) |
| | Min, | XX, XX | | XX, XX |
| | Max | | | |

ITT Population = all subjects who were randomized and receive at least 1 dose of IMP, according to the treatment group to which the subjects were randomized.

Baseline value is the last available measure prior to treatment.

[Source: Listings 2.2a] Change from Baseline at time point t: Change t = Value t - ValueBaseline.

#### Table 3.28 Summary of Change From Baseline in Left Ventricular End Diastolic Volume (LV EDV), Assessed by Echocardiography Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.29 Summary of Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by Echocardiography ITT Population

Table 3.30 Summary of Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by Echocardiography Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.31 Summary of Change From Baseline in Biplane Ejection Fraction (EF), Assessed by Echocardiography **ITT Population** 

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


#### Table 3.32 Summary of Change From Baseline in Biplane Ejection Fraction (EF), Assessed by Echocardiography Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.33
Summary of Change From Baseline in Left Ventricular Mass, Assessed by Echocardiography ITT Population

Table 3.34
Summary of Change From Baseline in Left Ventricular Mass, Assessed by Echocardiography
Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.35
Summary of Change From Baseline in Mitral Regurgitation Severity, Assessed by Echocardiography ITT Population

Table 3.36
Summary of Change From Baseline in Mitral Regurgitation Severity, Assessed by Echocardiography
Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.37

Report generated by program: /sasdir/xxxx.sas

Summary of Change From Baseline in Tricuspid Regurgitation Severity, Assessed by Echocardiography ITT Population

Table 3.38

Summary of Change From Baseline in Tricuspid Regurgitation Severity, Assessed by Echocardiography Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.39

Summary of Change From Baseline in Right Ventricular Fractional Area Change, Assessed by Echocardiography ITT Population

**Table 3.40** 

Summary of Change From Baseline in Right Ventricular Fractional Area Change, Assessed by Echocardiography Per-Protocol Population

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Table 3.41

Summary of Change From Baseline in Right Ventricular Systolic Pressure (RVSP), Assessed by Echocardiography ITT Population

Table 3.42

Summary of Change From Baseline in Right Ventricular Systolic Pressure (RVSP), Assessed by Echocardiography Per-Protocol Population

Report generated by program: /sasdir/xxxx.sas

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

### Table 3.43 Summary of Change From Baseline in Distance Walked (meters) During 6-minute Walking Test (6MWT) ITT Population

[From Table 3.1 mock, Change 2nd column header to: 6MWT, Change Timepoints to Week 4, Change footnote to Listing 2.3] [Remove

footnote for indexing to BSA]

[Change footnote [b] to:

[b] 95% confidence interval is based on the t-distribution and Lsmean of between treatment group difference from an ANCOVA model for the change from baseline which includes treatment group, ischemic/non-ischemic, and treatment-by-ischemic/non-ischemic interaction as factors and the baseline value as a continuous covariate. P-value corresponds to a 2-sided significance level of the between treatment group difference from the ANCOVA model.]

## Table 3.44 Summary of Change From Baseline in Distance Walked (meters) During 6-minute Walking Test (6MWT) Per-Protocol Population

[From Table 3.1 mock, Change 2nd column header to: 6MWT, Change Timepoints to Week 4, Change footnote to Listing 2.3]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.] [Remove

footnote for indexing to BSA]

[Change footnote [b] to:

[b] 95% confidence interval is based on the t-distribution and Lsmean of between treatment group difference from an ANCOVA model for the change from baseline which includes treatment group, ischemic/non-ischemic, and treatment-by-ischemic/non-ischemic interaction as factors and the baseline value as a continuous covariate. P-value corresponds to a 2-sided significance level of the between treatment group difference from the ANCOVA model.]

Table 3.45
Summary of Change From Baseline in Levels of NT-pro-BNP ITT Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

[From Table 3.1 mock, Change 2nd column header to: NT-pro-BNP, Change Timepoints to Weeks 1, 2, 4, and 6, Change footnote to Listing 2.3] [Remove footnote for indexing to BSA]

[Change footnote [b] to:

[a] Difference between treatments and inferential statistics based on log10 (NT-pro-BNP). 95% confidence interval is based on the t-distribution and Lsmean of between treatment group difference from a mixed model repeated measures for the change from baseline which includes treatment group, treatment-by-visit interaction, ischemic/non-ischemic as factors and the baseline value and baseline value-by-visit interaction as continuous covariates. P-value corresponds to a 2-sided significance level of the between treatment group difference from the mixed model repeated measures.]

[Change footnote [c] to:

[b] Linear trend test of log10 (NT-pro-BNP).]

## Table 3.46 Summary of Change From Baseline in Levels of NT-pro-BNP Per-Protocol Population

[From Table 3.1 mock, Change 2nd column header to: NT-pro-BNP, Change Timepoints to Weeks 1, 2, 4, and 6, Change footnote to Listing 2.3] [Remove footnote for indexing to BSA]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

[Change footnote [b] to:

[a] Difference between treatments and inferential statistics based on log10 (NT-pro-BNP). 95% confidence interval is based on the t-distribution and Lsmean of between treatment group difference from a mixed model repeated measures for the change from baseline which includes treatment group, treatment-by-visit interaction, ischemic/non-ischemic as

factors and the baseline value and baseline value-by-visit interaction as continuous covariates. P-value corresponds to a 2-sided significance level of the between treatment group difference from the mixed model repeated measures.]

[Change footnote [c] to: [b] Linear trend test of log10 (NT-pro-BNP).]

Table 3.47 Summary of Change From Baseline in Levels of hsTroponin ITT Population

[From Table 3.1 mock, Change 2nd column header to: hsTroponin, Change Timepoints to Weeks 1, 2, 4, and 6, Change footnote to Listing 6.4]

[Remove footnote for indexing to BSA]

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


### Table 3.48 Summary of Change From Baseline in Levels of hsTroponin Per-Protocol Population

[From Table 3.1 mock, Change 2nd column header to: hsTroponin, Change Timepoints to Weeks 1, 2, 4, and 6, Change footnote to Listing 6.4] [Remove footnote for indexing to BSA]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

### Table 3.49 Summary of Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score ITT Population

[From Table 3.1 mock, Change 2nd column header to: KCCQ, Change Timepoints to Week 4, Change footnote to Listing 2.3] [Remove footnote for indexing to BSA]

[Change footnote [b] to:

[b] 95% confidence interval is based on the t-distribution and Lsmean of between treatment group difference from an ANCOVA model for the change from baseline which includes treatment group, ischemic/non-ischemic, and treatment-by-ischemic/non-ischemic interaction as factors and the baseline value as a continuous covariate. P-value corresponds to a 2-sided significance level of the between treatment group difference from the ANCOVA model.]

Table 3.50
Summary of Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Per-Protocol Population

[From Table 3.1 mock, Change 2nd column header to: KCCQ, Change Timepoints to Week 4, Change footnote to Listing 2.3] [Remove footnote for indexing to BSA]

[Change first footnote to: Per-Protocol Population = all subjects who were randomized and receive at least 1 dose of IMP, without major protocol violations/deviations, according to the treatment group to which the subjects were randomized.]

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

#### [Change footnote [b] to:

[b] 95% confidence interval is based on the t-distribution and Lsmean of between treatment group difference from an ANCOVA model for the change from baseline which includes treatment group, ischemic/non-ischemic, and treatment-by-ischemic/non-ischemic interaction as factors and the baseline value as a continuous covariate. P-value corresponds to a 2-sided significance level of the between treatment group difference from the ANCOVA model.]

#### 4. PLASMA CONCENTRATION ANALYSIS

Table 4.1
Summary of Plasma Concentrations of Elamipretide and Metabolites (M1, M2) by Time Point Safety Population

| | Elamipretide | M1 | M2 |
|---|---|---|---|
| Concentration (unit) | (N=xx) | (N=xx) | (N=xx) |
| Day 1 | | | |
| Pre-dose | | | |
| n | XX | xx | XX |
| Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) |
| SD | XX.XX | XX.X | xx.xx |
| Median | XX.X | xx | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Geometric Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) |
| Post-dose | | | |
| N | XX | XX | XX |
| Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) |
| SD | XX.XX | XX.X | XX.XX |
| Median | XX.X | Xx | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Geometric Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) |
| Week 1 | Pre-dose | | |
| n | XX | XX | XX |
| Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) |
| SD | XX.XX | XX.X | XX.XX |
| Median | XX.X | XX | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Geometric Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) |
| Post-dose | | | |
| N | XX | XX | XX |
| Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) |
| SD | XX.XX | XX.X | XX.XX |
| Report generated by program: /sasdir/xxxx | .sas | | Draft YYYY |

| Geometric Mean (CV%) Steartrigsfortherapeutics, Inc. Protocol SPIHF-201 Mean (CV%) SD Median Min, Max Geometric Mean (CV%) Week 4 n | (xx.xx) | xx, xx<br>xx.x<br>(xx.x)<br>xx xx.x<br>(xx.x)<br>xx.x xx<br>xx, xx | (XX.XX) | - |
|---|---|---|---|---|
| Protocol SPIHF-201 Mean (CV%) SD Median Min, Max Geometric Mean (CV%) Week | (xx.xx) xx.xx xx.x xx, xx xx.x (xx.xx) xx xx.x (xx.xx) xx.xx (xx.xx) xx.xx xx.x (xx.xx) xx.xx xx.x xx, xx xx.x (xx.xx) xx xx.x | (xx.x) xx.x Xx Elamipretide™ xx, xx xx.x (xx.x) xx xx.x (xx.x) xx xx.x xx.x xx, xx | (xx.xx) (MRR-1631 xfor SC xx, xx xx.x (xx.xx) xx xx.x (xx.xx) xx xx.x (xx.xx) xx.xx xx, xx xx.x | Page n of N Median |
| Protocol SPIHF-201 Mean (CV%) SD Median Min, Max Geometric Mean (CV%) Week | xx.xx xx.x<br>xx, xx xx.x<br>(xx.xx)<br>xx xx.x<br>(xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x<br>(xx.xx)<br>xx xx.x | xx.x Xx Elamipretide™ xx, xx xx.x (xx.x) xx xx.x (xx.x) xx xx.x xx.x xx, xx | (MRR-1631 xfor SC<br>xx, xx xx.x<br>(xx.xx)<br>xx xx.x<br>(xx.xx)<br>xx xx.x<br>(xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x | Page n of N Median |
| Protocol SPIHF-201 Mean (CV%) SD Median Min, Max Geometric Mean (CV%) Week | xx, xx xx.x (xx.xx) | xx, xx<br>xx.x<br>(xx.x)<br>xx xx.x<br>(xx.x)<br>xx.x xx<br>xx, xx | xx, xx xx.x<br>(xx.xx)<br>xx xx.x<br>(xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x | Page n of N Median |
| Mean (CV%) SD Median Min, Max Geometric Mean (CV%) Week | (xx.xx)<br>xx xx.x<br>(xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x<br>(xx.xx)<br>xx xx.x | xx.x<br>(xx.x)<br>xx xx.x<br>(xx.x)<br>xx.x xx<br>xx, xx | (xx.xx)<br>xx xx.x<br>(xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x | Median |
| SD Median Min, Max Geometric Mean (CV%) Week | xx xx.x<br>(xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x<br>(xx.xx)<br>xx xx.x | (xx.x)<br>xx xx.x<br>(xx.x)<br>xx.x xx<br>xx, xx | xx xx.x<br>(xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x | |
| Median<br>Min, Max<br>Geometric Mean (CV%)<br>Week | (xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x<br>(xx.xx)<br>xx xx.x | xx xx.x<br>(xx.x)<br>xx.x xx<br>xx, xx | (xx.xx)<br>xx.xx xx.x<br>xx, xx xx.x | |
| Min, Max<br>Geometric Mean (CV%)<br>Week | xx.xx xx.x<br>xx, xx xx.x<br>(xx.xx)<br>xx xx.x | (xx.x)<br>xx.x xx<br>xx, xx | xx.xx xx.x<br>xx, xx xx.x | |
| Geometric Mean (CV%)<br>Week | xx, xx xx.x<br>(xx.xx)<br>xx xx.x | xx.x xx<br>xx, xx | xx, xx xx.x | XX.X |
| Week | (xx.xx)<br>xx xx.x | xx, xx | • | |
| | xx xx.x | | | Xx |
| 4 | | | (xx.xx) | XX.X |
| 4 n | , | XX.X | XX XX.X | Min, Max |
| Mean (CV%) | (xx.xx) | (xx.x) | (xx.xx) | XX, XX |
| SD | XX.XX XX.X | XX XX.X | XX.XX XX.X | XX, XX |
| Median | xx, xx xx.x | (xx.x) | XX, XX XX.X | XX, XX |
| Min, Max | (xx.xx) | XX.X XX | (xx.xx) | |
| Geometric Mean (CV%) | | XX, XX | | Geometric |
| Week | | XX.X | | Mean (CV%) |
| 6 n | | (xx.x) | | XX.X |
| Mean (CV%) | | | | (xx.xx) |
| SD | | | | XX.X |
| Median | | | | (xx.x) |
| Min, Max | | | | XX.X |
| Geometric Mean (CV%) | | | | (xx.xx) |
| Week 2 Pr | e-dose | | | |
| n | XX | XX | XX | |
| Mean (CV%) | xx.x (xx.xx) | xx.x (xx.x) | xx.x (xx.xx) | |
| SD xx.xx xx.x xx.xx Median xx.x xx xx.x | | | | |

N = number of subjects treated with Elamipretide. n

Values below Lower Limit of Quantification (LLQ) are set to LLQ/2.

Source: Listing 4.1

#### 5. EXTENT OF EXPOSURE TO STUDY MEDICATION

# Table 5.1 Extent of Exposure to Study Medication by Treatment Group Safety Population

| Elamipretide 4 mg | Elamipretide 40 mg | Placebo (N=xx) | All Subjects |
|-------------------|--------------------|----------------|--------------|
| (N=xx) | (N=xx) | | (N=xx) |

Draft YYYY


<sup>=</sup> number of subjects with data.

SD = standard deviation.

CV = coefficient of variation.

| Study Treatment Exposure (days) [a] | XX | XX | XX | XX |
|-------------------------------------|--------|----------|----------|--------|
| N | xxx.x | XXX.X | XXX.X | XXX.X |
| Mean SD | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | xxx.x | XXX.X | XXX.X | XXX.X |
| Min, Max | xxx, | xxx, xxx | xxx, xxx | xxx, |
| | XXX | | | XXX |
| | XX | xx | xx | xx |
| tudy Treatment Compliance (%) | XXX.X | XXX.X | XXX.X | XXX.X |
| Mean SD | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median<br>Min, Max | xxx.x | XXX.X | XXX.X | XXX.X |
| | xxx, | xxx, xxx | xxx, xxx | XXX, |
| | xxx | | | XXX |

SD = Standard deviation.

#### 6. ADVERSE EVENTS

Table 6.1

Overall Summary of Treatment-Emergent Adverse Events by Treatment Group

Safety Population

| | Elamipretide (N=xx) | 4 mg | Elamipretide 4<br>(N=xx) | ) mg | Placebo<br>(N=xx) | | All Subje<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|
| | # of<br>Subjects n<br>(%) | | # of<br>Subjects n<br>(%) | | # of<br>Subjects n<br>(%) | | # of<br>Subjects n<br>(%) | |
| | | E | | E | | E | | E |
| bjects with at least one TEAE | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | XX |
| ubjects with TEAEs Related to Study reatment [a] | xx (xx.x%) | xx | xx (xx.x%) | XX | xx (xx.x%) | xx | xx (xx.x%) | XX |
| ubjects with Serious TEAEs | xx (xx.x%) | xx | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | XX |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

n represents the number of subjects contributing to summary statistics. Percentages are based on n for each characteristic. Percentages are based on n.

<sup>[</sup>a] Study treatment exposure (days) = Treatment end date - treatment start date - number of days of missed doses + 1. Source: Listing 3.1

| Subjects with Serious TEAEs Related to Study Treatment [a] | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | XX |
|---|---|---|---|---|---|---|---|---|
| Subjects with TEAEs Leading to<br>Discontinuation of Study Drug | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) | XX | xx (xx.x%) | XX |
| Deaths - All<br>Causes | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | XX |

TEAE = Treatment-Emergent Adverse Event. An adverse event is considered treatment-emergent if the date of onset is on or after the date of first dose of study medication, or worsening during the treatment period + 30 days.

E = number of events

[a] Related = unlikely related, probably related or possibly related to study drug.

Source: Listing 5.1

Program: /data/dev/client29/SPIHF201/programs/statout/xxxxxxx.sas DDMMMYYYY:HH:MM (Page x of y)

Table 6.2
Incidence of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| | Elamipretide 4 mg<br>(N=xx) | Elamipretide 40 mg (N=xx) | Placebo<br>(N=xx) | All Subjects<br>(N=xx) n |
|---|---|---|---|---|
| System Organ Class<br>Preferred Term | n (%) | n (%) | n (%) | (%) |
| FIETETIEU TETM | | | | |
| At Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | | | | xx (xx.x%) |
| MedDRA SOC1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MedDRA SOC2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (xx.x%) xx |
| Preferred Term 2 Etc. | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (xx.x%) |

Report generated by program: /sasdir/xxxx.sas

-MM-DD HH:MM

TEAE = Treatment Emergent Adverse Event. An adverse event is considered treatment-emergent if the date of onset is on or after the date of first dose of study medication, or worsening during the treatment period + 30 days.

If more than one adverse event is coded to the same preferred term for a subject, the subject will be counted only once for that preferred term. If more than one preferred term is coded to the same System Organ Class for a subject, the subject will be counted only once for that System Organ Class. Adverse events coded using MedDRA version 20.0.

Source: Listing 5.1

Note to Programmer: SOCs sorted alphabetically. PTs sorted within SOCs in decreasing order of frequency in the all subject group.

Subjects having several AEs with the same SOC will be counted only once for that particular SOC.

Subjects having several AEs with the same PT will be counted only once for that particular PT.

Table 6.3
Incidence of Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term Safety Population

| System Organ Class<br>Preferred Term | Elamipretide 4 mg<br>(N=xx)<br>n (%) | Elamipretide 40 mg (N=xx) n (%) | Placebo<br>(N=xx)<br>n (%) | All Subjects<br>(N=xx) n<br>(%) |
|---|---|---|---|---|
| At Least One TESAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | | | | xx (xx.x%) |
| MedDRA SOC1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


| MedDRA SOC2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) xx |
|------------------|------------|------------|------------|---------------|
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (xx.x%) xx |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (xx.x%) |
| Etc. | | | | |

TESAE (Treatment Emergent Serious Adverse Event) = serious adverse events occurring on or after the date of first dose of study medication, or worsening during the treatment period + 30 days. The definition of serious adverse event is in Protocol Section 9.6. If more than one serious adverse event is coded to the same preferred term for a subject, the subject will be counted only once for that preferred term. If more than one preferred term is coded to the same System Organ Class for a subject, the subject will be counted only once for that System Organ Class.

Percentages are based on N.

Adverse events coded using MedDRA version 20.0.

Source: Listings 5.2

Note to Programmer: SOCs sorted alphabetically. PTs sorted within SOCs in decreasing order of frequency in the all subject group. Subjects having several SAEs with the same SOC will be counted only once for that particular SOC. Subjects having several SAEs with the same PT will be counted only once for that particular PT.

Table 6.4
Incidence of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Intensity
Safety Population

| System Organ | Elamipretide 4 mg | Elamipretide 40 mg | Placebo | All Subjects |
|---|---|---|---|---|
| Class | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Preferred M | Mild Moderate Severe Mild Mo | oderate Severe | Mild Moderate Severe | Moderate Severe<br>Mild |
| Term | n (%) n (%) _n (%) | n (%) n (%) n (%) | n (%) n (%) n (%) | n (%) n (%) n (%) |
| | | | | At Least One xx |
| XX XX<br>TEAE | xx xx xx xx (xx.x%) (xx.x%) | xx xx xx xx (xx.x%) (xx. | xx xx<br>x%) (xx.x%) (xx.x%) (xx.x%) (xx | .x%) (xx.x%) (xx.x%) (xx.x%) |
| MedDRA SOC1 | xx xx xx xx (xx.x%) (xx.x%) | xx xx xx xx (xx.x%) (xx. | xx xx xx xx<br>x%) (xx.x%) (xx.x%) (xx | xx xx xx xx xx (%x.x%) (xx.x%) |
| Report generat | ted by program: /sasdir/xxxx. | sas | | Draft YYYY |

| Preferred<br>Term 1<br>Preferred | xx<br>(xx.x%)<br>xx | xx<br>(xx.x%)<br>xx | xx<br>(xx.x%)<br>xx | xx | xx<br>xx | xx<br>(xx.x%) (xx.x%)<br>xx | xx<br>(xx.x%)<br>xx | xx<br>(xx.x%)<br>xx | xx<br>(%x.x%)<br>xx | (xx.x%) | xx<br>(xx.x%)<br>xx | xx<br>(xx.x%)<br>xx | xx<br>(xx.x%)<br>xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Term 2 | | (xx.x%) | | **** | | (xx.x%) (xx.x%) | | | | (xx.x%) | | (xx.x%) | |
| | (2221 • 21 0 ) | (2121 • 21 0 ) | (222.22) | | | (MM.MO) (MM.MO) | (222.20) | (222.220) | (222.220) | (2121 • 21 0 ) | (222.22.0) | (2121 • 21 0 ) | (2121 • 21 0 ) |
| MedDRA SOC2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | | XX | XX | XX |
| | (xx.x%) | (xx.x%) | (xx.x%) | | | (xx.x%) (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Preferred | XX | XX | XX | XX | XX | XX | XX | XX | XX | | XX | XX | XX |
| Term 1 | (xx.x%) | (xx.x%) | (xx.x%) | | | (xx.x%) (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Preferred | XX | XX | XX | XX | XX | XX | XX | XX | XX | | XX | XX | XX |
| Term 2 | (xx.x%) | (xx.x%) | (xx.x%) | | | (xx.x%) (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| | | | | | | | | | | | E | tc. | |

TEAE = Treatment Emergent Adverse Event. An adverse event is considered treatment-emergent if the date of onset is on or after the date of first dose of study medication, or worsening during the treatment period + 30 days. Only the worst grade of intensity is counted for multiple occurrences of the same adverse event for a given subject. Adverse events coded using MedDRA version 20.0. Source: Listing 5.1

### Note to Programmer: SOCs and PTs sorted alphabetically.

Table 6.5
Incidence of Study Treatment Related Adverse Events by System Organ Class, Preferred Term, and Intensity Safety
Population

| System<br>Organ Class | | | | 0 mg | | Placebo<br>(N=xx) | All Subjects (N=xx) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred<br>Term | Mild | Moderate | Severe n | Mild<br>n (%) | Moderate | Severe<br>n (%) | Mild | Moderate | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) |
| | <u>n (%)</u> | n (%) | (%) | 11 (0) | n (%) | | <u>n (%)</u> | <u>n (%)</u> | | | | |
| At Least<br>One Study<br>Treatment | xx<br>(xx.x%) | xx<br>(xx.x%) | XX | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx | xx | xx | xx |
| Related AE | | | (xx.x%) | | | | | | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


| MedDRA SOC1 Preferred Term 1 Preferred Term 2 | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>(xx.x%)<br>(xx.x%) | xx<br>xx | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>(xx.x%)<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>xx (xx.x%)<br>xx xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA SOC2 Preferred Term 1 Preferred Term 2 Etc. | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>(xx.x%)<br>(xx.x%) | XX<br>XX | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>(xx.x%)<br>(xx.x%) | xx<br>xx (xx.x%)<br>xx xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) |

Study Treatment Related AE is a treatment-emergent adverse event classified by investigators as unlikely related, probably related or possibly related to study drug.

Only the worst grade of intensity is counted for multiple occurrences of the same adverse event for a given subject. Adverse events coded using MedDRA version 20.0.

Source: Listing 5.1

#### Note to Programmer: SOCs and PTs sorted alphabetically.

Table 6.6
Incidence of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug
Safety Population

| Elamipretide 4 | mg Elamipretide 40 mg | Placebo (N= | xx) All Subjects |
|----------------|-----------------------|-------------|------------------|
| (N=xx) | (N=xx) | | (N=xx) |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

| System Organ Class | Not Related | Related n | Not Related | Related n | Not Related | Related n | Not Related | Related n |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | (%) n (%) | | (응) n (응) | | (%) n (%) | | (%) n (%) | |
| At Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MedDRA SOC1 Preferred Term 1 Preferred Term 2 | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| MedDRA SOC2 Preferred Term 1 Preferred Term 2 | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

TEAE = treatment Emergent Adverse Event. An adverse event is considered treatment-emergent if the date of onset is on or after the date of first dose of study medication, or worsening during the treatment period + 30 days.

Not Related = unrelated to study drug; Related = unlikely related, probably related or possibly related to study drug. If a subject had more than one occurrence in the same event category, only the most related occurrence was counted. Adverse events coded using MedDRA version 20.0.

Source: Listing 5.1

Note to Programmer: SOCs sorted alphabetically. PTs sorted within SOCs in decreasing order of frequency in the related-all subject column.

Table 6.7
Incidence of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug by System Organ Class and Preferred Term Safety Population

| - | | Elamipretide 4 mg | Elamipretide 40 mg (N=xx) Placebo | All Subjects |
|---|---|---|---|---|
| | | (N=xx) | (N=XX) | (N=xx) |
| System Organ Class | Preferred Term | n (%) | n (%) n (%) | n (%) |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

| | | | | | xx (xx.x%) |
|---|---|---|---|---|---|
| Any Adverse Event Leadi<br>Discontinuation of<br>Study Drug | ng to<br>Any | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| MedDRA SOC1 | Any | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | PT1 | (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | PT2 | (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <br>Any | ( ) | ( | ( | xx (xx.x%) |
| | PT1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MedDRA SOC2 | | (x (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | PT2 | (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Etc.

Percentages are based on N. Adverse events coded using MedDRA version 20.0. Source: Listing 5.3

Note to Programmer: SOCs sorted alphabetically. PTs sorted within SOCs in decreasing order of frequency in the all subject group.

Table 6.8
Deaths
Safety Population

| | | | | | Was Autopsy |
|---|---|---|---|---|---|
| Subject ID | Study Treatment | Age/Sex [a] | Date of Death | Study Day of Death [b] | Performed? (Yes/No) |
| XXXX | Elamipretide 4 mg | 73/F | vvvv-mmm-dd | XX | Xxx |

Draft YYYY


Elamipretide  $^{\text{TM}}$  (MTP-131 for SC Injection) Page n of N

xxxx Placebo 75/M yyyy-mmm-dd xx Xx

[a] Age is age at informed consent in years. F = Female, M = Male.

[Source: b]Study Day = date of death - date of first dose + 1. Listing 5.2

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

#### 7. CLINICAL LABORATORY EVALUATIONS

Table 7.1a Change From Baseline in Hematology Parameters by Visit Safety Population

| Parameter (unit) | Elam | ipretide 4 mg<br>(N=xx) | Elami | pretide 40 mg (N=xx) | | Placebo (N=xx) All Subject = xxx) | | |
|---|---|---|---|---|---|---|---|---|
| | Actual | Change From | Actual | Change From | Actual | Change From | Actual | Change From |
| Time Point | Value | Baseline | Value | Baseline | Value | Baseline | Value | Raseline |

| Baseline[a] | n Mean | XX | | XX | | XX | | XX | |
|---|---|---|---|---|---|---|---|---|---|
| | SD<br>Median | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | | XX.XXX | | XX.XXX | | XX.XXX | | XX.XXX | |
| | Min, | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | Max | XX.X, | | XX.X, | | XX.X, | | XX.X, | |
| | | XX.X | | XX.X | | XX.X | | XX.X | |
| | n Mean | XX | | XX | | XX | | XX | |
| | SD | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | Median | XX.XXX | XX XX.XX | XX.XXX | XX XX.XX | XX.XXX | XX XX.XX | XX.XXX | xx xx.xx |
| Week 1 | Min, | XX.XX | XX.XXX | XX.XX | XX.XXX | XX.XX | XX.XXX | XX.XX | XX.XXX |
| | Max | xx.x, | XX.XX | XX.X, | XX.XX | xx.x, | XX.XX | xx.x, | XX.XX |
| | | XX.X | XX.X, | XX.X | XX.X, | XX.X | XX.X, | XX.X | XX.X, |
| | ., | XX | XX.X | XX | XX.X | XX | XX.X | XX | XX.X |
| | n Mean | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | SD<br>Median | XX.XXX | XX XX.XX | XX.XXX | XX XX.XX | XX.XXX | XX XX.XX | XX.XXX | XX XX.XX |
| | | XX.XX | XX.XXX | XX.XX | XX.XXX | XX.XX | XX.XXX | XX.XX | XX.XXX |
| | Min, | xx.x, | XX.XX | xx.x, | XX.XX | xx.x, | XX.XX | xx.x, | XX.XX |
| Week 2 | Max | XX.X | XX.X, | XX.X | XX.X, | XX.X | XX.X, | XX.X | XX.X, |
| | | XX | XX.X | XX | XX.X | XX | XX.X | XX | XX.X |
| | n Mean | XX.XX | xx xx.xx | xx.xx | xx xx.xx | xx.xx | xx xx.xx | xx.xx | xx xx.xx |
| | SD | XX.XXX | XX.XXX | xx.xxx | XX.XXX | xx.xxx | XX.XXX | xx.xxx | XX.XXX |
| | Median | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX |
| | Min, | xx.x, | XX.X, | xx.x, | XX.X, | xx.x, | XX.X, | xx.x, | XX.X, |
| | Max | XX.X | XX.X | xx.x | XX.X | xx.x | XX.X | XX.X | xx.x |
| | | XX | | XX | | XX | | XX | |
| Week 4 | n Mean | xx.xx | XX XX.XX | xx.xx | XX XX.XX | xx.xx | XX XX.XX | xx.xx | XX XX.XX |
| | SD Mean | xx.xxx | XX.XXX | xx.xxx | XX.XXX | xx.xxx | XX.XXX | xx.xxx | XX.XXX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min, | XX.X, | XX.X, | XX.X, | XX.X, | XX.X, | XX.X, | xx.x, | XX.X, |
| | , | , | XX.X | , | XX.X | • | XX.X | , | XX.X |

Week 6

<Parameter 1> (unit)

| | | Elamipretide 4 mg<br>(N=xx) | Elamipretide 40 mg (N=xx) | | Placebo (N=xx) | All Subjects (N = xxx) |
|---|---|---|---|---|---|---|
| Parameter<br>(unit)<br>Time Point | | Actual Change From Value<br>Baseline | Actual Change From Value<br>Baseline | Actual<br>Value | Change From<br>Baseline | Actual Change From Value<br>Baseline |
| | Max | xx.x | xx.x | XX.X | | xx.x |

SD = Standard deviation.

[Source: Listinga] Baseline assessment is defined as last assessment prior to the first dose of study medication. 6.1

n represents the number of subjects contributing to summary statistics.

| Parameter | | | Week 1 | | | Week 2 | High | | Week 4 | | | Week 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <pre>(unit) Treatment Group <parameter 1=""> (unit)</parameter></pre> | Baselin<br><u>e</u> | Low<br>n (%) | Normal <u>n</u> (%) | High<br>n (%) | Low | Normal <u>r</u> (%) | <u>n (%)</u> | Low<br>n (%) | Normal<br><u>(%) n (</u> | | Low<br>n (%) | Normal<br><u>(%) n (</u> | |
| | N | | | | n (%) | | | | | | | | |
| Elamipretid | | | | | | | | | | | | | |
| e 4 mg | Low | XX XX | xx | xx | | | xx<br>(xx.x% | XX XX | XX | XX | xx xx | xx | XX |
| | Normal | (xx.x%<br>)<br>xx<br>(xx.x% | (xx.x%<br>)<br>xx | (xx.x%<br>)<br>xx | xx xx<br>(xx.x% | xx<br>(xx.x%<br>)<br>xx | )<br>xx<br>(xx.x% | (xx.x%<br>)<br>xx<br>(xx.x% | (xx.x%<br>)<br>xx | (xx.x%<br>)<br>xx | (xx.x%<br>)<br>xx<br>(xx.x% | )<br>(xx.x% | (xx.x%<br>)<br>xx |
| | High | )<br>xx<br>(xx.x% | (xx.x%<br>)<br>xx | (xx.x%<br>)<br>xx | )<br>xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | )<br>xx<br>(xx.x%<br>) | )<br>xx<br>(xx.x% | (xx.x%<br>)<br>xx | (xx.x%<br>)<br>xx | )<br>xx<br>(xx.x% | )<br>xx | )<br>xx |
| | N | )<br>xx xx<br>(xx.x% | (xx.x%<br>) | (xx.x% | ,<br>(xx.x%<br>) | ) | , | )<br>xx xx<br>(xx.x% | (xx.x%<br>) | (xx.x%<br>) | )<br>xx xx<br>(xx.x% | (xx.x% | (xx.x%<br>) |
| Elamipretid<br>e 40 mg | Low | )<br>XX | | | xx xx | | xx | )<br>xx | | | )<br>xx | | |
| | Normal | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) |
| | High | (xx.x% | xx<br>(xx.x%<br>) | xx<br>(xx.x% | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | (xx.x% | xx<br>(xx.x% | xx<br>(xx.x%<br>) | (xx.x% | xx<br>(xx.x% | xx<br>(xx.x% |
| | N | xx xx<br>(xx.x% | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | (xx.x%<br>) | xx<br>(xx.x% | (xx.x% | xx xx<br>(xx.x% | xx<br>(xx.x%<br>) | ,<br>(xx.x%<br>) | xx xx<br>(xx.x% | xx<br>(xx.x% | xx<br>(xx.x%<br>) |
| | Low | )<br>xx | | | xx xx<br>(*x.xx) | , | xx<br>(xx.x% | )<br>xx | | | )<br>xx | | |
| Placebo | Normal | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | )<br>xx | xx<br>(xx.x%<br>) | )<br>xx | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) |
| | High | (xx.x% | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | xx<br>(xx.x%<br>) | (xx.x%<br>)<br>xx | (xx.x% | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | (xx.x% | xx (xx.x% | xx<br>(xx.x%<br>) |
| | | | xx<br>(xx.x%<br>) | xx<br>(xx.x% | (xx.x%<br>) | xx<br>(xx.x%<br>) | (xx.x% | | xx<br>(xx.x%<br>) | xx<br>(xx.x%<br>) | | xx<br>(xx.x% | xx<br>(xx.x% |
| Report gener | ated hy nr | ogram• /s: | asdir/xxvv | ,<br>, sas | | , | | | , | , | Draft | ,<br>. v v | Y Y |
| -MM-DD HH: | | - <u>5</u> -2 / 50 | , | | | | | | | | 2 2 4 1 | | |

<Parameter 2> (unit)

#### Table 7.1b Shift Table of Hematology Parameters From Baseline to Post Baseline Visits

Safety Population

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

| Parameter | | Week 1 | Week 2 | | Week 4 | | Week 6 | |
|---|---|---|---|---|---|---|---|---|
| (Treatment unit) | | | Low | Normal High | Low | Normal High | Low | Normal High |
| | Baselin | Low Normal High | | J | | , | | - |
| Group | е | n (%) n (%) n (%) | | | n (%) n (% | s) n (%) n (%) n (% | ) n (%) n | (%) n (%) n (%) |

Percentages are based on N, number of subjects with assessment value at both the post-baseline visit and baseline. Source: Listing 6.1

Table 7.2a Change From Baseline in Blood Chemistry Parameters by Visit Safety Population

Note to Programmer: Same layout as Table 7.1a.

Source: Listing 6.2

Table 7.2b
Shift Table of Blood Chemistry Parameters From Baseline to Post Baseline Visits
Safety Population

Note to Programmer: Same layout as Table 7.1b.

Source: Listing 6.2

Table 7.3a Change From Baseline in Urinalysis Parameters by Visit Safety Population

Note to Programmer: Table layout is similar to Table 7.1a. The time points are baseline and Week 4. Only the parameters with continuous values will be presented.

Source: Listing 6.3

Table 7.3b Shift Table of Urinalysis Parameters From Baseline to Post Baseline Visits Safety Population

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

Note to Programmer: Table layout is similar Table 7.1b. Low, Normal, High replaced with Normal and Abnormal. Time points are baseline and Week 4. All the parameters in urinalysis will be presented. Source: Listing 6.3

Table 7. 4a Change From Baseline in Levels of hsTroponin by Visit Safety Population

Note to Programmer: Same layout as Table 7.1a. Include parameters: hsTroponin, Log hsTroponin. For Log hsTroponin, use Log Ratio for Change from Baseline.

Source: Listing 6.4

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM
## 8. ELECTROCARDIOGRAM EVALUATIONS

Table 8.1 Change From Baseline in Electrocardiogram (ECG) Parameters by Visit Safety Population

| | Elami | Elamipretide 4 mg<br>(N=xx) | | Elamipretide 40 mg<br>(N=xx) | | Placebo (N=xx) | | All Subjects (N<br>= xxx) |
|---|---|---|---|---|---|---|---|---|
| Parameter (unit) | Actual | Change From | Actual | Change From | Actual | Change From | Actual | Change From |
| Time Point <parameter 1=""></parameter> | Value | Baseline | Value | Baseline | Value | Baseline | Value | Baseline |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

(unit)

| Baseline[a] | n | xx | | XX | | XX | | xx | |
|---|---|---|---|---|---|---|---|---|---|
| | Mean | XX.XX | | xx.xx | | XX.XX | | XX.XX | |
| | SD | xx.xxx | | xx.xxx | | XX.XXX | | XX.XXX | |
| | Median | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | Min, | XX.X, | | XX.X, | | XX.X, | | XX.X, | |
| | Max | XX.X | | XX.X | | XX.X | | XX.X | |
| | | XX | | XX | | XX | | XX | |
| | ~ | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | n<br>Mean | XX.XXX | | XX.XXX | | XX.XXX | | XX.XXX | |
| r.r 1. 1 | SD | XX.XX | XX XX.XX | XX.XX | XX XX.XX | XX.XX | XX XX.XX | XX.XX | XX XX.XX |
| Week 1 | Median | XX.X, | XX.XXX | xx.x, | XX.XXX | XX.X, | XX.XXX | xx.x, | XX.XXX |
| | Min, | XX.X | xx.xx<br>xx.x, xx.x | XX.X | xx.xx<br>xx.x, xx.x | XX.X | XX.XX<br>XX.X, XX.X | XX.X | xx.xx<br>xx.x, xx.x |
| | Max | | AA.A, AA.A | | AA.A, AA.A | | AA.A, AA.A | | AA.A, AA.A |
| | Мах | XX.XX | XX XX.XX | XX<br>XX.XX | XX XX.XX | XX<br>XX.XX | XX XX.XX | XX.XX | XX XX.XX |
| | n | XX.XXX | XX.XXX<br>XX.XX | XX.XXX | XX.XXX<br>XX.XX | XX.XXX | XX.XXX<br>XX.XX | XX.XXX | XX.XXX<br>XX.XX |
| | Mean | XX.XX | XX.X, XX.X | XX.XX | XX.X, XX.X | XX.XX | XX.X, XX.X | XX.XX | XX.X, XX.X |
| | SD | XX.X, | AA.A, AA.A | XX.X, | AA.A, AA.A | XX.X, | AA.A, AA.A | XX.X, | AA.A, AA.A |
| Week 2 | Median | XX.X | xx xx.xx | XX.X | xx xx.xx | XX.X | xx xx.xx | XX.X | xx xx.xx |
| | Min, | XX | XX.XXX | XX | XX.XXX | XX | XX.XXX | XX | XX.XXX |
| | Max | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | XX.XXX | xx.x, xx.x | XX.XXX | XX.X, XX.X | XX.XXX | XX.X, XX.X | XX.XXX | xx.x, xx.x |
| | | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | n<br>Maara | XX.X, | XX | xx.x, | XX | xx.x, | XX | xx.x, | XX |
| | Mean<br>SD | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| 1 4 | Median | XX | | XX | | XX | | XX | |
| Week 4 | | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| | Min, | | | | | | | | |
| | Max | | | | | | | | |

Week 6

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

n Mean

Draft YYYY


| | | Elami | pretide 4 mg (N= | =xx) Elami | Placebo (N=xx) | All Subjects (N<br>= xxx) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter<br>(unit)<br>Time Point | | Actual<br>Value | Change From<br>Baseline | Actual<br>Value | Change From<br>Baseline | Actual<br>Value | Change From<br>Baseline | Actual<br>Value | Change From<br>Baseline |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Median | XX.XX | XX.XX XX.X, | XX.XX | XX.XX XX.X, | XX.XX | XX.XX XX.X, | XX.XX | xx.xx xx.x, |
| | Min, Max | XX.X, | XX.X | XX.X, | XX.X | XX.X, | XX.X | XX.X, | XX.X |
| | | XX.X | | XX.X | | XX.X | | XX.X | |

SD = Standard deviation. n represents the number of subjects contributing to summary statistics.

[Source: Listinga] Baseline assessment is defined as last assessment prior to the first dose of study medication. 7.2

Report generated by program: /sasdir/xxxx.sas Draft YYYY
-MM-DD HH:MM


### 9. VITAL SIGNS

Table 9.1 Change From Baseline in Vital Signs Safety Population

| | Elamipre | tide 4 n | ng (N=xx) | Elamipre | tide 40 mg ( $N=$ | xx) Pla | ncebo (N=xx) | All S | ubjects (N=xx |
|---|---|---|---|---|---|---|---|---|---|
| | | _ | | | | Actual<br><u>Value</u> | Change From<br>Baseline | Actual<br>Value | Change From Baseline |
| | Actual<br><u>Value</u> | | | Actual<br><u>Value</u> | Change From<br><u>Baseline</u> | | | xx xx.x<br>xx.xx xx.x | |
| n Mean<br>SD<br>Median<br>Min, Max<br>n Mean<br>SD<br>Median<br>Min, Max | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x<br>xx xx.x<br>xx.xx xx.x<br>xx.xx xx.x | xx.x<br>xx.x<br>xx.x | xx<br>xx.xx<br>xx.x, | n Mean<br>SD<br>Median<br>Min, Max<br>n Mean<br>SD<br>Median<br>Min, Max | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x<br>xx xx.x<br>xx.xx xx.x<br>xx.xx xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x |
| n Mean<br>SD<br>Median<br>Min, Max | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx.x<br>xx.x<br>xx.x | xx<br>xx.xx<br>xx.x, | n Mean<br>SD<br>Median<br>Min, Max | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x |
| n Mean<br>SD<br>Median<br>Min, Max | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx<br>xx.xx<br>xx.x, | xx.x<br>xx.x<br>xx.x | n Mean<br>SD<br>Median<br>Min, Max | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x | xx xx.x<br>xx.xx xx.x<br>xx.x, xx.x |
| | SD Median Min, Max n Mean SD Median Min, Max n Mean SD Median Min, Max | n Mean SD | Actual Value N Mean SD XX XX.X Median XX.XX XX.X N Mean XX XX.X SD XX.XX XX.X Median XX.X, XX.X Median XX.X, XX.X Median XX.X, XX.X Median XX.X, XX.X N Mean XX XX.X N Mean XX XX.X N Mean XX XX.X XX XX.X N Mean XX XX.X N Mean XX.X, XX.X XX XX XX.X XX XX XX.X XX XX XX XX.X XX X | Change From Baseline Actual Value Note the proof of th | Change From Baseline Actual Value Actual Value n Mean SD xx xx.x Median xx.xx xx.x Min, Max n Mean xx xx.x xx xx n Mean xx xx.x xx | Change From Baseline Actual Value Change From Baseline N Mean SD XX XX.X SD XX XX.X Median XX.XX XX.X Median XX.XX XX.X Min, Max XX.X, XX.X Min, Max XX.X, XX.X Min, Max XX.X, XX.X Min, Max XX.X, XX.X Min, Max XX.X, XX.X Median XX.X, XX.X XX.X Median XX.X, XX.X Median XX.X, XX.X Min, Max N Mean XX XX.X XX.X XX.X XX.X Median XX.X, XX.X Min, Max N Mean XX XX.X XX.X XX.X XX.X Median XX.X, XX.X XX.X XX.X Min, Max N Mean XX XX.X XX.X XX.X XX.X XX.X Median XX.X, XX.X XX.X XX.X XX.X XX.X XX.X XX | Change From Baseline | Change From Baseline | Change From Baseline |


| Week 6 | n Mean | XX XX.X | | XX | n Mean | XX XX.X | XX XX.X | XX XX.X | XX XX.X | XX XX.X |
|---|---|---|---|---|---|---|---|---|---|---|
| | SD | XX.XX XX.X | XX.X | XX.XX | SD | XX.XX XX.X | XX.XX XX.X | XX.XX XX.X | XX.XX XX.X | XX.XX XX.X |
| | Median | xx.x, xx.x | XX.X | xx.x, | Median | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Min, Max | | xx.x | | Min, Max | | | | | |

| | - | etide 4 mg<br>N=xx) | - | etide 40 mg<br>N=xx) | | acebo<br>N=xx) | | Subjects<br>J=xx) |
|---|---|---|---|---|---|---|---|---|
| Parameter (unit) | | | | | | | | |
| Time | Actual | Change From | Actual | Change From | Actual | Change From | Actual | Change From |
| Point | Value | Baseline | Value | Baseline | Value | Baseline | Value | Baseline |

SD = Standard deviation, BP = Blood pressure.

Note to Programmer: Repeat for Respiration Rate (breaths/min), Systolic BP (mmHg), Diastolic BP (mmHg), and Temperatures(°C)

Draft YYYY


n represents the number of subjects contributing to summary statistics. Source: Listing 7.1

### 10. PHYSICAL EXAMINATION

Table 10.1 Cardiovascular Physical Examination Results by Visit Safety Population

| | Elamipretide 4 mg | Elamipretide 40 mg | Placebo | All Subjects |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=XX) | (N=xx) |
| | n (%) | n (%) | n (%) | n (%) |
| Screening<br>Clinical Significant Abnormality Noted<br>Yes | ( xx.x%)<br>( xx.x%)<br>xx ( xx.x%) | ( xx.xx)<br>( %x.xx)<br>( %x.xx) | ( xx.x%)<br>( xx.x%)<br>xx ( xx.x%) | ( |
| No<br>Not Done | xx<br>xx | xx<br>xx | XX XX | xx xx |
| Baseline Clinical Significant Abnormality Noted Yes No Not Done | ( xx.x%)<br>( xx.x%)<br>xx ( xx.x%)<br>xx | ( xx.x%)<br>( xx.x%)<br>xx ( xx.x%)<br>xx | ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx | xx.x%) ( xx.x%) xx ( xx.x%) xx xx xx |
| eek 1 Clinical Significant Abnormality Noted Yes No Not Done eek 2 | ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx | ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx | ( xx.x%)<br>( xx.x%)<br>xx ( xx.x%)<br>xx xx | xx.x%) xx (xx.x%) xx (xx.x%) xx |
| Clinical Significant Abnormality Noted Yes No Not Done | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | ( |
| eek 4<br>Clinical Significant Abnormality Noted<br>Yes<br>No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (<br>XX XX.X%) |
| eport generated by program: /sasdir/xxxx.sa<br>MM-DD HH:MM | S | | D : | raft YYYY |


| Stealth BioTherapeutics, Inc. Protocol SPIHF-201 | | | Elamipretide™ (MTP-1 | 31 for SC Injection) Page n of N |
|---|---|---|---|---|
| Not Done | xx ( xx.x%)<br>xx ( xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Week 6 Clinical Significant Abnormality Noted Yes No Not Done | xx (xx.x%)<br>xx (xx.x%)<br>xx (xy.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xy.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | (<br>xx xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

% = 100\*n/N, where n = number of subjects in the specific row category and N = number of subjects in the column category. Source: Listing 7.3

( xx.x%)

Table 10.2 Physical Measurement Results by Visit Safety Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Y Y Y Y

Draft

( xx.x%)


| | Elamipretide 4 mg | Elamipretide 40 mg | Placebo (N=xx) | ) All Subjects |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | | (N=xx) |
| Screening | xx xx | | | XX XX |
| Steafth bightifes, the normality Protocol Noted have | (%x.xx)<br>(xx.xx)<br>(%x.xx) | xx xx<br>(xx.x%) xx | $xx$ <b>EXamipretide</b> <sup>TM</sup> (MT) $(xx.x^8)$ $xx$ | P-131 for SC Injection) (xx.x%) xx Page n of N (xx.x%) |
| Not Done | | (xx.x%) xx<br>(xx.x%) | (xx.x%) xx<br>(xx.x%) | |
| | XX | XX | xx | xx |
| Weight (kg) | XX.X | XX.X | XX.X | XX.X |
| n | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | xx, xx | xx, xx | xx, xx | XX, XX |
| Median<br>Min, Max | | | | |
| Height (cm) | xx | xx | xx | xx |
| n | xx.x | XX.X | XX.X | xx.x |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX, XX | XX, XX | XX, XX | XX, XX |
| Min, Max | | | | |
| | xx | XX | xx | xx |
| Body Mass Index (kg/m2) | XX.X | XX.X | XX.X | xx.x |
| n | xx.xx | XX.XX | XX.XX | XX.XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | xx, xx | XX, XX | xx, xx | xx, xx |
| Median | | | | |
| Min, Max | | | | |
| Baseline | xx xx | xx xx | xx xx | xx xx |
| Clinical Significant Abnormality | (xx.x%) xx | (xx.x%) xx | (xx.x%) xx | (xx.x%) xx |
| Noted n Yes | (xx.x%) xx | (xx.x%) xx | (xx.x%) xx | (xx.x%) xx |
| No | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Not Done | | | | |
| Weight (kg) | XX | XX | XX | XX |
| n | XX.X | XX.X | XX.X | XX.X |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | | | | |
| Median | XX.X | XX.X | XX.X | XX.X |

Draft YYYY

Report generated by program: /sasdir/xxxx.sas

-MM-DD HH:MM

| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
|---|---|---|---|---|
| Week 1 Clinical Significant Abnormality Noted | | | | |
| | | xx xx | xx xx | XX XX |
| n<br>Wasan | XX | (xx.x%) | (xx.x%) | (xx.x%) |
| Yes | xx (xx.x%) | xx | XX | XX |
| No | xx (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Not Done | xx (xx.x%) | xx | xx | XX |
| Weight (kg) | | (xx.x%) | (xx.x%) | (xx.x%) |
| n xx Mean xx.x | SD | XX | xx | XX |
| XX.XX | | XX.X | XX.X | XX.X |
| Median | XX.X | xx.xx | xx.xx | XX.XX |
| Min, Max | xx, xx | XX.X | XX.X | XX.X |
| Week 2 | | xx, | xx, | XX, |
| Clinical Significant Abnormality Noted | l | xx | xx | XX |
| n | XX | | | |
| Yes | xx (xx.x%) | | | |
| No | xx (xx.x%) | XX XX | XX XX | XX XX |
| Not Done | xx (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| | XX (XX.X%) | XX | XX | XX |
| Weight (kg) | a.p. | (xx.x%) | (xx.x%) | (xx.x%) |
| n xx Mean xx.x | SD | XX | XX | XX |
| XX.XX | | (xx.x%) | (xx.x%) | (xx.x%) |
| Median | XX.X | XX | XX | XX |
| Min, Max | xx, xx | XX.X | XX.X | XX.X |
| Week 4 | | XX.XX | XX.XX | XX.XX |
| Clinical Significant Abnormality Noted | l | XX.X | XX.X | XX.X |
| n | XX | XX, | XX, | XX, |
| Yes | xx (xx.x%) | XX | XX | XX |
| No | xx (xx.x%) | | | |
| Not Done | xx (xx.x%) | xx xx | xx xx | xx xx |
| Weight (kg) | | (xx.x%) | (xx.x%) | (xx.x%) |
| n xx Mean xx.x | SD | XX | XX | XX XX |
| XX.XX | | (xx.x%) | (xx.x%) | (xx.x%) |
| Median | XX.X | XX | XX | XX XX |
| Min, Max | xx, xx | (xx.x%) | (xx.x%) | (xx.x%) |
| Week 6 | m, m | XX | XX | XX XX |
| Clinical Significant Abnormality Noted | | XX.X | XX.X | XX.X |
| n | | XX.XX | XX.XX | XX.XX |
| | XX | XX.X | XX.X | XX.X |
| Yes | xx (xx.x%) | XX, | XX, | XX, |
| No | xx (xx.x%) | XX | XX | XX |
| | | ΛΛ | AA | AA |
| | | XX XX | XX XX | xx xx |
| | | (xx.x%) | (xx.x%) | (xx.x%) |


Stealth BioTherapeutics, Inc. Protocol SPIHF-201

Elamipretide  $^{\mathbb{T}M}$  (MTP-131 for SC Injection) Page n of N

 $\begin{array}{cccc} xx & & xx & & xx \\ (xx.x\%) & & (xx.x\%) & & (xx.x\%) \end{array}$ 

Draft YYYY

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM


| Not Done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|
| | Weight (kg) | n xx | XX XX | xx Mean |
| XX.X XX.X XX.X | xx.x SD xx.xx xx.xx | xx.xx xx.xx Median xx.x | XX.X XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX |

% = 100\*n/N, where n = number of subjects in the specific row category and N = number of subjects in the column category. Source: Listing 7.3

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


#### 11. CONCOMITANT MEDICATIONS/TREATMENTS

Table 11.1 Concomitant Medications by ATC and Preferred Drug Name Safety Population

| Elamipretide 4 mg (N=xx) | Elamipretide 40 mg<br>(N=xx) | Placebo (N=xx) | All Subjects<br>(N=xx) |
|---|---|---|---|
| n (응) | n (응) | n (응) | n (%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| (xx.x%) xx<br>(xx.x%) | (xx.x%) xx<br>(xx.x%) | (xx.x%) xx<br>(xx.x%) | (xx.x%) xx (xx.x%) |
| xx (xx.x%) xx<br>(xx.x%) xx | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) | xx (xx.x%) xx<br>(xx.x%) xx<br>(xx.x%) |
| | (N=xx) n (%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xx) (N=xx) n (%) n (%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xx) (N=xx) n (%) n (%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) |

ATC = Anatomic-Therapeutic-Chemical 3 Classification code.

[a] Preferred drug name via the World Health Organization Drug Dictionary (WHO-DD).

Percentages are based on N.

Included any medications taken during the study (from the date of first dose of investigational product to the date of last visit). Source: Listing 3.2

Note to Programmer: ATCs sorted alphabetically. All medications will be sorted alphabetically by medication class and medication subclass.

#### LISTINGS

### LISTINGS – SUBJECT DISPOSITION, DEMOGRAPHICS, AND BASELINE CHARACTERISTICS

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Listing 1.1
Study Completion or Early Discontinuation Status
All Randomized Subjects

| Subject<br>ID | Age/Sex[a] | Date of Randomization/ Treatment Assigned | Study Drug<br>Administered | Treatment<br>Start/End<br>Date | Study Completion Status/ Last Study Date [b] (Study Day) [c] | Reason for Early Discontinuation | Included in Safety/ITT/Per Protocol Population? |
|---|---|---|---|---|---|---|---|
| xxx-xxx<br>xxx-xxx<br>xxx-xxx<br>xxx-xxx | 73/F<br>66/M 69/F<br>xx/X xx/X | yyyy-mmm-dd Elamipretide 4 mg yyyy-mmm-dd Elamipretide 40 mg yyyy-mmm-dd Elamipretide 4 mg yyyy-mmm-dd Placebo yyyy-mmm-dd Placebo | Elamipretide 4 mg Elamipretide 40 mg Elamipretide 40 mg Placebo Placebo | yyyy-mmm-dd/<br>yyyy-mmm-dd/<br>yyyy-mmm-dd/<br>yyyy-mmm-dd/<br>yyyy-mmm-dd/<br>yyyy-mmm-dd/ | Completed yyyy-mmm-dd (xxx) Discontinued yyyy-mmm-dd (xxx) Discontinued yyyy-mmm-dd (xxx) Discontinued yyyy-mmm-dd (xxx) Discontinued yyyy-mmm-dd (xxx) Discontinued yyyy-mmm-dd (xxx) | Adverse event Sponsor decision, specific reason Withdrawal of consent Investigator reason, specific reason | Yes/Yes/Yes Yes/Yes/No No/No/No No/No/No Yes/Yes/No |

<sup>[</sup>a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Treatment Group and Subject ID.

Listing 1.2 Violations of Inclusion/Exclusion Criteria All Subjects

| Informed Consent | Date Informed | Satisfied All Inclusion/ | |
|---|---|---|---|
| Subject ID Form Signed | Consent Signed | Exclusion Criteria | Inclusion/Exclusion Criteria Failed |

Report generated by program: /sasdir/xxxx.sas

Draft YYYY

-MM-DD HH:MM

<sup>[</sup>b] Last Study Date = date of last visit.

<sup>[</sup>c] Study Day = study date - date of randomization + 1.

Elamipretide  $^{\text{TM}}$  (MTP-131 for SC Injection) Page n of N

xxx-xxx Yes yyyy-mmm-dd No INCL. # 3, EXCL # 6, Other: xxxxxxxx
xxx-xxx Yes yyyy-mmm-dd Yes

Note to Programmer: Listing is sorted by Randomized Treatment Group and Subject ID.

## Listing 1.3 Randomization Status All Subjects

| Subject ID | Randomized? | Randomized Treatment Assignment | Randomization Number | Randomization Date | Reason not Randomized |
|---|---|---|---|---|---|
| xxx-xxx | Yes | Elamipretide 4 mg | xxxxx | yyyy-mmm-dd | Reason not Randomized |
| xxx-xxx | No | | | 7777 | xxxxxxxxxxxxxxxxx |

Note to Programmer: Listing is sorted by Subject ID.

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Listing 1.4 Demographic Information All Randomized Subjects

| ignment Age/Sex | [a] Race | Ethnicity | (cm) | (kg) | (kg/m2) |
|---|---|---|---|---|---|
| mipretide | | | | | |
| g 73/F | White | Hispanic or Latino | xxx.x | xxx.x | xx.x |
| cebo 66/M | Black | Not Hispanic or Latino | xxx.x | xxx.x | xx.x |
| ıç | 73/F | 73/F White | 73/F White Hispanic or Latino | 73/F White Hispanic or Latino xxx.x | 73/F White Hispanic or Latino xxx.x xxx.x |

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group and Subject ID.

Listing 1.5
Medical and Surgical History
All Randomized Subjects

| Subject<br>ID | Randomized<br>Treatment Age/Se<br>Assignment [a] | Any<br>Medical/<br>x Surgical<br>History | Category | Diagnosis or<br>Surgery | Start Date | Is Condition Still<br>Present at<br>Screening? | End Date |
|---|---|---|---|---|---|---|---|
| xxx-xxx | Elamipretide 73/F 4 mg | Yes | Drug Allergy | xxxxxxxx | yyyy-mmm-dd | No | yyyy-mmm-dd |
| xxx-xxx | Elamipretide 66/M<br>40 mg | Yes | Hepatic<br>Psychiatric | xxxxxxxx | уууу-mmm-dd<br>уууу-mmm-dd | Yes<br>No | yyyy-mmm-dd |
| xxx-xxx Pla | acebo 78/F | No | | | | | |

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group and Subject ID.

## LISTINGS – EFFICACY

Listing 2.1

Cardiac MRI Assessments – Actual and Change from Baseline Values
ITT Population

Draft YYYY


| | oTherapeutics,In | | | $	extsf{Elamipretide}^{	extsf{TM}}$ | (MTP-131 for SC | |
|---|---|---|---|---|---|---|
| _ | PIFFeathlent | Age/Sex | 771 - 1 to - 4 - to - | Davidada | 77 - 7 | Pa(\$6 se 19 fie) |
| ID | Assignment [a] | Visit | Visit date | Parameter | Value | value) |
| xxx-xxx | Elamipretide | Screening | yyyy-mmm-dd | Left Ventricular End Systolic Volume | XXX.XX | |
| | | | | Left Ventricular End Systolic Volume ( | LV xxx.xx xxx.x | X |
| | | | | ESV), Indexed by BSA | | |
| | | | | Left Ventricular Ejection Fraction (LVEF) | XXX.XX XXX.XX | X |
| | | | | Left Ventricular End Diastolic Volume (LV EDV) | XXX.XX XXX.XX | X |
| | | | | Left Ventricular End Diastolic Volume (LV EDV), Indexed by BSA | xxx.xx xxx.x | |
| | | | | Left Ventricular Myocardial Mass (LV | xxx.xx xxx.x | X |
| | | | | Mass) | XXX.XX XXX.XX | X |
| | | | | Left Ventricular Myocardial Mass (LV Mass), Indexed by BSA | xxx.xx xxx.x | X |
| | | | | Left Ventricular Stroke Volume (LVSV)<br>Left Ventricular Cardiac Output (LVCO) | xxx.xx | |
| | | | | Right Ventricular End Systolic Volume | Xxxxxx | |
| | | | | (RV ESV) | XXX.XX | |
| | | | | Right Ventricular End Systolic Volume | XXX.XX | |
| | | | | (RV ESV), Indexed by BSA Right Ventricular End Diastolic Volume (RV EDV) | xxx.xx | |
| | | | | Right Ventricular End Diastolic Volume | | |
| | | | | (RV EDV), Indexed by BSA<br>Right Ventricular Myocardial Mass (RV | | |
| | | | | Mass) | | |
| | | | | Right Ventricular Myocardial Mass (RV Mass), Indexed by BSA | | |
| | | | | Right Ventricular Ejection Fraction | | |
| | | | | (RVEF) | | |
| | | | | Ischemic/Non-ischemic Status | | |
| | | | | LV ESV | | |
| | | | | LV ESV, Indexed by BSA | | |
| | | | | LVEF | | |
| | | | | | | XXX.XX |
| | | 1 1 | yyyy-mmm-dd | | | xxx.xx |
| | | Week 1 | | | | |
| | 4 | 70/5 | | (TM DOM) | | |
| | 3 | 73/F | | (LV ESV) | _ | |
| | enerated by progr<br>HH:MM | ram: /sasdir/xxxx.sas | | | Draft | YYYY |


| LV EDV | XXX.XX | XXX.XX |
|-------------------------|--------|--------|
| LV EDV, Indexed by BSA | XXX.XX | XXX.XX |
| LV Mass | XXX.XX | XXX.XX |
| LV Mass, Indexed by BSA | XXX.XX | XXX.XX |
| LVSV | XXX.XX | XXX.XX |
| LVCO | XXX.XX | XXX.XX |
| RV ESV | XXX.XX | XXX.XX |
| RV ESV, Indexed by BSA | XXX.XX | XXX.XX |
| RV EDV | XXX.XX | XXX.XX |
| | XXX.XX | XXX.XX |
| RV EDV, Indexed by BSA | XXX.XX | XXX.XX |
| RV Mass | XXX.XX | XXX.XX |
| RV Mass, Indexed by BSA | XXX.XX | XXX.XX |
| RVEF | XXX.XX | XXX.XX |
| LV ESV | XXX.XX | XXX.XX |
| LV ESV, Indexed by BSA | XXX.XX | XXX.XX |
| LVEF | XXX.XX | XXX.XX |
| LV EDV | XXX.XX | |
| LV EDV, Indexed by BSA | XXX.XX | XXX.XX |
| LV Mass | XXX.XX | XXX.XX |
| LV Mass, Indexed by BSA | XXX.XX | |
| LVSV | XXX.XX | XXX.XX |
| LVCO | XXX.XX | |
| RV ESV | XXX.XX | XXX.XX |
| | XXX.XX | XXX.XX |
| RV ESV, Indexed by BSA | XXX.XX | |
| RV EDV | XXX.XX | XXX.XX |
| RV EDV, Indexed by BSA | XXX.XX | |
| RV Mass | XXX.XX | XXX.XX |
| RV Mass, Indexed by BSA | | |
| RVEF | | |

yyyy-mmm-dd

Week 4

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

XXX-

Elamipretide 40 mg 65/M Screening

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date. Ischemic/Non-ischemic status only needs to be reported at Screening.

Listing 2.2

Draft YYYY


## Echocardiography Assessments- Actual and Change from Baseline Values ITT Population

| Subject 1 | Treatment | Age/Sex | | | | Change fro |
|---|---|---|---|---|---|---|
| xxx-xxx | Elamipretide | 73/F 4 | Screening | yyyy-mmm-dd | E/A (Ratio Between Early And Late Mitral xxx.xx | xxx.xx |
| | mg | | | | Inflow Velocity)<br>E/e' (Ratio Between Early Mitral<br>Inflow Velocity and Mitral Annular Early | xxx.xx |
| | | | | | Diastolic Velocity) Left Ventricular End Systolic Volume (LV ESV) | xxx.xx |
| | | | | | Left Ventricular End Systolic Volume<br>(LV ESV), Indexed by BSA<br>Biplane Ejection Fraction (EF) | |
| | | | | | Left Ventricular End Diastolic Volume xxx.xx (LV EDV) | xxx.xx |
| | | | | | Left Ventricular End Diastolic Volume (LV EDV), Indexed by BSA | xxx.xx |
| | | | | | Left Ventricular Global Longitudinal<br>Strain (LV GLS)<br>Left Atrial Volume (LAV) | |
| | | | | | Left Atrial Volume (LAV), Indexed by XXX.XX BSA Left Ventricular Mass (LVM) | xxx.xx |
| | | | | | Left Ventricular Mass (LVM), Indexed by BSA Mitral Regurgitation Severity (MRS) | xxx.xx |
| | | | | | Tricuspid Regurgitation Severity (TRS) Right Ventricular Fractional Area | xxx.xx |
| | | | | | Change (RV FAC) | xxx.xx |
| | | | | | Right Ventricular Systolic Pressure (RVSP) | xxx.xx |
| | | | | | E/A<br>E/e' | |
| | | | | | LV ESV | xxx.xx |
| | | | | | LV ESV, Indexed by BSA | xxx.xx |
| | | | | | EF | XXX.XX |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Elamipretide  $^{\text{TM}}$  (MTP-131 for SC Injection) Page n of N

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

| Baseline | | LV EDV<br>LV EDV, Indexed by BSA | xxx.xx ID |
|----------|-------------|----------------------------------|-----------|
| | yyyy-mmm-dd | LV GLS | XXX.XX |
| | | LAV | XXX.XX |
| | | LAV, Indexed by BSA | XXX.XX |
| | | LVM | XXX.XX |
| | | LVM, Indexed by BSA | XXX.XX |
| | | MRS | XXX.XX |
| | | | XXX.XX |
| | | | XXX.XX |

Assignment [a] Visit Visit date Parameter Value Baseline

| | | TRS | XXX.XX | |
|-------------|-------------|------------------------|--------|--------|
| | | RV FAC | XXX.XX | |
| | | RVSP | XXX.XX | |
| | | E/A | xxx.xx | |
| | | E/e' | xxx.xx | xxx.xx |
| | уууу-mmm-dd | LV ESV | xxx.xx | XXX.XX |
| ToTa a la 1 | | | xxx.xx | XXX.XX |
| Week 4 | | LV ESV, Indexed by BSA | xxx.xx | XXX.XX |
| | | EF | xxx.xx | XXX.XX |
| | | LV EDV | xxx.xx | XXX.XX |
| | | LV EDV, Indexed by BSA | xxx.xx | XXX.XX |
| | | LV GLS | xxx.xx | xxx.xx |
| | | LAV | xxx.xx | XXX.XX |
| | | LAV, Indexed by BSA | xxx.xx | XXX.XX |
| | | LVM | XXX.XX | xxx.xx |
| | | LVM, Indexed by BSA | XXX.XX | xxx.xx |
| | | MRS | XXX.XX | XXX.XX |
| | | TRS | XXX.XX | XXX.XX |
| | | RV FAC | XXX.XX | XXX.XX |
| | | RVSP | xxx.xx | XXX.XX |
| | | E/A | xxx.xx | XXX.XX |
| | | E/e' | xxx.xx | XXX.XX |
| | | LV ESV | xxx.xx | XXX.XX |
| | | | XXX.XX | XXX.XX |
| | | LV ESV, Indexed by BSA | XXX.XX | XXX.XX |
| | | EF | XXX.XX | XXX.XX |
| | | LV EDV | XXX.XX | XXX.XX |
| | | LV EDV, Indexed by BSA | xxx.xx | XXX.XX |
| | | LV GLS | xxx.xx | XXX.XX |
| | 1.1 | LAV | xxx.xx | XXX.XX |
| | yyyy-mmm-dd | LAV, Indexed by BSA | XXX.XX | XXX.XX |
| | | LVM | XXX.XX | XXX.XX |
| | | LVM, Indexed by BSA | XXX.XX | XXX.XX |
| Week 6 | | MRS | XXX.XX | XXX.XX |
| | | TRS | XXX.XX | XXX.XX |
| | | RV FAC | | XXX.XX |
| | | RVSP | | |
| | | LVOL | | |

XXX-

Elamipretide 65/M 40 mg Screening

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

## Listing 2.3 Exploratory Assessments – Actual and Change from Baseline Values ITT Population

| | | | | | | | Was a 6MWT |
|---|---|---|---|---|---|---|---|
| Subjec | t Treatment | Age/Se | X | | | Change from | performed? |
| ID | Assignment | [a] | Visit | Visit date Parameter | Value | Baseline [b] | [c] |

| xxx-xxx | Elamipretide<br>4 mg | 73/F | Baseline | yyyy-mmmdd | | | | Yes |
|---|---|---|---|---|---|---|---|---|
| Stealth Bi<br>Protocol S | OTherapeutics, | Inc. | | | Distance Walked (meters) During 6-minute Walking Test (6MWT) Levels of NT-pro-BNP (Log value) Kansas City Cardiomyopathy Questionnaire (KCCQ) Score | xRkamipretide™<br>xxx.xx<br>(xx.xx)<br>xxx.xx | (MTP-131 for SC | C Injection)<br>Page n of N |
| | | | Week 1 | yyyy-mmmdd | NT-pro-BNP (Log value) | xxx.xx (xx.xx) | xxx.xx (xx.xx) | |
| | | | Week 2 | yyyy-<br>mmmdd | NT-pro-BNP (Log value) | xxx.xx<br>(xx.xx) | xxx.xx<br>(xx.xx) | |
| | | | Week 4 | уууу-mmmdd | 6MWT | | | No |
| | | | | | NT-pro-BNP (Log value) | xxx.xx | xxx.xx | |
| | | | | | KCCQ | xxx.xx<br>(xx.xx)<br>xxx.xx | xxx.xx<br>(xx.xx)<br>xxx.xx | |
| | | | Week 6 | yyyy-mmmdd | NT-pro-BNP (Log value) | xxx.xx (xx.xx) | xxx.xx (xx.xx) | |
| xxx-xxx | Elamipretide<br>40 mg | 65/M | Baseline | | | | | |

<sup>[</sup>a] Age is age at informed consent. Sex: M = Male, F = Female.

## Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

## Listing 2.4.1 Six-Minute Walk Test – Part I ITT Population

| Subje ct Assignment ID t | | | УУУ<br>ymmm<br>-dd | | | tal<br>oxygen<br>used | O2<br>Flo<br>w, | | М | Pressu<br>re<br>(mmHg) | Rate<br>(beat<br>s/ | (breaths / min) | (%<br>) | (Borg<br>) | (Borg |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Age/S<br>ex<br>[a] | <u>Visit</u><br>Baseli<br>ne | Vis<br>it<br>dat<br><u>e</u> | Was a 6MWT perform ed? Yes | If No,<br>Reason | Supplemen | If<br>Yes | Tim<br><u>e</u><br>Pre | Vita<br>ls<br><u>Time</u><br>HH:M | Blood | Heart | Respirat<br>ory Rate | Sp<br>O2 | Dyspn<br>ea | Fatio |

Report generated by program: /sasdir/xxxx.sas

-MM-DD HH:MM

<sup>[</sup>b] Log ratio for log-transformed parameters.

<sup>[</sup>c] Assessed only at Baseline and Week 4.

| ${\tt Elamipretide^{\tt TM}}$ | (MTP-131 | for | SC | Inje | ect | cio | า) |
|-------------------------------|----------|-----|----|------|-----|-----|----|
| | | | ī | Page | n | ٥f | N |

| xxxxx | Elamipret<br>ide 4 mg | | | | | | during<br>test? Yes | Typ exx. x, xxx xxx | xxx/xx<br>x | min)<br>xxx | xx | xx<br>x | xx.x | xx.x |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Elamipret<br>ide 40 mg | 65/M | Week 4 Baseli | УУУ<br>ymmm<br>-dd | No | New<br>unstab<br>le<br>angina<br>or MI | No | | | | | | | |

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

Listing 2.4.2 Six-Minute Walk Test – Part II ITT Population

Subje

ct

Sit If

Subject at Yes, Any Any

Experience If any Time Interruptio Clinically

Vis Sta Sto Total any If Other Point Subje n Require Significan Treatment Age/S it rt p Distan Interrupti Yes, , Durin ct Discontinua t Subje Assignmen ex dat Tim Tim Tim ce ons During Reas Speci g First tion of Abnormalit ct ID t [a] Visit e e e e Walked 6MWT? on fy Test? Sat 6MWT? ies Noted?

xxx- Elamipret Baseli yyy Pre HH: HH: xxx Yes Leg Yes HH:MM Yes
xxx ide 4 mg ne y- MM MM Cram mmm
ps

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft

YYYY

Stealth BioTherapeutics, Inc. Protocol SPIHF-201

Elamipretide  $^{\text{TM}}$  (MTP-131 for SC Injection) Page n of N

73/F -dd

Week 4 yyy Pos HH: HH: xxx No y- t MM MM mmm dd

Elamipret Baseli xxx ide 40 mg 65/M ne

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

## Listing 2.5.1 Kansas City Cardiomyopathy Questionnaire – Page 1 ITT Population

| | | Activity |
|---|---|---|
| Subject Treatment Assignment [a] xxx-xxx Elamipretide 4 mg | Block | Carrying Without ID or Jogging Weeks Ago, |
| | Week 4 yyyy- Moderately mmmdd Limited Baseline | Much<br>Better |
| xxx-xxx Elamipretide<br>40 mg | 65/M | Not at All<br>Limited |

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

Listing 2.5.2
ITT Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


#### Elamipretide $^{\text{TM}}$ (MTP-131 for SC Injection) Page n of N

| Subject<br>ID | Treatment<br>Assignment | Age/Sex<br>[a] | Visit | | Many Times Visitve date Swelling? | _ | How Many Times<br>Has Fatigue<br>Limited Your<br>Ability? | How Much Has<br>Fatigue<br>Bothered You? | How Many Times Has Shortness of Breath Limited Your Ability? |
|---|---|---|---|---|---|---|---|---|---|
| xxx-xxx | Elamipretide<br>4 mg | 73/F | Baseline | yyyymmmdd | Every morning | Quite a bit bothersome | All of the time | Quite a bit bothersome | All of the time |
| | | | Week 4 | yyyymmmdd | 1-2 times a week | Slightly<br>bothersome | Less than once<br>a week | Slightly<br>bothersome | Less than once<br>a week |

xxx-xxx Elamipretide Baseline 40 mg 65/M

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

Listing 2.5.3
ITT Population

sdir/xxxx.sas Draft YYYY -MM-DD HH:MM

| Subject<br>ID | Treatment<br>Assignment | Age/Sex<br>[a] | Visit | Sh | ortness of<br>eath<br>Bothered | How Many Times Forced Ptb31515mp SC I: Sitting Up Par Because of Shortness of Breath? | How Sure Are<br>nfwotfingt You<br>goingwoffingt to<br>Do if Heart<br>Failure Gets<br>Worse? | Understand What Things You are Able to Do to Keep Heart Failure Symptoms from Getting Worse? | | If You Had to<br>Spend the<br>Rest of Your<br>Life with<br>Heart<br>Failure, How<br>Would You<br>Feel? |
|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxx | Elamipretide<br>4 mg | 73/F | Baseline | yyyymmmdd | Quite a bit<br>bothersome | Every night | Not very<br>sure | Somewhat<br>understand | It has<br>limited my<br>enjoyment<br>of life<br>quite a bit | Mostly<br>dissatisfied |
| | | | Week 4 | yyyymmmdd | Slightly<br>bothersome | 1-2 times a week | Mostly sure | Mostly<br>understand | It has slightly limited my enjoyment of life | Mostly<br>satisfied |

xxx-xxx Elamipretide Baseline 40 mg 65/M

sdir/xxxx.sas

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

# Listing 2.5.4 Kansas City Cardiomyopathy Questionnaire – Page 4 ITT Population

| Treatment | Age/Se | X | | Activity |
|------------|--------|-------|----------------|----------|
| Assignment | [a] | Visit | How Often Have | |

Draft YYYY -MM-DD HH:MM

#### Elamipretide $^{\mathbb{T}\!M}$ (MTP-131 for SC Injection) Page n of N

| Subject ID xxx- xxx | Elamipretide<br>4 mg | 73/F | Baseline | e Visit<br><u>date</u><br>yyyymmmdd | You Felt<br>Discouraged? | Hobbies, Recreational Activities Severely Limited | Working or<br>Doing Household<br>Chores of Your | Visiting Family<br>d or Friends Out Re<br>Home with Loved | lationships |
|---|---|---|---|---|---|---|---|---|---|
| | | | Week 4 | | | | Limited | Moderately | |
| xxx-xxx | Elamipretide<br>40 mg | 65/M | Baseline | yyyymmmdd | | | | | Did not limit<br>at all |

<sup>[</sup>a] Age is age at informed consent. Sex: M = Male, F = Female.

Draft YYYY -MM-DD HH:MM

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.


sdir/xxxx.sas

Listing 2.5.5
Kansas City Cardiomyopathy Questionnaire – Summary Scores ITT Population

| | | Sympt | | | Overal Clinic |
|---|---|---|---|---|---|
| | Sympt | om Symptom om | Total Self- | Quali | l al |
| Age/S | Visi Physical Stabili | Frequen Burde | Sympt Effica | ty of Social | Summar Summar |
| ıbje Treatment ex | t Limitati ty | cy n | om cy | Life Limitat: | i y y |
| ID Assignment [a] Visit | date on Score Score | | Score Score | Score on | Score Score Score |
| xx- Elamipreti Baseli yyyy | xxx de 4 mg ne - | | | = | |
| | mmm- | | | | |
| 73/F | dd | | | | |
| Mook | 4 уууу | | | | |
| week | mmmdd | | | | |
| | minida | | | xxx- Elami | ipreti |
| aseli | | | xxx de 40 mg | 65/M ne | rprecr |
| 32011 | | | AAA de 40 mg | 03/M He | |

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Randomized Treatment Group, Subject ID, and Visit Date.

#### LISTINGS - STUDY DRUG AND PRIOR/CONCOMITANT MEDICATIONS

Listing 3.1 Study Drug Injection Records Safety Population

If Incomplete Injection,

Total Volume

Vial Any

Injected (mL, Reason(s) for

Entire

Subject Study Drug Dose Number(s) Date of Time of Incomplete % of Incomplete Dose ID Treatment Injected (mg) Used Injection Injection Injections? Expected) Injection Injected xxx-xxx Elamipretide Yes xxx.xx xxxx- yyyy-mmm- hh:mm Yes 0.5 mL, 50% xxxxxxxxxxxx Yes

XXXX,

xxxx-xxxx

xxx-xxx Placebo No,

Reason: XXXXXX

Study

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft Y Y Y Y

### Note to Programmer: Listing is sorted by Randomized Treatment Group and Subject ID.

Listing 3.2
Prior and Concomitant Medications by Subject
Safety Population

| Subject<br>ID | Study<br>Treatment | Age/Sex | Medication<br>Class/Preferred<br>Term<br>(Investigator<br>Text) | Reason | Dose | Unit | Route | Frequency | Prior/<br>Concomita<br>nt[b] | Start Date<br>End Date /<br>Ongoing | Date of<br>First dose<br>of Study<br>Treatment |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx-xxx | Elamipret<br>ide 4 mg | 73/F | XXXXXXXXXXX<br>(XXXXXXXXXXX)<br>XXXXXXXXXXXX | xxxxxx | xxxxx | xxxxx | xxxxx | xxx | Y/N | yyyy-mmm-dd<br>Ongoing | yyyy-mmm-dd |
| | | | (XXXXXXXXXX) | XXXXXX | xxxxx | xxxxx | xxxxx | xxx | N/Y | yyyy-mmm-dd<br>yyyy-mmm-dd | yyyy-mmm-dd |
| xxx-xxx | Placebo | 65/M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxx | xxxxx | xxxxx | xxxxx | XXX | Y/Y | уууу-mmm-dd<br>уууу-mmm-dd | уууу-mmm-dd |

<sup>[</sup>a] Age is age at informed consent. Sex: M = Male, F = Female.

Concomitant = any medications taken during the study (from the date of first dose of investigational product to the date of last visit).

Note to Programmer: Listing is sorted by Study Treatment, Subject ID

#### LISTINGS - PLASMA CONCENTRATION

Listing 4.1
Plasma Concentrations of Elamipretide and Metabolites (M1, M2)
Safety Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

<sup>[</sup>b] Prior = any medications taken prior to the date of first dose of investigational product.
| | | | | | Pl | asma Concentrati | ion (unit) |
|---|---|---|---|---|---|---|---|
| Subject ID | Treatment Assignment | Age/Sex [a] | Date | Time label | Elamipretio | le M1 | M2 |
| xxx-xxx | Elamipretide 4 mg | 73/F | yyyy-mmm-dd | Day 1 Pre-dose | XXX.XX | XXX.XX | XXX.XX |
| | | | | Day 1 Post-dose | xxx.xx | XXX.XX | XXX.XX |
| | | | | Week 1 Pre-dose | xxx.xx | xxx.xx | xxx.xx |
| | | | | Week 1 Post-dose | xxx.xx | xxx.xx | xxx.xx |
| | | | | Week 2 Pre-dose | xxx.xx | xxx.xx | xxx.xx |
| | | | | Week 2 Post-dose | xxx.xx | xxx.xx | xxx.xx |
| | | | | Week 4 | xxx.xx | xxx.xx | xxx.xx |
| | | | | Week 6 | xxx.xx | xxx.xx | xxx.xx |

xxx-xxx

Elamipretide 40 mg

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Subject ID, Visit Date, and Time.

### LISTINGS – ADVERSE EVENTS

Listing 5.1 Adverse Events Safety Population

| | | | System Organ | Onset Date | | Treatment : | for | |
|---|---|---|---|---|---|---|---|---|
| | | | Class/Preferred | (Study day)/ | | AE? | | |
| | | Age/ | Term | Resolution | Intensity/ | Medication | Action | |
| Subject | Study | Sex | (Investigator | Date(Study Day)/ | Relationship | or | Taken with | Serious |
| ID | Treatment | [a] | Term) | ongoing [b] | to Study Drug Outcome | Procedure : | Study Drug | AE [c] |

Draft YYYY


| xxx-xxx | Elamipretide<br>4 mg | 73/F | ************************************** | yyyy-mmm-dd<br>(xxx) yyyy-<br>mmm-dd (xxx) | Severe<br>Probably<br>related | Recovered/Resolved | Yes<br>Medica | Interrupted<br>ation | Yes |
|---|---|---|---|---|---|---|---|---|---|
| | | | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | yyyy-mmm-dd<br>(xxx) ongoing | Severe<br>Unlikely<br>related | Not recovered/not resolved | Yes | None Procedure | No |
| xxx-xxx | Placebo | 65/M | xxxxxxxxxx<br>xxxxxxxxx<br>(xxxxxxxxx) | yyyy-mmm-dd (xxx)<br>yyyy-mmm-dd (xxx)<br>yyyy-mmm-dd (xxx) | xxxxx<br>xxxxxxxxxx | xxxx/xxxx xxxxxxxx | xxx | xxxxxxxx | xxx xxx |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | yyyy-mmm-dd<br>(xxx) | xxxxx/<br>xxxxxxxxxx | | | xxxxxxx | |

Note to Programmer: Listing is sorted by Subject ID, AE Onset Date.

Listing 5.2 Serious Adverse Events Safety Population

| Subject | Study | Age/ | System Organ<br>Class/Preferred<br>Term<br>(Investigator | Onset Date (Study day)/Resolution Date(Study Day)/ | Intensity/ Relationship t Study Drug/Dat of last study treatment prior to the event | Treatment f<br>AE?<br>Medication<br>or | or Action Taken with Study | Seriousness<br>criteria |
|---|---|---|---|---|---|---|---|---|
| ID | Treatment | Sex [a] | Term) | ongoing [b] | | Procedure D | rug | [c] |

Draft YYYY


AE = adverse event.

<sup>[</sup>a] Age is age at informed consent in years. F = Female, M = Male.

<sup>[</sup>b] Study Day = Onset/Resolution date - date of first dose of study drug + 1. [c] Serious AE criteria are defined in protocol Section 9.6.

| xxx-xxx | Elamipret<br>ide 4 mg | 73/F | XXXXXXXXXXX<br>XXXXXXXXX<br>(XXXXXXXXXX) | yyyy-mmm-dd (xxx)<br>yyyy-mmm-dd (xxx) | Severe Recovered Probably Yes /Resolved Medication related yyyy-mmm-dd Additional case details Relevant diagnostic tests | Interrupted Stopped: yyyy-mmm-dd hh:mm AE abated Restarted: yyyy-mmm-dd hh:mm AE reoccurred | Hospitaliza tion/prolon gation. Admission on yyyymmm-dd Discharged on yyyy-mmm-dd |
|---|---|---|---|---|---|---|---|
| xxx-xxx | | | | | | | |
| | Placebo | 65/M | XXXXXXXXXXX<br>XXXXXXXXX<br>(XXXXXXXXXX) | yyyy-mmm-dd<br>(xxx) ongoing | Severe Not Yes Unlikely recovered Procedure related /not resolved yyyy-mmm-dd Additional case details Relevant diagnostic tests | None | Death on<br>yyyy-mmm-dd<br>Autopsy<br>performed |
| xxx-xxx | Placebo | 65/M | XXXXXXXXXXXX<br>XXXXXXXXXX<br>(XXXXXXXXXX) | yyyy-mmm-dd<br>(xxx) ongoing | Severe Not Yes Unlikely recovered Procedure related /not resolved yyyy-mmm-dd | Permanently<br>discontinued<br>Last dose<br>date<br>yyyy-mmm-dd | xxxxxx |

<sup>[</sup>a] Age is age at informed consent in years. F = Female, M = Male.

Note to Programmer: Listing is sorted by Study Treatment, and Subject ID.

Listing 5.3

Adverse Events Leading to Discontinuation of Study Drug Safety Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

<sup>[</sup>b] Study Day = Onset/Resolution date - date of first dose of study drug + 1. [c] Serious AE criteria are defined in protocol Section 9.6.

| System Organ<br>Class/Preferred Term<br>(Investigator Term) | Subject<br>ID | Study<br>Treatment | Age/<br>Sex<br>[a] | Onset Date (Study day)/Resolution Date(Study Day)/ ongoing [b] | Intensity/<br>Relationship<br>to Study Drug | Outcome | Treatment fo AE? Medication or Procedure AE | Serious |
|---|---|---|---|---|---|---|---|---|
| (XXXXXXXXXX<br>XXXXXXXXX<br>(XXXXXXXXXX) | xxx-xxx | Elamipretide<br>4 mg | 73/F | yyyy-mmm-dd d<br>(xxx)<br>yyyy-mmm-dd (xxx) | Severe<br>Probably<br>related | Recovered/Resolved | Yes<br>Medication | Yes |
| (MAMAMA) | xxx-xxx | Elamipretide<br>40 mg | 78/M | yyyy-mmm-dd (xxx)<br>ongoing | Severe<br>Possibly<br>related | Not recovered/not resolved | Yes<br>Procedure | No |
| XXXXXXXXXXX<br>XXXXXXXXX<br>(XXXXXXXXXX) | xxx-xxx | Placebo | 65/M | yyyy-mmm-dd (xxx)<br>yyyy-mmm-dd (xxx) | xxxxx<br>xxxxxxxxxxx | xxxx/xxxx<br>xxxxxxxx | xxx<br>xxxx | XXX |
| (MMMMMAA) | | Elamipretide<br>4 mg | 68/F | yyyy-mmm-dd (xxx)<br>yyyy-mmm-dd (xxx) | xxxxx/<br>xxxxxxxxxxx | | | XXX |

#### AE = adverse event.

- [a] Age is age at informed consent in years. F = Female, M = Male.
- [b] Study Day = Onset/Resolution date date of first dose of study drug + 1. [c] Serious AE criteria are defined in protocol Section 9.6.

Note to Programmer: Include all AEs with Action taken with study drug = permanently discontinued. Sorted by PT in decreasing order of total frequency, Study Treatment, and Subject ID.

### LISTINGS - LABORATORY DATA

# Listing 6.1 Hematology Results by Subject and Visit Safety Population

| Timepoint | | Sample | <u>Value</u> | Markedly Abnorma | l Criteria |
|---|---|---|---|---|---|
| Subject Study Age/Sex Parameter ID Treatment Screening [a] (Unit) | Sample Date yyyy-mmm-dd | <u>Time</u> | xxx.xx | | Result<br>(N/H/L) |
| Report generated by program: /sasdir/xxxx.sas | | | | Draft | У У У У |

| Elamipret | | | Baseline | yyyy-mmm-dd yyyy- | hh:mm | XXX.XX | Reference Range | N N |
|---|---|---|---|---|---|---|---|---|
| xxx-xxx 4 mg | 73/F | | Week 1 | mmm-dd yyyy-mmm-dd | hh:mm | xxx.xx | Low - high | L |
| | | XXXXXX | Week 2 | yyyy-mmm-dd yyyy- | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | (xxx) | Week 4 | mmm-dd yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | | Week 6 | yyyy-mmm-dd yyyy- | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | | Screening | mmm-dd yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | | Baseline | yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | | Week 1 | yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | Н |
| | | | Week 2 | yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | XXXXXX | Week 4 | yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | (xxx) | Week 6 | yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | | | yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | |
| | | | | yyyy-mmm-dd | hh:mm | xxx.xx | xxxx - xxxx | |
| | | | Screening | | hh:mm | xxx.xx | xxxx - xxxx | N |
| | | | Baseline | | hh:mm | xxx.xx | xxxx - | N |
| | | | Week 1 | | hh:mm | xxx.xx | xxxx xxxx | N |
| | | | Week 2 | | hh:mm | xxx.xx | - xxxx | N |
| xxx-xxx Placebo | 65/M | | Week 4 | | hh:mm | | xxxx - | N |
| AAA AAA TIUCCDO | 00/11 | XXXXXX | Week 6 | | | | XXXX XXXX | N |
| | | (xxx) | | | | | - xxxx | |
| | | | | | | | xxxx - | |
| | | | | | | | xxxx xxxx | |
| | | | | | | | - xxxx | |

N = Normal, H=High, L=Low are based on comparison to the reference ranges. [a] Age is age at informed consent. Sex: M = Male, F = Female.

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


Stealth BioTherapeutics, Inc. Protocol SPIHF-201

Note to Programmer: Listing is sorted by Study Treatment, Subject ID, Parameter, and Timepoint.

Listing 6.2 Blood Chemistry Results by Subject and Visit Safety Population

Note to Programmer: Same layout as Listing 6.1.

Listing 6.3 Urinalysis Results by Subject and Visit Safety Population

Note to Programmer: Layout similar to Listing 6.1. The time points are Screening, Baseline, and Week 4.

Listing 6.4
Levels of hsTroponin by Subject and Visit Safety
Population

Note to Programmer: Layout similar to Listing 6.1. The time points are Baseline, Week 1, Week 2, Week 4, and Week 6. Change "Value" column to "Value (Log Value)".

#### LISTINGS – OTHER SAFETY DATA

Listing 7.1
Vital Signs by Subject and Visit Safety
Population

Report generated by program: /sasdir/xxxx.sas -MM-DD +HH:MM

| Subject | Study | Age/<br>Sex | | | | Temperature | Systolic | Diastolic | Heart Rate | Respiration<br>Rate<br>(breaths/min) |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Treatment<br>Elamipretide | [a] | Timepoint | Date | Time | (°C) | (mmHg) | (mmHg) | (BPM) | |
| xxx-xxx | 4 mg | 73/F | Screening<br>Baseline | yyyy-mmm-dd<br>yyyy-mmm-dd | hh:mm<br>hh:mm | xx.x<br>xx.x | XXX | XXX<br>XXX | xxx<br>xxx | xxx |
| | | | Week 1 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | XXX | XXX |
| | | | Week 2 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | XXX | XXX |
| | | | Week 4 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | xxx | XXX |
| | | | Week 6 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | XXX | xxx |
| xxx-xxx | Placebo | 65/M | Screening | yyyy-mmm-dd | hh:mm | XX.X | XXX | xxx | xxx | xxx |
| | | | Baseline | yyyy-mmm-dd | hh:mm | xx.x | XXX | XXX | XXX | xxx |
| | | | Week 1 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | xxx | xxx |
| | | | Week 2 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | XXX | XXX |
| | | | Week 4 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | XXX | XXX |
| | | | Week 6 | yyyy-mmm-dd | hh:mm | XX.X | XXX | XXX | XXX | XXX |

Blood Pressure

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

BPM = Beats per minute.

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Study Treatment, Subject ID, and Timepoint.

Listing 7.2a
Electrocardiogram (ECG) by Subject and Visit Safety
Population

| Subject ID xxx-xxx | Study Treatment Elamipretide 4 mg | Age/Sex [a]<br>73/F | Timepoint Screening Baseline Week 1 Week 2 Week 4 Week 6 | Date_yyyy-<br>mmm-dd<br>yyyy-mmm-dd<br>yyyy-mmm-dd<br>yyyy-mmm-dd<br>yyyy-mmm-dd | Time Heart hh:mm xxx hh:mm xxx hh:mm xxx hh:mm xxx hh:mm xxx hh:mm xxx | Rate PR (msec) xxx xxx xxx xxx xxx xxx xxx | QRS (msec) xxx xxx xxx xxx xxx xxx xxx | QT (msec) xxx xxx xxx xxx xxx xxx | QTCF(msec) xxx xxx xxx xxx xxx xxx |
|---|---|---|---|---|---|---|---|---|---|
| xxx-xxx | Placebo | 65/M | Screening<br>Baseline<br>Week 1<br>Week 2<br>Week 4<br>Week 6 | yyyy-mmm-dd<br>yyyy-mmm-dd<br>yyyy-mmm-dd<br>yyyy-mmm-dd<br>yyyy-mmm-dd | hh:mm xxx hh:mm xxx hh:mm xxx hh:mm xxx hh:mm xxx | XXX<br>XXX<br>XXX<br>XXX | xxx<br>xxx<br>xxx<br>xxx | XXX<br>XXX<br>XXX<br>XXX | xxx<br>xxx<br>xxx<br>xxx |

<sup>[</sup>a] Age is age at informed consent. Sex: M = Male, F = Female. QTcF

Note to Programmer: Listing is sorted by Study Treatment, Subject ID and Timepoint.

Listing 7.2b
Electrocardiogram (ECG) by Subject and Visit with QRS Duration of <= 110 msec Safety
Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

<sup>=</sup> Fridericia corrected QT interval.

# Listing 7.2c Electrocardiogram (ECG) by Subject and Visit with QRS Duration of >110 msec Safety Population

Listing 7.3

Electrocardiogram (ECG) by Subject and Visit

Subjects with Either an Increase of >60 msec Between Baseline and End of Treatment in Their QT or QTcF or an Absolute QT or QTcF value >500 msec at Any Point in Time

During the Study

Safety Population

| | Subject ID Study Treatment Elamipretide 4 g | Age/Sex [a]<br>73/F | Timepoint Date Screening yyyy-mmm-dd | | Time Heart Rat | | | | <u> </u> |
|---|---|---|---|---|---|---|---|---|---|
| mg | Bramipreerae 4 | 7371 | - | yyyy-mmm-aa<br>yyyy-mmm-dd | hh:mm xxx | xxx | xxx | xxx | xxx |
| | | | Week 1 | yyyy-mmm-dd | hh:mm xxx | XXX | xxx | xxx | xxx |
| | | | Week 2 | yyyy-mmm-dd | hh:mm xxx | XXX | XXX | XXX | XXX |
| | | | Week 4 | yyyy-mmm-dd | hh:mm xxx | xxx | XXX | xxx | xxx |
| | | | Week 6 | yyyy-mmm-dd | hh:mm xxx | XXX | xxx | xxx | XXX |
| xxx-xxx | Placebo | 65/M | Screening | yyyy-mmm-dd | hh:mm xxx | XXX | XXX | XXX | XXX |
| | | | Baseline : | yyyy-mmm-dd | hh:mm xxx | xxx | xxx | xxx | xxx |
| | | | Week 1 | yyyy-mmm-dd | hh:mm xxx | xxx | XXX | xxx | xxx |
| | | | Week 2 | yyyy-mmm-dd | hh:mm xxx | xxx | XXX | xxx | xxx |
| | | | Week 4 | yyyy-mmm-dd | hh:mm xxx | xxx | XXX | xxx | xxx |
| | | | Week 6 | yyyy-mmm-dd | hh:mm xxx | XXX | XXX | xxx | xxx |

[a] Age is age at informed consent. Sex: M = Male, F = Female. QTcF

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


<sup>=</sup> Fridericia corrected QT interval.

-MM-DD HH:MM

Note to Programmer: Listing is sorted by Study Treatment, Subject ID and Timepoint.

Listing 7.4

Cardiovascular Physical Examination and Physical Measurements by Subject and Visit Safety
Population

Subject Study Age/Sex ID Cardiovascular Physical Examination Physical Measurements Treatment [a] Visit Elamipretide 73/F xxx-xxx 4 mg Screening Baseline Week 1 Week 2 Week 4 Week 6 Clinical Clinical Significant Physical Significant Date Examination performed? abnormalities noted? Measurements Performed? abnormalities noted? Weight (kg) Height (cm) BMI (kg/m2) yyyymmm-dd Yes No Yes No xxx.x xxx.x xxx.x yyyymmm-dd Yes No Yes No xxx.x xxx.x xxx.x yyyymmm-dd Yes No Yes No xxx.x xxx.x xxx.x yyyymmm-dd Yes No Yes No xxx.x xxx.x xxx.x yyyymmm-dd No No No ууууmmm-dd Yes No Yes No XXX.X XXX.X XXX.X xxx-xxx Placebo 65/M Screening Report generated by program: /sasdir/xxxx.sas Draft YYYY

| Baseline | уууу- |
|----------|----------------------------------------------|
| | mmm-dd Yes No Yes No xxx.x xxx.x xxx.x yyyy- |
| Week 1 | mmm-dd Yes No Yes No xxx.x xxx.x xxx.x yyyy- |
| | mmm-dd Yes No Yes No xxx.x xxx.x xxx.x yyyy- |
| Week 2 | mmm-dd No No No |
| | уууу- |
| Week 4 | mmm-dd Yes Yes Yes xxx.x xxx.x xxx.x yyyy- |
| F-7 1 C | mmm-dd Yes |
| Week 6 | No |
| | Yes |
| | No xxx.x xxx.x xxx.x |

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Study Treatment, Subject ID, and Timepoint.

Listing 7.5
Injection Site Reaction (Nurse/Investigator Assessment)
Safety Population

| | | | | Surety 1 opular | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject | Study Age/S | ex | | Assessment Not | Injection | | | |
| ID | Treatment | [a] | Date | Completed | Site | Other, Specify | Parameter | Grade |
| | Elamipretide | | | | | | Pain or | |
| xxx-xxx | 4 mg | 73/F | | | | | Tenderness | |
| | | | | | Upper Right | | Erythema or | 1 |
| | | | | | | | Redness | |
| | | | | | Upper Left | | Induration or | 2 |
| | | | yyyy-mmm-dd yyyy- | | | | Swelling | |
| | | | mmm-dd yyyy-mmm-dd | | Lower Right | | | 3 |
| | | | yyyy-mmm-dd | | Lower Left | | Pruritus | 4 |
| | | | yyyy-mmm-dd yyyy- | | | | | |
| | | | mmm-dd | | | | | |
| | | | minit da | | Other | Xxxxxx | | |
| xxx-xxx | | | | | | | | |
| | Placebo | 65/M | yyyy-mmm-dd | | Upper Right | | | |
| | | | yyyy-mmm-dd | | Upper Left | | | |
| | | | yyyy-mmm-dd | | Lower Right | | | |

Report generated by program: /sasdir/xxxx.sas
D r a f t Y Y Y Y -MM-DD HH:MM


yyyy-mmm-dd

Lower Left

yyyy-mmm-dd yyyy-

mmm-dd

Other Xxxxxx

[a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Study Treatment, Subject ID, and Timepoint.

Listing 7.6 Injection Site Reaction Self-Assessment Questionnaire

| | | | | | Safety Pop | ulation | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject S | Study<br>Treatment | Age/Sex<br>[a] | Date | Day | Was the ISR Self- Assessment Questionnaire completed by the subject? | Pain? | Burning<br>Sensati<br>on? | Cold<br>Sensati<br>on? | Itching | Redness | Swellin<br>g? | Bruisin<br>g? |
| | Elamipretide | [~] | 2400 | 241 | 0.10 000,000. | Not at | 011. | 0111 | • | <u> </u> | 9. | |
| xxx-xxx | 4 mg | 73/F | | 1 | Yes | all | | | | | | |
| | | | yyyy-mmm-dd<br>yyyy-mmm-dd | 2 | Yes | | А | Moderat | | | | |
| | | | yyyy-mmm-dd | 3 | Yes | | little | ely | | | | |
| | | | yyyy-mmm-dd<br>yyyy-mmm-dd | 4 | Yes | | | | Very | Extreme<br>ly | | |
| | | | 1111 | 5 | No | | | | | ± | | |
| | | | yyyy-mmm-dd | 6 | Yes | | | | | | | |

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY

1111 00 11111111

| Placebo | 65/M | yyyy-mmm-dd | 1 | Yes |
|---------|------|-------------|---|-----|
| | | yyyy-mmm-dd | 2 | Yes |
| | | yyyy-mmm-dd | 3 | No |
| | | yyyy-mmm-dd | 4 | Yes |
| | | yyyy-mmm-dd | 5 | Yes |
| | | yyyy-mmm-dd | 6 | Yes |

<sup>[</sup>a] Age is age at informed consent. Sex: M = Male, F = Female.

Note to Programmer: Listing is sorted by Study Treatment, Subject ID, and Timepoint.

Listing 7.7 Comments All Subjects

| Thi Subjects | | | | | |
|---|---|---|---|---|---|
| Subject ID | Study Treatment | Age/Sex [a] | Visit | Comments Applies To | Comments |
| XXX-XXX | Elamipretide 4 mg | 73/F | xxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | xxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | xxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxx-xxx | | | | | |
| | Placebo | 65/M | xxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | xxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |

<sup>[</sup>a] Age is age at informed consent. Sex: M = Male, F = Female.

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Note to Programmer: Listing is sorted by Study Treatment, Subject ID, Visit and CRF page.

### **FIGURES**

Figure 1a
Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Elamipretide 4 mg Group (By Subject) ITT
Population

Note: x-axis: Change time points to Screening, Week 1, and Week 4

Figure 1a
Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Elamipretide 4 mg
Group (By Subject)



Figure 1b

Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Elamipretide 4 mg Group (By Subject)
Per-Protocol Population

Figure 1c Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Elamipretide 40 mg Group (By Subject) ITT Population

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

#### Figure 1d Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Elamipretide 40 mg Group (By Subject) Per-Protocol Population

Figure 1e Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Placebo Group (By Subject) ITT Population

Figure 1f Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, for Placebo Group (By Subject) Per-Protocol Population

Figure 1g
LS Mean Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, (By Treatment Group)
ITT Population

Figure 1h
LS Mean Change From Baseline in Left Ventricular End Systolic Volume (LV ESV), Assessed by MRI, (By Treatment Group) PerProtocol Population

Note: For Figures 1g and 1h, only 3 lines, one for Elamipretide 4mg, one for Elamipretide 40 mg, and one for Placebo group. Add SE bar to the plot. Change Subject Number legend to Treatment Group legend.

Figure 2a to Figure 2h (LVEF assessed by MRI)

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Figure 3a to Figure 2h (LV EDV assessed by MRI)

Figure 4a to Figure 4h (LVSV assessed by MRI)

Figure 5a to Figure 5h (LVCO assessed by MRI)

Figure 6a to Figure 6h (LV Myocardial Mass assessed by MRI)

Figure 7a to Figure 7h (RV ESV assessed by MRI)

Figure 8a to Figure 8h (RV EDV assessed by MRI)

Figure 9a to Figure 9h (RVEF assessed by MRI)

Figure 10a to Figure 10h (E/A assessed by Echocardiography)

Figure 11a to Figure 11h (E/e' assessed by Echocardiography)

Figure 12a to Figure 12h (LA Volume assessed by Echocardiography)

Figure 13a to Figure 13h (LV GLS assessed by Echocardiography)

Figure 14a to Figure 14f (LV EDV assessed by Echocardiography)

Figure 15a to Figure 15f (LV ESV assessed by Echocardiography)

Figure 16a to Figure 16f (LVEF Biplane assessed by Echocardiography)

Figure 17a to Figure 17f (LV Mass assessed by Echocardiography)

Figure 18a to Figure 18f (Mitral Regurgitation Severity assessed by Echocardiography)

Figure 19a to Figure 19f (Tricuspid Regurgitation Severity assessed by Echocardiography)

Figure 20a to Figure 20f (RV fractional area change assessed by Echocardiography)

Figure 21a to Figure 21f (RV systolic pressure assessed by Echocardiography)

Figure 22a to Figure 22h (6MWT)

Figure 23a to Figure 23f (NT-pro-BNP)

Figure 24a to Figure 24h (Log10 NT-pro-BNP)

Figure 25a to Figure 25h (hs Troponin)

Figure 26a to Figure 26h (KCCQ)

Figure 27a Mean Plasma Concentration-Time Profile of Elamipretide (Linear Scale) Safety Population



Source: Table 4.1

#### Programmer note:

- 1. AXES: Display nominal time of sample on the X axis (label "Time After Dosing"). Display mean concentration value on the Y axis (label "Mean Plasma Concentration +/- SD <unit>")
- 2. Nominal time points marked on the x axis are Day 1 Pre-Dose, Day 1 45 min Post-Dose, Week 1 Pre-Dose, Week 1 45 min Post-Dose, Week 2 Pre-Dose, Week 2 45 min Post-Dose, Week 4, and Week 6

Report generated by program: /sasdir/xxxx.sas -MM-DD HH:MM

Draft YYYY


3. PLOT TYPE: line and symbol plot with error bars (+/- SD)

Figure 27b
Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M1 (Linear Scale) Safety
Population

Figure 27c Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M2 (Linear Scale) Safety Population

Figure 27d Log Mean Plasma Concentration-Time Profile of Elamipretide (Semi-logarithmic Scale) Safety Population



Source: Table 4.1 and Listing 4.1  $\,$ 

Programmer note:

- 1. AXES: Display nominal time of sample on the X axis (label "Time After Dosing"). Display mean of log concentration value on the Y axis (label "Log Mean Plasma Concentration <unit>")
- 2. Nominal time points marked on the x axis are Day 1 Pre-Dose, Day 1 45 min Post-Dose, Week 1 Pre-Dose, Week 1 45 min Post-Dose, Week 2 Pre-Dose, Week 2 45 min Post-Dose, Week 4, and Week 6
- 3. PLOT TYPE: line and symbol plot

Figure 27e Log Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M1 (Semi-logarithmic Scale) Safety Population

Report generated by program: /sasdir/xxxx.sas

# Figure 27f Log Mean Plasma Concentration-Time Profile of Elamipretide Metabolite M2 (Semi-logarithmic Scale) Safety Population

Figure 27g
Individual Plasma Concentration-Time Profile of Elamipretide (Linear Scale)
Safety Population

#### Similar to Figure 27a without +/- SD source:

#### Listing 4.1

Programmer note:

- 1. All individual profiles superimpose on the same graph
- 2. AXES: Display actual time of sample on the X axis (label "Time After Dosing"). Display concentration value on the Y axis (label "Plasma Concentration, <unit>")
- 3. Nominal time points marked on the x axis are Day 1 Pre-Dose, Day 1 45 min Post-Dose, Week 1 Pre-Dose, Week 1 45 min Post-Dose, Week 2 Pre-Dose, Week 2 45 min Post-Dose, Week 4, and Week 6
- 4. PLOT TYPE: line plot.

Figure 27h Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M1 (Linear Scale) Safety Population

Figure 27i Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M2 (Linear Scale) Safety Population

Figure 27j Individual Plasma Concentration-Time Profile of Elamipretide (Semi-logarithmic Scale) Safety Population

## Similar to Figure 27d

Source: Listing 4.1 Programmer note:

Report generated by program: /sasdir/xxxx.sas

-MM-DD HH:MM

- 1. All individual profiles superimpose on the same graph
- 2. AXES: Display actual time of sample on the X axis (label "Time After Dosing"). Display log concentration value on the Y axis (label "Log Plasma Concentration, <unit>")
- 3. Nominal time points marked on the x axis are Day 1 Pre-Dose, Day 1 45 min Post-Dose, Week 1 Pre-Dose, Week 1 45 min Post-Dose, Week 2 Pre-Dose, Week 2 45 min Post-Dose, Week 4, and Week 6
- 4. PLOT TYPE: line plot.

## Figure 27k

Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M1 (Semi-logarithmic Scale)
Safety Population

Figure 271

Individual Plasma Concentration-Time Profile of Elamipretide Metabolite M2 (Semi-logarithmic Scale)
Safety Population

Similar to Figure 1a

Figure 28a

QTc for Subjects with a QTc value >500 msec at Any Point in Time During the Study (By Subject) Safety Population

Note:

- 1. x-axis: Change time points to Screening, Baseline, Weeks 1,2, 4, and 6
- 2. Only generate figure if there is at least one subject who meets the criteria

Report generated by program: /sasdir/xxxx.sas -MM-DD +HH:MM